

#### CLINICAL STUDY PROTOCOL

Study Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Efficacy

and Safety of Sofosbuvir/Velpatasvir Fixed Dose Combination in Subjects with Chronic HCV Infection who have received a Liver

Transplant

Sponsor: Gilead Sciences, Inc.

333 Lakeside Drive

Foster City, CA 94404, USA

**IND Number:** This is a non-IND study

**EudraCT Number:** 2016-000416-15 **Clinical Trials.gov** Not Available

Identifier:

**Indication:** Hepatitis C Virus Infection

Protocol ID: GS-US-342-2104

Gilead Study Director Name: Brian McNabb, M.D.

or Medical Monitor: Telephone:

Fax: PPD PPD

Protocol Version/Date: Original: 19 February 2016

# CONFIDENTIALITY STATEMENT

The information contained in this document, particularly unpublished data, is the property or under control of Gilead Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Gilead Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# TABLE OF CONTENTS

| TA | BLE O | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF I | N-TEXT TABLES | 5 |
| PRO | OTOCO | OL SYNOPSIS | 6 |
| GL | OSSAF | RY OF ABBREVIATIONS AND DEFINITION OF TERMS | 10 |
| 1. | INTR | RODUCTION | 13 |
| | 1.1. | Background | |
| | 1.1. | Sofosbuvir/Velpatasvir Fixed Dose Combination (SOF/VEL FDC) | |
| | | 1.2.1. General Information | |
| | | 1.2.2. Additional Clinical Experience | |
| | 1.3. | Rationale for This Study | |
| | 1.4. | Rationale for Dose Selection | |
| | 1.5. | Risk/Benefit Assessment for the Study | |
| | 1.6. | Compliance | |
| 2. | OBJE | ECTIVES | 39 |
| 3. | STUI | DY DESIGN | 40 |
| | 3.1. | Treatment Plan and Regimen | 40 |
| | 3.2. | Visit Schedule | |
| | 3.3. | HCV Virologic Response-Based Stopping Criteria | |
| | 3.4. | Stopping Rules for Individual Subjects | 41 |
| | 3.5. | Discontinuations. | |
| | 3.6. | Assessments for Premature Discontinuation from Study | |
| | 3.7. | Criteria for Discontinuation of Study Treatment | |
| | 3.8. | Biomarker Testing | |
| | | 3.8.2. Biomarker Samples for Optional Pharmacogenomics Research | |
| 4 | CI ID | JECT POPULATION | |
| 4. | | | |
| | 4.1. | Number of Subjects and Subject Selection | |
| | 4.2.<br>4.3. | Inclusion Criteria | |
| | | Exclusion Criteria. | |
| 5. | INVE | ESTIGATIONAL MEDICINAL PRODUCTS | 49 |
| | 5.1. | Enrollment and Study Drug Supply | |
| | 5.2. | Description and Handling of SOF/VEL FDC | |
| | | 5.2.1. Formulation | |
| | | 5.2.2. Packaging and Labeling | |
| | 5.3. | 5.2.3. Storage and Handling Dosage and Administration | |
| | 5.4. | Prior and Concomitant Medications | |
| | J. <b>T.</b> | 5.4.1. Colony Stimulating Agents | |
| | 5.5. | Management of Rejection | |
| | 5.6. | Study Drug Accountability | 52 |
| | | 5.6.1. Study Drug Return and Disposal | 53 |
| 6. | STUI | DY PROCEDURES | 54 |
| | 6.1. | Screening Assessments | 54 |
| | J.1. | 6.1.1 Screening Visit (Day 28 to Day 0) | |

| | 6.2. | Treatment Assessments | 56 |
|---|---|---|---|
| | | 6.2.1. Baseline/Day 1 Visit | 56 |
| | | 6.2.2. Week 2 (± 3 days) | 57 |
| | | 6.2.3. Weeks 4 and 8 (± 3 days) | 58 |
| | | 6.2.4. Week 12 (± 3 days) or Early Termination (ET) | |
| | | 6.2.5. Unscheduled Visit | |
| | 6.3. | Post-treatment Assessments | |
| | | 6.3.1. Post-treatment Week 4 (±5 days) | |
| | | 6.3.2. Post-treatment Week 12 (± 5 days) | |
| | 6.4. | Confirmatory Visit | |
| | 6.5. | End of Study. | |
| | 6.6. | Procedures and Specifications. | |
| | 0.0. | 6.6.1. Clinical Laboratory Analytes | |
| | | 6.6.2. Medical History | |
| | | 6.6.3. Complete Physical Examination. | |
| | | 6.6.4. Vital Signs | |
| | | 6.6.6. Child-Pugh Score | |
| | | 6.6.7. 12-Lead ECG | |
| | | 6.6.8. HCV Viral RNA Sequencing/ Phenotyping (Archive) | |
| | | 6.6.9. Single Pharmacokinetic (PK) Sample | |
| | | 6.6.10. Pharmacogenomics Testing | |
| | | 6.6.11. Sample Storage | |
| | | 6.6.12. Pregnancy Testing | 64 |
| 7. | ADV | ERSE EVENTS AND TOXICITY MANAGEMENT | 65 |
| • | | | |
| | 7.1. | Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events | |
| | | 7.1.1. Adverse Events | |
| | | 7.1.2. Serious Adverse Events | 65 |
| | | 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as | |
| | | Adverse Events or Serious Adverse Events | |
| | 7.2. | Assessment of Adverse Events and Serious Adverse Events | |
| | | 7.2.1. Assessment of Causality for Study Drugs and Procedures | |
| | | 7.2.2. Assessment of Severity | 67 |
| | 7.3. | Investigator Requirements and Instructions for Reporting Adverse Events and Serious | |
| | | Adverse Events to Gilead | 67 |
| | 7.4. | Gilead Reporting Requirements | 69 |
| | 7.5. | Toxicity Management | 69 |
| | | 7.5.1. Subject Stopping Rules | 69 |
| | 7.6. | Special Situations Reports | |
| | | 7.6.1. Definitions of Special Situations | |
| | | 7.6.2. Instructions for Reporting Special Situations | |
| O | CTAT | ISTICAL CONSIDERATIONS | |
| 8. | SIAI | ISTICAL CONSIDERATIONS | 12 |
| | 8.1. | Analysis Objectives and Endpoints | 72 |
| | | 8.1.1. Analysis Objectives | 72 |
| 7. A 7 7 7 7 7 8. S 8 | | 8.1.2. Primary Endpoint | 72 |
| | | 8.1.3. Secondary Endpoints | 72 |
| | | 8.1.4. Other Endpoints of Interest | |
| | 8.2. | Analysis Conventions. | |
| | | 8.2.1. Analysis Sets | |
| | 8.3. | Data Handling Conventions | |
| | 8.4. | Demographic Data and Baseline Characteristics | |
| | 8.5. | Efficacy Analysis | |
| | | · · · · y = =====- y === · | |

| | | 8.5.1. | Primary Analysis | 74 |
|---|---|---|---|---|
| | | 8.5.2. | Secondary Analyses | |
| | 8.6. | Safety A | Analysis | 75 |
| | | 8.6.1. | Extent of Exposure | 75 |
| | | 8.6.2. | Adverse Events | 75 |
| | | 8.6.3. | Laboratory Evaluations | 76 |
| | | 8.6.4. | Other Safety Evaluations | 76 |
| | 8.7. | Pharma | cokinetic Analysis | 76 |
| | 8.8. | Sample | Size | 77 |
| 9. | RESP | ONSIBIL | ITIES | 78 |
| | 9.1. | Investio | ator Responsibilities | 78 |
| | J.1. | 9.1.1. | Good Clinical Practice. | |
| | | 9.1.2. | Independent Ethics Committee (IEC) Review and Approval | |
| | | 9.1.3. | Informed Consent | |
| | | 9.1.4. | Confidentiality | |
| | | 9.1.5. | Study Files and Retention of Records | |
| | | 9.1.6. | Case Report Forms | |
| | | 9.1.7. | Study Drug Return and Disposal | |
| | | 9.1.8. | Inspections. | |
| | | 9.1.9. | Protocol Compliance | |
| | 9.2. | Sponsor | Responsibilities | |
| | | 9.2.1. | Protocol Modifications | |
| | | 9.2.2. | Study Report and Publications | 82 |
| | 9.3. | Joint In | vestigator/Sponsor Responsibilities | |
| | | 9.3.1. | Payment Reporting | 82 |
| | | 9.3.2. | Access to Information for Monitoring | |
| | | 9.3.3. | Access to Information for Auditing or Inspections | 83 |
| | | 9.3.4. | Study Discontinuation | 83 |
| 10. | REFE | ERENCES | | 84 |
| 11. | APPE | ENDICES | | 8 |
| | | | | 0.4 |
| | | ndix 1. | Investigator Signature Page | |
| | | ndix 2. | Study Procedures Table | |
| | | ndix 3. | GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities | |
| | | ndix 4. | Child-Pugh-Turcotte Classification of the severity of cirrhosisa | |
| | | ndix 5. | Banff Criteria* Programmy Programing Definition for Family of Childhousing Potential and | 114 |
| | Appe | ndix 6. | Pregnancy Precautions, Definition for Female of Childbearing Potential, and | 114 |
| | | | Contraceptive Requirements | 1 1 7 |

# LIST OF IN-TEXT TABLES

| Table 1-1. | GS-US-342-1138: SVR12 Overall and by HCV Genotypes | 17 |
|---|---|---|
| Table 1-2. | NGMN, NG, EE, and VEL Plasma PK Parameters Following Administration of | |
| | NGM/EE alone or with VEL | 32 |
| Table 1-3. | Summary of LH, FSH, and Progesterone Concentrations Following Administration | |
| | of NGM/EE alone or with VEL | 33 |
| Table 1-4. | Summary of Changes in SOF/VEL PK following administration with | |
| | Representative H2RAs and PPIs | 35 |
| Table 5-1. | List of Disallowed/ Use with Caution Medications | |

# PROTOCOL SYNOPSIS

# Gilead Sciences, Inc. 333 Lakeside Drive Foster City, CA 94404, USA

| Study Title: | A Phase 2, Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed Dose Combination in Subjects with Chronic HCV Infection who have received a Liver Transplant |
|---|---|
| IND Number:<br>EudraCT Number:<br>Clinical Trials.gov<br>Identifier: | This is a non-IND study 2016-000416-15<br>Not Available |
| Study Centers<br>Planned: | Approximately 18 centers in the United Kingdom, Spain and Switzerland |
| Number of Subjects<br>Planned: | Approximately 80 subjects with chronic hepatitis C virus (HCV) infection who have received a liver transplant. |
| Target Population: | Male and non-pregnant/non-lactating female subjects with chronic hepatitis C virus (HCV) infection who have received a liver transplant, ages 18 years or older. |
| | The enrollment target for subjects with genotype 3 HCV infection is approximately 20%. The enrollment target for subjects with Metavir stage 3 or 4 fibrosis/cirrhosis or corresponding fibrosis degree is approximately 20%. |
| Duration of<br>Treatment: | Enrolled subjects will receive study treatment for 12 weeks |
| Objectives: | The primary objectives of this study are: |
| | • To evaluate the efficacy of study treatment with sofosbuvir (SOF)/velpatasvir (VEL, GS-5816) fixed dose combination (FDC) for 12 weeks as measured by the proportion of subjects with sustained virologic response 12 weeks after cessation of study treatment regimen(SVR12) |
| | • To evaluate the safety and tolerability of the study treatment regimen |
| | The secondary objectives of this study are: |
| | <ul> <li>To determine the proportion of subjects who attain SVR at</li> <li>4 weeks after cessation of the study treatment regimen (SVR4)</li> </ul> |

- To evaluate the kinetics of circulating HCV RNA during study treatment and after cessation of study treatment regimen
- To evaluate the emergence of viral resistance to SOF and VEL (GS-5816) during study treatment and after cessation of study treatment regimen

The exploratory objective of this study is:



#### Study Design:

Approximately 80 subjects with chronic hepatitis C virus (HCV) infection who have received a liver transplant will be enrolled and treated with SOF/VEL FDC tablet once daily for 12 weeks.

The enrollment target for subjects with genotype 3 HCV infection is approximately 20%. The enrollment target for subjects with Metavir stage 3 or 4 fibrosis/cirrhosis or corresponding fibrosis degree is approximately 20%.

# Substudies and Registry Studies:

# Pharmacogenomics (PG) Substudy

In consenting participants, blood samples will be drawn at Baseline or during the study for pharmacogenomics research.

# Diagnosis and Main Eligibility Criteria:

Chronic HCV infected, post-liver transplant, male and non-pregnant/non-lactating female subjects without cirrhosis or with compensated cirrhosis, ages 18 years or older.

Refer to Sections 4.2 and 4.3 of the protocol for detailed Inclusion and Exclusion Criteria.

# Study Procedures/ Frequency:

Screening assessments will be completed within 28 days of the Baseline/Day 1 visit. (Screening period may be extended up to 42 days for those requiring liver biopsy, or additional HCV genotype testing or for extenuating circumstances.)

All subjects will complete the following study visits: Screening, Baseline/Day 1, on-treatment visits at the end of Weeks 2, 4, 8, and 12, and post-treatment visits at Weeks 4 and 12 after completion of study treatment.

Screening assessments will include physical examination, medical history, height, weight, vital signs, 12-lead ECG, adverse events related to screening procedures, concomitant medications, safety laboratory tests (including hematology, chemistry, and coagulation),

HCV RNA, serology (HIV, HCV, HBV), hemoglobin A1c (HbA1c), assessment of the presence or absence of cirrhosis, screening for hepatocellular carcinoma, serum  $\beta$ -hCG (females of child bearing potential only), IL28B genotyping, urinalysis and urine drug screen.

On-treatment assessments include adverse events (AEs), concomitant medications, study medication pill count, physical examination, weight, vital signs, safety laboratory tests, HCV RNA, and urine pregnancy tests (females of child bearing potential only).

Post-treatment assessments include AEs, concomitant medications, vital signs, safety laboratory tests, HCV RNA, and urine pregnancy tests (females of child bearing potential only).

Samples for viral RNA sequencing / phenotyping will be collected at Baseline and every visit thereafter. Samples will be collected during on-treatment visits for pharmacokinetic (PK) analysis of study drug.

For subjects who provide their additional and specific consent, an appropriate blood sample will be collected at the Baseline/Day 1 visit for PG (this sample may be drawn after Baseline/Day 1 if necessary).

Plasma samples may be collected at Baseline/Day 1, Week 12, or ET visits and PPD

Test Product, Dose, and Mode of Administration:

SOF/VEL FDC is manufactured as a 400/100mg FDC tablet for oral administration. Subjects will take 1 tablet once daily with or without food for 12 weeks.

# Criteria for Evaluation:

Safety: AEs and laboratory tests will be collected throughout the study.

Efficacy: Efficacy will be evaluated using scheduled assessments of HCV RNA

performed using COBAS® AmpliPrep®/COBAS® TaqMan® HCV

Quantitative Test, v2.0.

Pharmacokinetics: A single PK blood sample will be collected at each on-treatment visit

for all subjects.

The PK of SOF (and metabolites) and VEL may be assessed.

Statistical Methods: The primary efficacy endpoint for the study is SVR12 in all enrolled

and treated subjects.

In the primary efficacy analysis, point estimate and 95% confidence

interval of SVR12 will be computed.

Secondary efficacy endpoints include SVR4 and the proportion of subjects with virologic failure.

All continuous endpoints (except for safety endpoints) will be summarized using an 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum). All categorical endpoints will be summarized by number and percentage of subjects who meet the endpoint definition.

Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical values or 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data.

With a sample size of 80, a two-sided 95% exact confidence interval will extend at most 23% in length.

This study will be conducted in accordance with the guidelines of Good Clinical Practice (GCP) including archiving of essential documents.

#### GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS

° C degrees Celsius ° F degrees Fahrenheit

ACR Acute Cellular Rejection

AE adverse event

ALT alanine aminotransferase
ANC absolute neutrophil counts
APRI AST: platelet ratio index

APTT activated partial thromboplastin time

AST aspartate aminotransferase AUC area under the curve

AUC<sub>tau</sub> area under the plasma concentration versus time curve over the dosing interval (tau)

β-hCGβ-human chorionic gonadotropinBLQbelow the lower limit of quantification

BMI body mass index
CI confidence interval
CLcr creatinine clearance

Cmax the maximum observed serum/plasma/peripheral blood mononuclear (PBMC)

concentration of drug

CK creatine kinase

CPT Child-Pugh-Turcotte Classification

CRF case report form(s)

CRO Contract (or clinical) research organization

CSA colony stimulating agents
DAA direct acting antiviral

DCV daclatasvir (HCV NS5A Inhibitor)

DDI drug-drug interaction

DSPH Drug Safety and Public Health

EC Ethics committee
ECG electrocardiogram
EDC electronic data capture

eCRF electronic case report form(s)
ESA erythropoiesis-stimulating agents

ET early termination EU European Union

EudraCT European clinical trials database

FAS full analysis set

FDA (United States) Food and Drug Administration

FDC fixed dose combination

FSH follicle stimulating hormone

GCP Good Clinical Practice (Guidelines)

GM-CSF Granulocyte macrophage colony stimulating factor

GSI Gilead Sciences, Inc.
GT genotype (viral)

H2RA Histamine-2 receptor antagonist

Hb Hemoglobin
HbA1C Hemoglobin A1C

hCG human chorionic gonadotropin HDPE high-density polyethylene

HCV Hepatitis C virus

HIV Human Immunodeficiency Virus

HLGT high-level group term HLT high-level term

IB investigator's brochure
ICF Informed Consent Form

ICH International Conference on Harmonisation

IEC independent ethics committee

IFN interferon

IL28B interleukin-28B gene

IMP Investigational Medicinal Product

IND Investigational New Drug (Application)

INR international normalized ratio of prothrombin time

IRB institutional review board

IUD intrauterine device

IWRS interactive web response system

LAM lactational amenorrhea method

LDV ledipasvir

LFT liver function test
LH luteinizing hormone

LLN lower limit of the normal range LLOQ lower limit of quantification

LLT lower-level term
LT liver transplantation

MELD Model for End Stage Liver Disease

MedDRA Medical Dictionary for Regulatory Activities

mg Milligram
min Minute
mL milliliter

mmHg millilimeter mercury

MCV mean cellular volume
NDA New Drug Application

ng nanogram

ng•h/mL nanograms times hours per milliliter

NG norgestrel NGM norgestimate

NGM/EE norgestimate/ethinyl estradiol

NGMN norelgestromin

NS (3/4A/5A/5B) Non-structural protein OC oral contraceptive

PCR Polymerase chain reaction Peg-IFN Pegylated-Interferon- $\alpha$ 

pg pictogram

pg•h/mL picograms times hours per milliliter

P-gp P-glycoprotein
PK pharmacokinetic
PPI Proton pump inhibitor

PT Preferred term or prothrombin time

RBC Red blood cell count

RBV ribavirin

RNA ribonucleic acid

SADR serious adverse drug reaction

SAE serious adverse event
SAP Statistical Analysis Plan
SD Standard deviation
SOC System Organ Class

SOF Sovaldi® or Sofosbuvir, formerly GS-7977

SOF/VEL SOF/VEL fixed dose combination

SUSAR Suspected Unexpected Serious Adverse Reaction

SVR Sustained virologic response

 $t_{max}$  The time (observed time point) of  $C_{max}$ 

 $t_{1/2}$  An estimate of the terminal elimination half-life of the drug in

serum/plasma/PBMC, calculated by dividing the natural log of 2 by the terminal

elimination rate constant  $(\lambda_z)$ 

ULN upper limit of the normal range

US United States
VA Veterans Affairs

VEL Velpatasvir, formerly GS-5816

WBC White blood cell count

#### 1. INTRODUCTION

# 1.1. Background

Hepatitis C virus (HCV) infection is a global health challenge with an estimated 150 million individuals infected worldwide {World Health Organization (WHO) 2014}. Chronic HCV infection remains a leading cause of chronic hepatitis, cirrhosis, and liver cancer and a primary indication for liver transplantation in the Western world. In the United States, between 1995 and 2010 there were 52,000 HCV-associated liver transplants {Biggins et al 2012}. These patients universally experience postoperative recurrence of HCV {Feray et al 1992, Wiesner et al 2003, Wright et al 1992}, and are particularly vulnerable to complications associated with HCV recurrence including cirrhosis, fibrosing cholestatic hepatitis, graft loss, liver re-transplantation, and death {Berenguer 2002, Crespo et al 2012, Gane 2008, Prieto et al 1999, Wiesner et al 2003}, {Berenguer et al 2000, Charlton et al 2004, Firpi et al 2009, Forman et al 2002}. Therefore, treating HCV recurrence is of great importance to patients who have undergone a liver transplantation.

Interferon with ribavirin regimens have been studied as a means to either prevent or treat HCV reoccurrence in patients awaiting transplants and those who have already received transplants, respectively{Calmus et al 2012, Carrion et al 2007, Crippin et al 2002, Forns et al 2003, Samuel et al 2003, Terrault 2008, Wang et al 2006}. Not only are sustained virologic response rates low in these trials, but interferon based therapy is often poorly tolerated in this complex population. The development of Sovaldi® (sofosbuvir, SOF), a nucleotide analog HCV NS5B polymerase inhibitor, represents a major advance in the treatment of HCV as SOF based regimens are shorter in duration, better tolerated and result in higher SVR rates than prior therapies. SOF is currently approved in the US for the treatment of genotype (GT) 1, 2, 3 and 4 HCV infection and in the European Union for GT1-6, with different regimens and durations dependent on the HCV genotype {Gilead Sciences Inc 2013}. SOF is also approved in both the US and Europe to be used in combination with ribavirin in patients awaiting liver transplantation in order to prevent HCV reoccurrence, and in Europe in patients who have already received liver transplants {Gilead Sciences Inc 2013}. SVR 12 rates in the case of HCV recurrence and post-transplant virologic response rates in the case of prevention of HCV recurrence range from 60-70%, and represent significant advances. However, there remains room for more potent therapies to improve upon these results in this complex population.

The next wave of therapies for the treatment of HCV includes combinations of direct acting antivirals (DAAs) including SOF that offer even higher response rates without the need for pegylated interferon (PEG-IFN), and often without the need for ribavirin, depending on patient characteristics and HCV genotype. The first of these treatments, a fixed dose combination (FDC) of SOF and the HCV nonstructural protein 5A (NS5A) inhibitor ledipasvir (LDV) has been approved in the US for genotypes 1, 4, 5, and 6 {Gilead Sciences Inc 2015} and Europe for genotypes 1, 3, 4, 5 and 6 infections {Gilead Sciences International Limited 2014}. LDV/SOF has been studied in combination with ribavirin in patients after liver transplantation in 2 phase 2 trials: SOLAR 1 which was primarily conducted in the US and SOLAR 2 which was conducted in Europe, Canada, Australia, and New Zealand {Charlton et al 2015, Manns et al 2016}. In both

trials, post-transplant patients with genotypes 1 and 4 HCV with and without cirrhosis were treated with 12 or 24 weeks of LDV/SOF with ribavirin. In SOLAR 1 SVR 12 rates were 96-98% in patients with no or CPT class A cirrhosis, while they were 60-88% in patients with CPT class B or C cirrhosis. In SOLAR 2 SVR 12 rates were 93-100% in genotype 1 HCV patients with no or CPT class A cirrhosis, while they were 50-100% in patients with CPT class B or C cirrhosis. Currently, LDV/SOF in combination with ribavirin is approved in Europe for the treatment of genotypes 1, 4, 5, 6 HCV in patients after liver transplantation. There are no currently approved ribavirin-free regimens for treatment of HCV in patients with who have had a liver transplant. LDV/SOF (without ribavirin) for 12 weeks (in patients without cirrhosis) or 24 weeks (in patients with cirrhosis) may be considered for patients who are ineligible for or intolerant to ribavirin.

Most HCV drug development efforts have been focused on GT1 HCV infection as this is the most prevalent HCV genotype in developed countries {Gower et al 2014}. However, over half of all HCV infections are non-GT1: estimates from 2 recent meta-analyses indicate GT3 HCV is the next most common accounting for 22-30% of infections, while GT2 and GT4 each account for approximately 8 to 13%, GT6 for approximately 2 to 5%, and GT5 for approximately 1% of HCV infections worldwide. Among patients with liver transplantation, non-GT1 HCV infections are also high. In the US, about 20% of HCV infections among liver transplant recipients are non-GT1 (Campos-Varela et al 2015, Lim 2015). In Spain, approximately 15% of HCV infections among patients with liver transplants are non-GT1 (10% GT1a, 75% GT1b, 2% GT2, 5% GT3, and 5% GT4){Forns et al 2003}. The number of non-GT1 HCV infections is even higher in other countries that perform liver transplantation, and reflects the country specific background prevalence's of HCV genotypes. In the United Kingdom, 40% of HCV infections among patients with liver transplants are GT3, 40% of HCV infections are non-GT-1 among Korean liver transplant recipients, and 45% are non-GT1 among Australia and New Zealand liver transplant recipients) {Kim et al 2016, Zekry et al 2003}. The availability of a welltolerated, all oral, ribavirin-free, short duration therapy such as SOF/VEL that is effective across all HCV genotypes would be a major advance for the treatment of HCV infection globally. This is particularly true for patients with liver transplants who often have reduced blood cell counts or GFRs at baseline, making them susceptible to ribavirin-associated toxicities. There are no approved ribavirin-free regimens for these patients, regardless of genotype

# 1.2. Sofosbuvir/Velpatasvir Fixed Dose Combination (SOF/VEL FDC)

SOF/ velpatasvir (VEL, GS-5816) fixed-dose combination (SOF/VEL FDC) combines two HCV specific DAAs into a single tablet for the treatment of chronic HCV infection.

SOF is a nucleotide analog HCV NS5B polymerase inhibitor currently approved in the US and other regions for the treatment of HCV infection as described in Section 1.1. VEL (formerly known as GS-5816) is a HCV NS5A inhibitor that has demonstrated activity against HCV in phase 1, phase 2, and phase 3 studies. VEL showed activity against genotypes 1, 2, 3 and 4 HCV in a phase 1, 3 day, monotherapy study. Phase 2 studies of SOF + VEL administered as single agents have demonstrated that the combination of SOF 400 mg and VEL 100 mg administered for 12 weeks is well tolerated and results in high SVR rates across a broad range of HCV

genotypes. The SOF/VEL FDC (400/100 mg) is a co-formulation of SOF 400 mg and VEL 100 mg which is currently being developed as a treatment for HCV through several completed and several ongoing phase 3 trials described in detail in Section 1.2.2.2.

The development of SOF/VEL may have a major impact on the global prevalence and burden of HCV as it may represent a simple, well tolerated, highly efficacious pangenotypic treatment for all HCV infected patients.

#### 1.2.1. General Information

Please refer to the Investigator's Brochure (IB) for additional information on SOF/VEL, and the individual components, including:

- In-Vitro Anti-Hepatitis C Virus Activity
- Nonclinical Pharmacokinetics and In Vitro Metabolism
- Nonclinical Pharmacology and Toxicology
- Clinical Experience

# **1.2.2.** Additional Clinical Experience

#### 1.2.2.1. SOF/VEL Phase 2 and 3 Studies

Four Phase 3 studies have been completed evaluating the efficacy and safety of SOF/VEL in subjects with genotype 1-6 HCV infection. Three studies enrolled subjects without cirrhosis or with compensated cirrhosis, GS-US-342-1138 (ASTRAL-1), GS-US-342-1139 (ASTRAL-2) and GS-US-342-1140 (ASTRAL-3); and one study enrolled subjects with decompensated cirrhosis GS-US-342-1137 (ASTRAL-4). Three Phase 3 trials enrolling patients with HIV-1 coinfection (GS-US-342-1202 [ASTRAL-5]), patients who failed to achieve SVR 12 in previous Gilead sponsored HCV treatment studies (GS-US-342-1553), and patients who received placebo during ASTRAL-1 (GS-US-342-1446) are currently ongoing. Summaries of results from the completed Phase 3 studies and descriptions of the ongoing Phase 3 studies are presented below.

#### 1.2.2.1.1. Study GS-US-342-1138 (ASTRAL-1)

#### Design

This ongoing Phase 3, randomized, double-blind, placebo-controlled, multicenter, international study is assessing the antiviral efficacy, safety, and tolerability of 12 weeks of SOF/VEL treatment compared with 12 weeks of SOF/VEL placebo treatment in subjects with chronic genotype 1, 2, 4, 5, or 6 hepatitis C virus (HCV) infection. This study was conducted in Belgium, Canada, France, Germany, Hong Kong, Italy, United Kingdom, United States.

Subjects with genotype 1, 2, 4, or 6 HCV infection were randomized in a 5:1 ratio to treatment with SOF/VEL for 12 weeks (SOF/VEL 12 Week group) or SOF/VEL placebo for 12 weeks (Placebo 12 Week group). Subjects with genotype 5 HCV infection were enrolled to the SOF/VEL 12 Week group. Randomization was stratified by HCV genotype (1, 2, 4, 6, and indeterminate) and the presence or absence of cirrhosis at screening.

# Disposition

A total of 740 subjects were enrolled and treated; 624 subjects in the SOF/VEL 12 Week group and 116 subjects in the Placebo 12 Week group.

The majority of subjects (99.3%) completed study treatment. Five subjects (0.7%) prematurely discontinued study treatment; 2 subjects in the SOF/VEL group and 3 subjects in the placebo group. The reasons for premature discontinuation of study drug for subjects in the SOF/VEL 12 Week group were an AE (1 subject) and lost to follow-up (1 subject) and for subjects in the Placebo 12 Week group were AEs (2 subjects) and investigator discretion (1 subject).

# **Demographics and Baseline Characteristics**

Demographics and baseline disease characteristics were generally balanced between the SOF/VEL 12 Week and Placebo 12 Week groups.

In the SOF/VEL 12 Week group, the majority of subjects were male (59.9%), and 21.6% of subjects had a body mass index (BMI)  $\geq$  30 kg/m², 19.4% had cirrhosis and most subjects (73.9%) had baseline HCV RNA  $\geq$  800,000 IU/mL. Of the 624 subjects who received SOF/VEL, 328 subjects (52.6%) had genotype 1 HCV infection (210 subjects [33.7%] with HCV genotype 1a and 118 subjects [18.9%] with HCV genotype 1b), 104 subjects (16.7%) had genotype 2 HCV infection, 116 subjects (18.6%) had genotype 4 HCV infection, 35 subjects (5.6%) had genotype 5 HCV infection, and 41 subjects (6.6%) had genotype 6 HCV infection.

#### **Efficacy Results**

The SOF/VEL 12 Week group met the primary endpoint of an SVR12 rate that was statistically superior relative to the prespecified performance goal of 85% (p < 0.001). The SVR12 rate was as follows:

SOF/VEL 12 Week group: 99.0% (95% CI: 97.9% to 99.6%) of subjects (618 of 624) achieved SVR12.

Table 1-1 presents the SVR12 results for the SOV/VEL 12 Week group overall and by HCV genotype. A total of 6 of 624 subjects (1.0%) who received SOF/VEL did not achieve SVR12. Two subjects had relapse determined at post-treatment week 4; one treatment-naive subject with genotype 1a HCV infection without cirrhosis and one treatment experienced subject with genotype 1b infection and cirrhosis. Four additional subjects (3 with genotype 1 and 1 with genotype 5) did not achieve SVR12 (1 subject withdrew consent, 2 subjects had not returned for the post-treatment Week 12 visit, and 1 subject died prior to the post-treatment Week 4 visit).

| | | SOF/VEL<br>12 Weeks | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Total (All Genotypes) (N = 624) | GT-1a<br>(N = 210) | GT-1b<br>(N = 118) | GT-1<br>Total<br>(N = 328) | GT-2<br>(N = 104) | GT-4<br>(N = 116) | GT-5<br>(N = 35) | GT-6<br>(N = 41) |
| SVR12 | 618/624<br>(99.0%) | 206/210<br>(98.1%) | 117/118<br>(99.2%) | 323/328<br>(98.5%) | 104/104<br>(100.0%) | 116/116<br>(100.0%) | 34/35<br>(97.1%) | 41/41<br>(100.0%) |

Table 1-1. GS-US-342-1138: SVR12 Overall and by HCV Genotypes

GT = genotype

The SVR4 results for subjects with genotype 1, 2, 4, 5, or 6 HCV infection were the same as the SVR12 results with the exception of 1 subject with genotype 1a HCV infection who achieved SVR4 but had not returned for his post-treatment Week 12 visit at the time of the interim analysis.

HCV RNA declined rapidly with similar decreases in HCV RNA observed across all HCV genotypes in the SOF/VEL 12 Week group. Consistent with the rapid and sustained decline in HCV RNA, > 88.5% of subjects in the SOF/VEL 12 Week group had HCV RNA < LLOQ at Week 4. Time to virologic suppression was not associated with treatment outcome overall or in any genotype.

#### Virologic Resistance

Deep sequence analyses indicated that subjects in the SOF/VEL 12 Week group had a diverse population of HCV with more than 30 subtypes across genotypes 1, 2, 4, 5, 6, and 7.

Approximately 42% and 9% of subjects in the SOF/VEL 12 Week group had baseline NS5A resistance-associated variants (RAVs) and NS5B RAVs, respectively. Baseline NS5A or NS5B RAVs had no impact on SVR12, with high SVR12 across all subtypes/genotypes regardless of the presence of NS5A RAVs or NS5B RAVs. Two subjects had virologic failure and both had baseline NS5A RAVs. At virologic failure time points, both subjects developed additional NS5A RAVs (Y93N and Y93H) that conferred a high (> 700) fold shift in EC<sub>50</sub> to VEL. No NS5B RAVs were detected at baseline or post-treatment in either subject with virologic failure.

# **Safety Results**

Treatment with SOF/VEL was well tolerated. Subjects in the SOF/VEL 12 Week treatment group had similar type, incidence, and severity of AEs as subjects in the Placebo 12 Week group.

Grade 3 (severe) and Grade 4 (life-threatening) AEs were rare, 19 of 624 (2.9%) in the SOF/VEL 12 Week group and 1 of 116 (0.9%) in the Placebo 12 Week group. Two subjects (0.3%) in the SOF/VEL 12 Week group had Grade 4 AEs. One subject had a Grade 4 AE of malignant lung neoplasm and 1 subject had a Grade 4 AE of sudden death. Both events were assessed by the investigators as unrelated to study drugs.

SAEs were rare and occurred in 15 subjects (2.4%) in the SOF/VEL 12 Week group. All SAEs were assessed by the investigators as unrelated to study drugs. No placebo treated subjects had SAEs. No trends in SAE type or onset time were observed, and no SAE was reported in > 1 subject. No SAEs led to treatment discontinuation. One subject death was reported in the study. This subject completed 12 weeks of treatment with SOF/VEL and died in his sleep on post-treatment Day 8. The death was assessed as not related to study drug by the investigator. One subject (0.2%) in the SOF/VEL 12 Week group discontinued study treatment due to a Grade 3 AE of anxiety and 2 subjects (1.7%) in the Placebo 12 Week group discontinued study treatment due to meeting the prespecified stopping criteria of elevated ALT and/or AST levels > 5 × nadir.

Most laboratory abnormalities were Grade 1 or 2 in severity. Subjects in the SOF/VEL 12 Week group had Grade 3 or 4 chemistry abnormalities of elevated AST (Grade 3; 1 subject [0.2%]), elevated creatine kinase (Grade 3; 2 subjects [0.3%], Grade 4; 2 subjects [0.3%]), hyperglycemia (Grade 3, 15 subjects [2.4%]), and elevated lipase (Grade 3; 14 subjects [2.2%], Grade 4, 2 subjects [0.3%]). Among subjects in the SOF/VEL 12 Week, all Grade 3 or 4 creatinine kinase elevations were transient, all Grade 3 or 4 lipase elevations were asymptomatic and generally transient, and Grade 3 or 4 hyperglycemia occurred in subjects with a medical history of diabetes. The most frequently observed Grade 3 or 4 laboratory abnormalities observed in placebo treated subjects were elevated ALT (Grade 3; 6 subjects [5.2%] and Grade 4; 2 subjects [1.7%]) consistent with ongoing HCV infection.

No notable changes from baseline in vital signs (systolic blood pressure, diastolic blood pressure, or pulse) were observed during the study. No trends in ECG findings suggestive of cardiotoxicity were observed.

#### **Conclusions**

The conclusions from this interim analysis were as follows:

- The study met its primary efficacy endpoint demonstrating that the SVR12 rate of 99.0% (95% CI: 97.9% to 99.6%) in genotype 1, 2, 4, 5, and 6 HCV-infected subjects treated for 12 weeks with SOF/VEL was statistically superior to the pre-specified SVR12 performance goal of 85% (p<0.001).
- High SVR12 rates were achieved across all HCV genotypes and subgroups
  - Among subjects with cirrhosis, the SVR rate was 99.2%
  - Among subjects with prior treatment failure, the SVR rate was 99.5%
  - Among subjects with baseline NS5A RAVs, the SVR12 rate was 99.2%
- Treatment with SOF/VEL for 12 Weeks was generally well tolerated with a safety profile similar to that of placebo treatment. There was a low incidence of SAEs, discontinuations due to AEs and no clinically relevant laboratory abnormalities.

# 1.2.2.1.2. Study GS-US-342-1139 (ASTRAL-2)

# **Study Design**

This ongoing Phase 3, randomized, open-label, multicenter study is assessing the antiviral efficacy, safety, and tolerability of 12 weeks of SOF/VEL treatment compared with 12 weeks of SOF+RBV treatment in subjects with chronic genotype 2 HCV infection. The study was conducted in the United States (US).

Subjects with genotype 2 HCV infection were randomized (1:1) to treatment with SOF/VEL for 12 weeks (SOF/VEL 12 Week group) or SOF+RBV for 12 weeks (SOF+RBV 12 Week group). Randomization was stratified by the presence or absence of cirrhosis at screening and prior treatment experience (treatment naive vs. treatment experienced).

# **Disposition**

A total of 266 subjects were randomized and treated; 134 in the SOF/VEL 12 Week group and 132 in the SOF+RBV 12 Week group. The majority of subjects (99.2%) completed study treatment. Two subjects (0.8%), 1 in each treatment group, prematurely discontinued study treatment. One subject in the SOF/VEL 12 Week group discontinued study treatment on Day 1 (after receiving 1 dose of study drug) due to AEs of disturbance in attention, headache, and anxiety. One subject in the SOF+RBV 12 Week group completed the Week 10 study visit, but did not return for any subsequent study visits and was assumed to be lost to follow-up; the last confirmed dosing date was Day 71.

# **Demographics and Baseline Characteristics**

Overall, demographics and baseline disease characteristics were balanced across both treatment groups. The majority of subjects were male (59.4%), and 32.7% of subjects had a BMI  $\geq 30 \text{ kg/m}^2$ . A total of 38 subjects (14.3%) had cirrhosis at screening. Overall, the majority of subjects had HCV RNA  $\geq 800,000 \text{ IU/mL}$  (79.7%). Overall, 14.7% (39 subjects) were treatment experienced.

#### **Efficacy Results**

The SOF/VEL 12 Week group met the primary endpoint of an SVR12 rate that was noninferior to the SVR12 rate in the SOF+RBV 12 Week group. The SVR12 rates were as follows:

- SOF/VEL 12 Week group: 99.3% (95% CI: 95.9% to 100%) of subjects (133 of 134) achieved SVR12
- SOF+RBV 12 Week group: 93.9% (95% CI: 88.4% to 97.3%) of subjects (124 of 132) achieved SVR12

The strata-adjusted difference (95% CI) in the proportions was 5.2% (0.2% to 10.3%). Since the lower bound of the 2-sided 95% CI for the difference between groups was greater than the

prespecified noninferiority margin of -10%, the efficacy of SOF/VEL for 12 weeks was demonstrated to be statistically noninferior to SOF+RBV for 12 weeks. There was sufficient evidence to demonstrate the statistical superiority of treatment with SOF/VEL for 12 weeks over SOF+RBV for 12 weeks for SVR12 (p = 0.018; CMH test stratified by cirrhosis status and prior treatment experience).

In the SOF/VEL 12 Week group, 1 of 134 subjects (0.7%) did not achieve SVR12: the subject discontinued study treatment on Day 1 (after receiving 1 dose) due to AEs of difficulty concentrating, headache, and anxiety. The subject never achieved HCV RNA < LLOQ. In the SOF+RBV 12 Week group, 8 of 132 subjects (6.1%) did not achieve SVR12. Of these, 6 subjects relapsed and 2 were lost to follow-up. Four relapses occurred by the post-treatment Week 4 visit and 2 relapses occurred between the post-treatment Week 4 and 12 visits. The low number of virologic failures in the study precluded meaningful subgroup analysis of SVR.

The SVR4 results were similar to the SVR12 results with the exception of 3 subjects in SOF+RBV 12 Week group: 1 subject was lost to follow-up after post-treatment Week 4 and 2 subjects relapsed between the post-treatment Week 4 and Week 12 visits.

HCV RNA levels (log<sub>10</sub> IU/mL) declined rapidly with similar decreases in HCV RNA observed in both treatment groups. After 1 week of treatment, the mean change from baseline in HCV RNA levels was –4.51 log<sub>10</sub> IU/mL in both treatment groups. The decreases in HCV RNA were maintained from Weeks 2 through 12. Consistent with the rapid and sustained decline in HCV RNA, 90.2% of subjects in both treatment groups had HCV RNA < LLOQ at Week 4. There was a lack of correlation of time to suppression with virologic outcome in the SOF/VEL 12 week group as all subjects who completed treatment achieved SVR regardless of the time to suppression.

#### Virologic Resistance

Deep sequencing analyses indicated that genotype 2a and 2b were the predominant HCV subtypes in subjects who were randomized and treated in this study. Approximately 60% and 10% of subjects in the SOF/VEL 12 Week group had pretreatment NS5A and NS5B RAVs, respectively. The most prevalent NS5A RAV observed was L31M in 51% of subjects. Despite the presence of pretreatment NS5A and NS5B RAVs, no subjects in the SOF/VEL 12 Week group experienced virologic failure in this study. Two of the 6 subjects who relapsed in the SOF+RBV 12 Week group had low levels of the NS5B NI RAV L159F detectable at failure.

#### **Safety Results**

Overall, treatment with SOF/VEL or SOF+RBV for 12 weeks was generally safe and well tolerated. A smaller percentage of subjects in the SOF/VEL 12 Week group experienced any AE (68.7%, 92 of 134) compared with the SOF+RBV 12 Week group (76.5%, 101 of 132), including treatment-related AEs (SOF/VEL, 33.6%; SOF+RBV, 56.8%) and AEs leading to modification or interruption of any study drug (SOF/VEL, 0; SOF+RBV, 9.8%).

The most common AEs (ie, AEs reported in > 10% of subjects in either group) were reported by a smaller percentage of subjects in the SOF/VEL 12 Week group compared with the SOF+RBV 12 Week group, including fatigue (14.9% vs 35.6%), headache (17.9% vs 22.0%), nausea (10.4% vs 14.4%), and insomnia (4.5% vs 13.6%).

Most AEs were Grade 1 (mild) or Grade 2 (moderate) in severity. Grade 3 (severe) AEs were rare (SOF/VEL, 2.2%; SOF+RBV, 2.3%). No Grade 4 (life-threatening) AEs were reported. Anxiety was the only Grade 3 AE reported in > 1 subject in the SOF/VEL 12 Week group (n = 2, 1.5%).

Serious adverse events (SAEs) were also rare (1.5%, 4 of 266 subjects [2 in each treatment group]). No SAE was reported in > 1 subject. All SAEs were considered by the investigators to be not related to study drug. Two non-treatment-emergent deaths were reported during the study (metastatic lung cancer and cardiac arrest after treatment completion). No pregnancies were reported during the study. Only 1 subject permanently discontinued any study drug (SOF/VEL) due to AEs. After receiving 1 dose of SOF/VEL, the subject, who had a medical history of depression, insomnia and post-traumatic stress disorder, discontinued study treatment due to Grade 3 AEs of difficulty concentrating, headache, and anxiety that were assessed as related to study drugs by the investigator.

Most subjects had at least 1 laboratory abnormality reported, with the majority being Grade 1 (104 of 266 subjects, 39.1%) or Grade 2 (70 of 266 subjects, 26.3%) in severity. A smaller percentage of subjects had Grade 3 laboratory abnormalities in the SOF/VEL 12 Week group (7.5%, 10 subjects) compared with the SOF+RBV 12 Week group (13.6%, 18 subjects). This difference was accounted for primarily by the expected decreases in hemoglobin observed with RBV therapy. No subjects in the SOF/VEL 12 Week group had a Grade 3 or 4 hematology laboratory abnormality. The only Grade 3 hematology laboratories abnormality in the SOF+RBV 12 Week group were decreased hemoglobin (5.3%, 7 subjects) and increased lymphocytes (0.8%, 1 subject). The most common Grade 3 or 4 chemistry laboratory abnormalities in both treatment groups were increased serum glucose (hyperglycemia) and increased lipase. Grade 3 increases in lipase were reported for 7 subjects (5.3%) in the SOF/VEL 12 Week group and 2 subjects (1.5%) in the SOF+RBV 12 Week group. Grade 4 increases in lipase were reported for 1 subject (0.8%) in each treatment group. All of the Grade 3 lipase elevations were transient and asymptomatic, with no cases of clinical pancreatitis. In the SOF/VEL 12 Week group, 1 subject each experienced a Grade 3 or 4 increase in creatine kinase following workout sessions. Grade 3 hyperbilirubinemia was only observed in the SOF+RBV 12 Week group and was consistent with RBV-associated hemolysis. Grade 4 chemistry laboratory abnormalities were reported for lipase and creatine kinase.

No notable changes in vital signs (systolic blood pressure, diastolic blood pressure, and pulse) or ECGs were reported during the study.

#### **Conclusions**

The conclusions from this interim analysis were as follows:

• The study met its predefined primary efficacy endpoint, demonstrating that the SVR12 rate of 99.3% with SOF/VEL for 12 weeks was noninferior to the SVR12 rates of 93.9% with SOF+RBV for 12 weeks.

- Treatment with SOF/VEL for 12 weeks led to a statistically superior SVR12 rate compared with SOF+RBV for 12 weeks (p = 0.018).
- No subjects treated with SOF/VEL experienced virologic failure, including subjects with cirrhosis (14%), prior treatment failure (14%), and baseline NS5A RAVs (60%).
- SOF/VEL was generally well tolerated and, compared with SOF+RBV, lacked toxicities associated with RBV. No treatment-emergent deaths, Grade 4 AEs, treatment-related SAEs, or clinically relevant laboratory abnormalities were observed.

1.2.2.1.3. Study GS-US-342-1140 (ASTRAL-3)

#### **Study Design**

This ongoing, Phase 3, randomized, open-label, multicenter study is assessing the antiviral efficacy, safety, and tolerability of 12 weeks of SOF/VEL treatment compared with 24 weeks of SOF+RBV treatment in subjects with chronic genotype 3 HCV infection. This study was conducted in Australia, Canada, France, Germany, Italy, New Zealand, United Kingdom, and United States.

Subjects with genotype 3 HCV infection were randomized (1:1) to treatment with SOF/VEL for 12 weeks (SOF/VEL 12 Week group) or SOF+RBV for 24 weeks (SOF+RBV 24 Week group). Randomization was stratified by the presence or absence of cirrhosis at screening and prior treatment experience (treatment naive vs treatment-experienced).

# **Disposition**

A total of 552 subjects were randomized and treated (277 subjects in the SOF/VEL 12 Week group and 275 subjects in the SOF+RBV24 Week group). A total of 21 subjects (7.6%) in the SOF+RBV 24 Week group discontinued treatment compared with 2 subjects (0.7%) in the SOF/VEL 12 Week group. The most common reason for discontinuation of treatment for subjects in the SOF+RBV 24 Week group was AEs (9 subjects, 3.3%).

#### **Demographics and Baseline Characteristics**

The majority of subjects were male (62.3%), and 20.3% of subjects had a BMI  $\geq$  30 kg/m<sup>2</sup>. Overall, the majority of subjects had HCV RNA  $\geq$  800,000 IU/mL (69.7%). A total of 163 subjects (29.5%) had cirrhosis at screening. Overall, 25.7% (142 subjects) were treatment experienced.

#### **Efficacy Results**

The study met the primary efficacy endpoint. The SVR12 rate for the SOF/VEL 12 Week group was statistically noninferior to the SVR12 rate for the SOF+RBV 24 Week group. The SVR12 rates were as follows:

- SOF/VEL 12 Week group: 95.3% (95% CI: 92.1% to 97.5%) of subjects (264 of 277) achieved SVR12.
- SOF+RBV 24 Week group: 80.4% (95% CI: 75.2% to 84.9%) of subjects (221 of 275) achieved SVR12.

The strata-adjusted difference (95% CI) in the proportions was 14.8% (9.6% to 20.0%). The superiority of treatment with SOF/VEL for 12 weeks over SOF+RBV for 24 weeks for SVR12 was also demonstrated (p < 0.001; CMH test stratified by cirrhosis status and prior treatment experience).

In the SOF/VEL 12 Week group, 13 of 277 subjects (4.7%) did not achieve SVR12. Of these, no subjects had on-treatment virologic failure, 11 subjects relapsed, and 2 subjects were lost to follow-up. In the SOF+RBV 24 Week group, 54 of 275 subjects (19.6%) did not achieve SVR12. Of these, 1 subject had on-treatment virologic failure (nonresponse), 38 subjects relapsed, and 15 subjects did not achieve SVR12 for reasons other than virologic failure. These 15 subjects included 6 subjects who were lost to follow-up or who did not attend a post-treatment Week 12 visit, 4 subjects who withdrew from the study due to AEs, 2 subjects who withdrew consent from the study, 2 subjects who died, and 1 subject who only received 2 days of study drug, did not achieve HCV RNA < LLOQ on treatment, and did not meet the protocol definition for virologic failure.

Most relapses occurred by the post-treatment Week 4 visit. In the SOF/VEL 12 Week group, 8 of 11 relapses occurred by post-treatment Week 4, and 3 of 11 relapses occurred between post-treatment Weeks 4 and 12.

Across the 2 treatment groups, the SVR12 rates consistently favored the SOF/VEL 12 Week group over the SOF+RBV 24 Week group. Within each treatment group, the SVR12 rates for most subgroups were generally consistent with those observed in the overall population. In the SOF/VEL 12 Week group, the SVR12 rates for subjects with and without cirrhosis were 91.3% (73 of 80) and 97.0% (191 of 197), respectively, and the SVR12 rates for treatment-naive and treatment-experienced subjects were 97.1% (200 of 206) and 90.1% (64 of 71), respectively. In the SOF+RBV 24 Week group, subjects with cirrhosis had considerably lower SVR12 rates (66.3%; 55 of 83) than subjects without cirrhosis (87.2%; 163 of 187), and subjects with prior treatment experience had considerably lower SVR12 rates (63.4%; 45 of 71) than treatment-naive subjects (86.3%; 176 of 204).

HCV RNA levels ( $\log_{10}$  IU/mL) declined rapidly, with similar decreases in HCV RNA observed in both treatment groups. Consistent with the rapid and sustained decline in HCV RNA, 91.7% of subjects in the SOF/VEL 12 Week group and 88.2% of subjects in the SOF+RBV 24 Week group had HCV RNA < LLOQ at Week 4. Time to virologic suppression did not impact virologic outcomes in the SOV/VEL 12 Week group: SVR12 rates were 96.0% and 95.7% among those subjects with HCV RNA < LLOQ and those with HCV RNA  $\geq$  LLOQ at Week 4, respectively.

# **Virologic Resistance**

Pretreatment NS5A and NS5B NI RAVs were present in 16% and 4% of subjects, respectively, in the SOF/VEL 12 Week group. There was a numerically lower SVR12 rate in SOF/VEL-treated subjects with baseline NS5A RAVs compared with subjects without NS5A RAVs (88% vs 97%, respectively). All subjects with NS5B NI RAVs in the SOF/VEL 12 Week group achieved SVR12.

A total of 10 subjects in the SOF/VEL 12 Week group relapsed, and 1 subject was reinfected. All 10 subjects had the NS5A RAV Y93H detected at relapse time points. No SOF/VEL-treated subjects had NS5B NI RAVs emerge at relapse. The NS5B NI RAVs (N142T, L159F, or V321A) emerged in 7 of 39 subjects in the SOF+RBV 24 Week group who had virologic failure.

#### **Safety Results**

Overall, treatment with SOF/VEL for 12 weeks or SOF+RBV for 24 weeks was generally safe and well tolerated. A lower percentage of subjects in the SOF/VEL 12 Week group experienced any AE (88.4%; 245 of 277) compared with the SOF+RBV 24 Week group (94.5%; 260 of 275).

Most AEs were Grade 1 (mild) or Grade 2 (moderate) in severity. Grade 3 (severe) AEs were reported for 4.3% (12 subjects) in the SOF/VEL 12 Week group and 7.3% (20 subjects) in the SOF+RBV 24 Week group. Grade 4 (life-threatening) AEs were reported for no subjects in the SOF/VEL 12 Week group and 1.1% (3 subjects) in the SOF+RBV 24 Week group (death due to natural causes in 1 subject, cerebrovascular accident in 1 subject, and multiple gunshot wounds in 1 subject).

Of the most common AEs (ie, AEs reported in  $\geq$  10% of subjects in either treatment group), a lower percentage of subjects in the SOF/VEL 12 Week group compared with the SOF+RBV 24 Week group experienced fatigue (25.6% vs 38.2%), insomnia (11.2% vs 26.9%), nausea (16.6% vs 21.1%), irritability (8.3% vs 14.5%), cough (5.1% vs 12.7%), pruritus (2.9% vs 12.7%), and dyspepsia (3.2% vs 10.9%).

Serious adverse events were reported for 2.2% (6 subjects) in the SOF/VEL 12 Week group and 5.5% (15 subjects) in the SOF+RBV 24 Week group. No SAE was reported in > 1 subject, and no SOV/VEL-treated subject had a treatment-related SAE. Three subject deaths were reported during the study (1 treatment-emergent death due to natural causes, 1 treatment-emergent death due to multiple gunshot wounds, and 1 nontreatment-emergent death due to an unknown cause); all 3 subjects were in the SOF+RBV 24 Week group. A total of 9 subjects (in the SOF+RBV 24 Week group) prematurely discontinued study drugs due to an AE. The most common AE resulting in discontinuation of study drug in the SOF+RBV 24 Week group was insomnia (1.1%, 3 subjects).

Most subjects had at least 1 laboratory abnormality reported, with the majority being Grade 1 (36.3%; 200 of 551 subjects) or Grade 2 (29.6%; 163 of 551 subjects) in severity. A lower percentage of subjects had Grade 3 laboratory abnormalities in the SOF/VEL 12 Week group (5.8%, 16 of 276) compared with the SOF+RBV 24 Week group (14.2%, 39 of 275). This difference was accounted for primarily by the expected decreases in hemoglobin observed during treatment with RBV. Grade 4 laboratory abnormalities were similarly low in the SOF/VEL 12 Week group (1.4%, 4 of 276) compared with the SOF+RBV 24 Week group (2.9%, 8 of 275).

The only Grade 3 or 4 hematology laboratory abnormality in the SOF/VEL 12 Week group occurring in more than 1 subject was decreased lymphocytes (1.1%, 3 of 276 subjects). One subject had normal lymphocytes throughout treatment and a Grade 3 decrease at the post-treatment Week 4 visit. The other 2 subjects had Grade 2 or 3 decreased lymphocytes at baseline that transiently decreased by 1 grade during treatment.

The most common Grade 3 or 4 chemistry laboratory abnormalities in both treatment groups were increased lipase, increased serum glucose (hyperglycemia), and increased creatine kinase. Grade 3 or 4 increases in lipase were reported for 9 subjects (3.3%) in the SOF/VEL 12 Week group and 5 subjects (1.8%) in the SOF+RBV 24 Week group. All of the Grade 3 or 4 increases in lipase were asymptomatic, with no cases of clinical pancreatitis. Grade 3 increases in serum glucose (hyperglycemia) were reported for 4 subjects (1.4%) in the SOF/VEL 12 Week group and 5 subjects (1.8%) in the SOF+RBV 24 Week group. All subjects with Grade 3 increased serum glucose had either a medical history of diabetes or HbA $_{1c} \ge 6.0\%$  at screening. Grade 3 or 4 increases in creatine kinase were reported for 2 subjects (0.7%) in the SOF/VEL 12 Week group and 4 subjects (1.5%) in the SOF+RBV 24 Week group. All of the Grade 3 or 4 creatine kinase elevations were transient and asymptomatic; the majority were associated with exercise. Grade 3 or 4 increases in total bilirubin (hyperbilirubinemia) were observed only in the SOF+RBV 24 Week group (Grade 3: 2 subjects, 0.7%; Grade 4: 1 subject, 0.4%). The timing and magnitude of the increases in total bilirubin were consistent with RBV-induced hemolysis.

No notable changes in vital signs (systolic blood pressure, diastolic blood pressure, and pulse) were reported during the study.

#### **Conclusions**

The conclusions from this interim analysis were as follows:

- The study met its predefined primary efficacy endpoint: subjects with genotype 3 HCV infection in the SOF/VEL 12 Week group achieved an SVR12 rate of 95.3% that was statistically noninferior to the SVR12 rate of 80.4% achieved by subjects with genotype 3 HCV infection in the SOF+RBV 24 Week group.
  - The superiority of treatment with SOF/VEL for 12 weeks over SOF+RBV for 24 weeks for SVR12 was also demonstrated (p < 0.001).
- Across the 2 treatment groups, the SVR12 rates consistently favored the SOF/VEL 12 Week group over the SOF+RBV 24 Week group.
  - For subjects with cirrhosis, the SVR12 rates (SOF/VEL 12 Weeks vs SOF+RBV 24 Weeks) were 91.3% and 66.3%, respectively.
  - For treatment-experienced subjects, the SVR12 rates (SOF/VEL 12 Weeks vs SOF+RBV 24 Weeks) were 90.1% and 63.4%, respectively.
- Among the 16% of SOF/VEL-treated subjects with baseline NS5A RAVs, the SVR12 rate was numerically lower (88%) compared with subjects without baseline NS5A RAVs (SVR12 rate of 97%).
- SOF/VEL was generally well tolerated and, compared with SOF+RBV, lacked toxicities
  associated with RBV. No treatment-emergent deaths, Grade 4 AEs, treatment-related SAEs,
  discontinuations due to AEs, or clinically relevant laboratory abnormalities were observed in
  SOF/VEL-treated subjects.

# 1.2.2.1.4. Study GS-US-342-1137 (ASTRAL-4)

# **Study Design**

This ongoing, Phase 3, randomized, open-label, multicenter study is assessing the antiviral efficacy, safety, and tolerability of SOF/VEL±RBV for 12 weeks and SOF/VEL for 24 weeks in subjects with chronic HCV infection and Child-Pugh-Turcotte (CPT) class B cirrhosis. The study was conducted in the US.

Subjects with genotype 1 to 6 HCV infection with CPT class B cirrhosis were randomized (1:1:1) to SOF/VEL for 12 weeks (SOF/VEL 12 Week group), SOF/VEL+RBV for 12 weeks (SOF/VEL+RBV 12 Week group), or SOF/VEL for 24 weeks (SOF/VEL 24 Week group). Randomization was stratified by HCV genotype (1, 2, 3, 4, 5, 6, and indeterminate).

# **Disposition**

A total of 267 subjects were included in the Safety and Full Analysis Sets (90 subjects in the SOF/VEL 12 Week group, 87 subjects in the SOF/VEL+RBV 12 Week group, and 90 subjects in the SOF/VEL 24 Week group).

Of the 90 subjects in the SOF/VEL 12 Week group, 89 subjects (98.9%) completed study drug and 1 subject (1.1%) discontinued due to an AE.

Of the 87 subjects in the SOF/VEL+RBV 12 Week group, 82 subjects (94.3%) completed study drug; 4 subjects (4.6%) discontinued due to AEs and 1 subject (1.1%) discontinued due to virologic failure (pharmacokinetic [PK] data for this subject indicated noncompliance with study drugs).

Of the 90 subjects in the SOF/VEL 24 Week group, 84 subjects (93.3%) completed study drug; 4 subjects (4.4%) discontinued due to AEs, 1 subject (1.1%) discontinued due to virologic failure, and 1 subject (1.1%) discontinued due to noncompliance with study drug.

#### **Demographics and Baseline Characteristics**

Overall, demographics and baseline disease characteristics were balanced across the treatment groups. Of the 267 subjects randomized and treated, 207 subjects (77.5%) had genotype 1 HCV infection, 12 subjects (4.5%) had genotype 2 HCV infection, 39 subjects (14.6%) had genotype 3 HCV infection, 8 subjects (3.0%) had genotype 4 HCV infection, and 1 subject (0.4%) in the SOF/VEL 24 Week group had genotype 6 HCV infection. The majority of subjects were male (69.7%), and 42.3% of subjects had a BMI  $\geq$  30 kg/m<sup>2</sup>. Most subjects (55.1%) had prior treatment experience and the majority of subjects had HCV RNA  $\geq$  800,000 IU/mL (55.8%).

#### **Efficacy Results**

The SVR12 rates were as follows:

- SOF/VEL 12 Week group: 83.3% (95% CI: 74.0% to 90.4%) of subjects (75 of 90) achieved SVR12
- SOF/VEL+RBV 12 Week group: 94.3% (95% CI: 87.1% to 98.1%) of subjects (82 of 87) achieved SVR12
- SOF/VEL 24 Week group: 85.6% (95% CI: 76.6% to 92.1%) of subjects (77 of 90) achieved SVR12

All 3 treatment groups met their primary efficacy endpoints with SVR12 rates that were statistically superior compared with the assumed spontaneous rate of 1%. The p-value was < 0.001 for the comparison with the SVR12 for each treatment group.

Among subjects with genotype 1 HCV infection, the SVR12 rate was higher for those in the SOF/VEL+RBV 12 Week group (95.6%, 65 of 68) compared with the SOF/VEL 12 Week group (88.2%, 60 of 68) or the SOF/VEL 24 Week group (91.5%, 65 of 71). Similarly, among subjects with genotype 3 HCV infection, the SVR12 rate was higher for those in the SOF/VEL+RBV 12 Week group (84.6%, 11 of 13) compared with the SOF/VEL 12 Week group (50.0%, 7 of 14) or the SOF/VEL 24 Week group (50.0%, 6 of 12).

All subjects with genotype 2, 4, or 6 HCV infection achieved SVR12 across all treatment groups with the exception of 1 subject with genotype 2 HCV infection in the SOF/VEL 24 Week group who died 39 days after completing 28 days of treatment.

Most virologic failures were due to relapse. One subject with genotype 3 HCV infection in the SOF/VEL+RBV 12 Week group had on-treatment breakthrough with PK data showing undetectable plasma drug levels consistent with non-adherence to study drug and 1 subject with genotype 3 HCV infection in the SOF/VEL 24 Week group had on-treatment breakthrough.

There was 1 subject (1.5%) with genotype 1 HCV infection with virologic failure in the SOF/VEL+RBV 12 Week group compared with 5 subjects (7.4%) in the SOF/VEL 12 Week group and 3 subjects (4.2%) in the SOF/VEL 24 Week group. Among subjects with genotype 3 HCV infection, the lowest rate of virologic failure was observed in the SOF/VEL+RBV 12 Week group with 2 failures (15.4%) compared with 6 (42.9%) in the SOF/VEL 12 Week group and 5 (41.7%) in the SOF/VEL 24 Week group.

There were no virologic failures in subjects with genotype 2, 4, or 6 HCV infection in any of the treatment groups.

Treatment with SOF/VEL+RBV for 12 weeks resulted in high SVR12 rates irrespective of genotype, prior treatment history, baseline HCV RNA, and presence of pretreatment NS5A or

NS5B RAVs. Furthermore, there was no impact of demographic factors such as age, sex, BMI, or IL28B genotype on treatment outcome in the SOF/VEL+RBV 12 Week group.

Overall, 108 subjects (47.2%) had an improvement in CPT score (range: 1–5 points) while 99 subjects (43.2%) had no change. A minority of subjects (9.6%, 22 subjects) experienced an increase (worsening) in CPT score from baseline to post-treatment Week 12. A higher percentage of subjects receiving SOF/VEL for 24 weeks (54.7%) compared with subjects receiving SOF/VEL±RBV for 12 weeks (40.7%–46.6%) had improvements in CPT score from baseline to post-treatment Week 12; this difference likely reflects the longer time of observation with HCV RNA suppression. The improvements in CPT score were largely due to improvements in bilirubin and albumin.

Overall, the majority of subjects who achieved SVR12 also had a decrease (improvement) (55.5%, 127 of 229 subjects) in MELD score between baseline and post-treatment Week 12 (range: 1-11 points). Among subjects who had MELD score < 15 at baseline and achieved SVR12, 197 of 203 subjects (97.0%) remained < 15 at post-treatment Week 12. A total of 16 subjects (61.5%) with baseline MELD score  $\geq$  15 who achieved SVR12 improved to < 15. Improvements in MELD score were largely due to improvements in total bilirubin.

# Virologic Resistance

Pretreatment NS5A RAVs were observed in 26% to 29% of subjects across the treatment groups. The presence of pretreatment NS5A RAVs did not impact treatment outcome in the SOF/VEL+RBV 12 Week group. Slightly lower SVR rates were observed in subjects with genotype 1 HCV infection with NS5A RAVs treated with SOF/VEL for 12 or 24 weeks compared to subjects without pretreatment NS5A RAVs. No virologic failures were observed in subjects with genotype 2, 4, or 6 HCV infection. The small numbers of subjects with genotype 3 HCV infection with pretreatment NS5A RAVs precluded meaningful subgroup analysis. The presence of pretreatment NS5B RAVs did not impact treatment outcome in any treatment group.

The majority of subjects had NS5A RAVs present at virologic failure with Y93H being the most common variant. NS5B NI RAVs were less common and typically observed at low levels. Of the 9 subjects with genotype 1 HCV infection with virologic failure, 6 had NS5A RAVs at failure (5 treatment emergent and 1 maintained from pretreatment). Two genotype 1 HCV-infected subjects had L159F and S282T NS5B NI RAVs present at failure; both of these subjects had multiple NS5A RAVs at pretreatment that reduce susceptibility to VEL. All 13 subjects with genotype 3 HCV infection with virologic failure had Y93H at failure (10 were treatment emergent). Three genotype 3 HCV-infected subjects had low levels of NS5B NI RAVs emerge at virologic failure.

#### **Safety Results**

Overall, treatment with SOF/VEL±RBV for 12 weeks or SOF/VEL for 24 weeks was generally safe and well tolerated. Adverse events were consistent with the expected clinical sequelae in the setting of decompensated cirrhosis and, in addition, with the known toxicities of RBV in the SOF/VEL+RBV 12 Week group.

A smaller percentage of subjects in the SOF/VEL 12 Week and SOF/VEL 24 Week groups experienced any AE (81.1% in each group) compared with the SOF/VEL+RBV 12 Week group (90.8%). The higher frequency of AEs observed in the SOF/VEL+RBV 12 Week group was primarily due to AEs consistent with RBV-associated toxicity. No treatment-related Grade 3 AEs were reported in > 1 subject in any group or overall.

Most AEs were Grade 1 (mild) or Grade 2 (moderate) in severity. Overall, the most commonly reported Grade 3 or 4 AEs were hepatic encephalopathy and sepsis (5 subjects each), which are consistent with the natural history of disease progression in a population with decompensated liver disease.

Serious adverse events (SAEs) occurred in 17.6% of subjects in similar proportions across treatment groups, and only 1 subject (0.4%) experienced SAEs considered related to SOF/VEL. The most commonly reported SAEs were hepatic encephalopathy and sepsis (5 subjects each). Nine deaths occurred during the study, 2 of which were treatment emergent, and none of which was assessed as related to study drugs. One subject in the SOF/VEL 24 Week group underwent a liver transplantation on post-treatment Day 8 after completing 35 days of treatment.

Nine subjects discontinued all study drugs due to an AE (SOF/VEL 12 Week group: 1.1%, 1 subject; SOF/VEL+RBV 12 Week group: 4.6%, 4 subjects; SOF/VEL 24 Week group: 4.4%, 4 subjects). No AE leading to discontinuation of study drugs was reported in > 1 subject. A total of 31.0% (27 of 87) of subjects had modified or interrupted RBV dosing due to AEs, and 10.3% (9 of 87) of subjects permanently discontinued RBV due to AEs while continuing SOF/VEL.

The majority of subjects had at least 1 Grade 3 or 4 laboratory abnormality (42.7% and 12.4%, respectively) with the highest rates observed in the SOF/VEL+RBV group (Grade 3: 43.7%; Grade 4 18.4%) due to a higher rate of hematologic abnormalities. The most commonly observed Grade 3 or 4 hematology laboratory abnormalities were decreased lymphocytes, hemoglobin, and platelet counts, all of which are a known effect of RBV therapy or expected in a subject population with decompensated liver disease.

The most commonly observed Grade 3 or 4 chemistry laboratory abnormalities were increased glucose and increased total bilirubin. All of the Grade 3 or 4 increased glucose abnormalities occurred in subjects with a history of diabetes mellitus or had elevated glucose at baseline or continuing through the post-treatment period. The majority of subjects with Grade 3 or 4 increased total bilirubin (71.7%, 22 of 31 subjects) were in the SOF/VEL+RBV 12 Week group, primarily in a pattern that was consistent with RBV-induced hemolysis.

No notable changes in vital signs (systolic blood pressure, diastolic blood pressure, and pulse) were reported during the study. No trends in electrocardiogram findings suggestive of cardiotoxicity were observed.

#### **Conclusions**

The conclusions from this interim analysis were as follows:

- Treatment with SOF/VEL±RBV for 12 or 24 weeks in subjects with decompensated cirrhosis resulted in high SVR12 rates:
  - In the SOF/VEL 12 Week group, the SVR12 rate was 83.3% (75 of 90 subjects).
  - In the SOF/VEL+RBV 12 Week group, the SVR12 rate was 94.3% (82 of 87 subjects).
  - In the SOF/VEL 24 Week group, the SVR12 rate was 87.8% (79 of 90 subjects).
- The SVR12 rates were highest in subjects treated with SOF/VEL+RBV for 12 weeks with few virologic failures:
  - In subjects with genotype 1 HCV infection, the virologic failure rate was 1.5% (1 of 68 subjects).
  - In subjects with genotype 3 HCV infection, the virologic failure rate was 15.4%
     (2 of 13 subjects), of which 1 subject had on-treatment breakthrough with PK data showing undetectable plasma drug levels consistent with non-adherence to study drug.

Overall, there were no virologic failures in subjects with genotype 2, 4, or 6 HCV infection.

- The SVR12 rates between the SOF/VEL 12- and 24-week treatment durations were similar across all genotypes.
- The presence of pretreatment NS5A and NS5B RAVs did not impact treatment outcome with SOF/VEL+RBV for 12 weeks.
- Approximately half of subjects who achieved SVR12 experienced an early improvement in CPT and MELD scores, primarily related to improvements in synthetic function (albumin) and decreases in bilirubin.
- SOF/VEL was generally well tolerated in these subjects with decompensated liver disease, as evidenced by low rates of study treatment discontinuation and the majority of Grade 3 and 4 AEs, SAEs, and laboratory abnormalities being consistent with clinical sequelae of advanced liver disease and RBV toxicity.
- 1.2.2.1.5. Study GS-US-342-1202 (ASTRAL-5)

#### **Study Design**

This ongoing, Phase 3, open-label, multicenter study is assessing the antiviral efficacy, safety, and tolerability of SOF/VEL for 12 weeks in subjects with chronic HCV infection and HIV-1 coinfection. This study is being conducted in the US, New Zealand, and Australia.

Approximately 100 subjects with genotype 1 to 6 HCV infection with HIV-1 coinfection on a stable regiment of HIV antiretroviral therapy (ARV) are all scheduled to receive SOF/VEL for 12 weeks. The primary outcome is the proportion of subjects who achieve SVR 12.

# 1.2.2.1.6. Study GS-US-342-1553

# **Study Design**

This ongoing, open-label, multicenter study is assessing the antiviral efficacy, safety, and tolerability of SOF/VEL±RBV for 24 weeks in subjects with chronic HCV infection who have participated in prior Gilead sponsored HCV treatment studies. This study is being conducted in the US, New Zealand, and Australia.

Approximately 150 subjects with and without cirrhosis with genotype 1 to 6 HCV infection who did not achieve SVR 12 in previous Gilead sponsored HCV treatment studies will all receive SOF/VEL + RBV for 24 weeks). The primary outcome is the proportion of subjects who achieve SVR 12.

# 1.2.2.1.7. Study GS-US-342-1446

#### **Study Design**

This ongoing, open-label, multicenter study is assessing the antiviral efficacy, safety, and tolerability of SOF/VEL for 12 weeks in subjects who received placebo in study GS-US-342-1138 (ASTRAL 1). This study is being conducted in the US, Canada, Europe, and Asia.

Approximately 100 subjects with genotype 1, 2, 4, 5, and 6 HCV infection who received placebo in ASTRAL 1 will all receive SOF/VEL 12 weeks. The primary outcome is the proportion of subjects who achieve SVR 12.

# 1.2.2.2. Clinical Pharmacology Studies

#### 1.2.2.2.1. Study GS-US-281-1058

GS-US-281-1058 is an open-label, Phase 1, multiple-dose drug-drug interaction (DDI) study in healthy female subjects of childbearing age evaluating the effect of VEL on the pharmacokinetics of a representative hormonal oral contraceptive medication, norgestimate/ethinyl estradiol (NGM/EE, OC). Following screening, eligible subjects were enrolled in a lead-in period (Part A) of 28 days during which they completed dosing with the hormonal oral contraceptive (OC) prior to baseline assessments and initiation of Cycle 1 (Part B). Subjects with a documented history of taking OC for at least 1 menstrual cycle could be enrolled directly into Cycle 1. The PK, safety, and tolerability of OC and OC + VEL were assessed in Part B of the study, which consisted of 2 cycles: subjects received OC alone during Cycle 1, and OC plus VEL 100 mg once daily during days 8-14 of Cycle 2. Fifteen subjects were

enrolled, and 13 completed the study. Two subjects were discontinued from the study prior to initiation of Cycle 2 (OC+VEL) for laboratory abnormalities.

Table 1-2 presents the steady-state PK parameters and statistical comparisons of NGM metabolites norelgestromin (NGMN) and norgestrel (NG) and EE following administration alone or in combination with VEL. Steady-state VEL PK parameters were also assessed. Norgestimate was not quantifiable for all subjects at most time points. Similar systemic exposure of NGMN and NG were achieved following NGM/EE administration with VEL relative to administration of NGM/EE alone. A modest increase in EE C<sub>max</sub> was observed when administered with VEL with no change in overall exposure (AUC) or C<sub>tau</sub>. The magnitude of increase in EE C<sub>max</sub> when administered with VEL is similar to that observed with the concomitant administration of other drugs such as voriconazole and etravirine, which did not warrant dose adjustment {Andrews et al 2008, Janssen Pharmaceuticals Inc. 2013}. VEL exposures were consistent with historical data (Studies GS-US-281-0115, GS-US-342-0104).

Table 1-2. NGMN, NG, EE, and VEL Plasma PK Parameters Following Administration of NGM/EE alone or with VEL

| | Mean ( | GLSM Ratio | |
|---|---|---|---|
| PK Parameter | NGM/EE Alone<br>(N = 15) | NGM/EE + VEL<br>(N = 13) | (90% CI) NGM/EE + VEI<br>vs. NGM/EE |
| Norelgestromin | | | |
| AUC <sub>tau</sub> (pg•h/mL) | 17,700 (16.7) | 15,700 (11.2) | 0.90 (0.82, 0.98) |
| C <sub>max</sub> (pg/mL) | 1650 (16.8) | 1600 (13.7) | 0.97 (0.88, 1.07) |
| C <sub>tau</sub> (pg/mL) | 454 (18.5) | 416 (14.3) | 0.92 (0.83, 1.03) |
| Norgestrel | | • | · |
| AUC <sub>tau</sub> (pg•h/mL) | 47,000 (34.4) | 43,000 (32.4) | 0.91 (0.73, 1.15) |
| C <sub>max</sub> (pg/mL) | 2410 (30.6) | 2330 (31.5) | 0.96 (0.78, 1.19) |
| C <sub>tau</sub> (pg/mL) | 1760 (34.4) | 1640 (35.7) | 0.92 (0.73, 1.18) |
| Ethinyl Estradiol | | • | |
| AUC <sub>tau</sub> (pg•h/mL) | 666 (30.7) | 686 (27.3) <sup>a</sup> | 1.04 (0.87, 1.24) |
| C <sub>max</sub> (pg/mL) | 57.5 (27.3) | 80.0 (28.4) <sup>a</sup> | 1.39 (1.17, 1.66) |
| C <sub>tau</sub> (pg/mL) | 14.8 (39.3) | 12.4 (43.9) <sup>a</sup> | 0.83 (0.65, 1.06) |
| Velpatasvir | | • | |
| AUC <sub>tau</sub> (ng•h/mL) | | 4680 (35.1) | |
| C <sub>max</sub> (ng/mL) | | 626 (22.0) | |
| C <sub>tau</sub> (ng/mL) | | 68.3 (47.6) | |

Note: preliminary data presented to 3 significant figures.

a N = 12

Luteinizing hormone (LH), follicle stimulating hormone (FSH), and progesterone concentrations were similar in both treatment cycles, as presented in Table 1-3. Luteinizing hormone and progesterone median values were lower than those expected for ovulatory or luteal phases, respectively {Barditch-Crovo et al 1999, Quest Diagnostics 2013a, Quest Diagnostics 2013b}. Follicle stimulating hormone was lower or within the expected range for the ovulatory phase {Quest Diagnostics 2013a}. These results are consistent with a possible decrease in serum LH and FSH by hormonal contraceptives and absence of ovulation, as assessed by very low progesterone values on cycle Day 21.

Table 1-3. Summary of LH, FSH, and Progesterone Concentrations Following Administration of NGM/EE alone or with VEL

| | Median (Q1, Q3) | |
|---|---|---|
| PD Analyte | <b>OC Alone (N = 15)</b> | OC + GS-5816 (N = 13) |
| LH (mIU/mL) | 8.0 (2.9, 12.7) | 9.3 (5.4, 14.4) |
| FSH (mIU/mL) | 3.6 (2.0, 5.9) | 2.6 (2.2, 5.1) |
| Progesterone (ng/mL) | 0.24 (0.17, 0.39) | 0.27 (0.18, 0.80) |

Based on these results, no loss in contraceptive efficacy is expected upon administration of combined oral contraceptives containing norgestimate/ethinyl estradiol with VEL. Study GS-US-334-0146 previously demonstrated that the use of SOF with contraceptives (e.g., norgestimate/ethinyl estradiol) is permitted. Accordingly, the use of hormonal contraceptives with VEL as a single agent or as part of SOF/VEL FDC is permitted.

# 1.2.2.2.2. Drug-Drug Interaction Studies with SOF/VEL and Gastric Acid Suppressants

GS-US-342-1346 and GS-US-342-1709 were open-label, Phase 1, single-dose drug-drug interaction studies in healthy volunteers evaluating the effect of gastric acid suppressants (H2RAs and PPIs) on the PK of SOF/VEL. A summary of results from these studies are presented in the Table 1-4 below.

Study GS-US-342-1346 demonstrated that simultaneous or staggered (12 hour) administration of SOF/VEL, administered under fasting conditions, with famotidine 40 mg resulted in no change to the AUC of SOF or VEL, suggesting that SOF/VEL can be administered simultaneously or staggered with H2RAs at doses comparable to famotidine 40 mg. Study GS-US-342-1346 also demonstrated that simultaneous or staggered (12 hour) administration of SOF/VEL, administered under fasting conditions, with omeprazole 20 mg resulted in a reduction in VEL AUC of 37% and 56%, respectively. The AUC of SOF also decreased 29% to 44%, respectively, though these effects are secondary to the impact of PPIs on VEL, as SOF does not demonstrated pH-dependent solubility. Based on these data, the use of SOF/VEL under fasting conditions with PPIs is not recommended.

Study GS-US-342-1709 evaluated the effect of omeprazole 20 mg or 40 mg on the PK of SOF/VEL when SOF/VEL is administered with food. Administration of SOF/VEL with food and

omeprazole did not alter the overall exposure (AUC) of SOF or its metabolites, regardless of timing or dose of omeprazole. Administration of SOF/VEL with food and omeprazole resulted in a decrease in VEL exposure. The smallest decrease in VEL exposure (AUC: 26%, C<sub>max</sub>: 33%) was observed following administration of SOF/VEL with food 4 hours before omeprazole 20 mg. A slightly greater decrease in VEL exposure (AUC: 38%, C<sub>max</sub>: 48%) was observed when SOF/VEL was administered with food 2 hours after omeprazole 20 mg. The largest decline in VEL exposure (AUC: 53%, C<sub>max</sub>: 56%) was observed following SOF/VEL administration with food 4 hours before omeprazole 40 mg.

Collectively, these studies indicate that PPIs can impact the PK of SOF/VEL. Administration of SOF/VEL with food reduces the effect of omeprazole on SOF/VEL PK. The overall exposure of SOF and its metabolites were not affected by omeprazole 20 mg when SOF/VEL was administered with food, and the reduction in VEL exposure was less when administered with food (26% to 38%) compared to fasted administration (37% to 56%). Staggering timing of omeprazole 20 mg and SOF/VEL administration also modestly impacted VEL exposure; VEL AUC was least impacted when administered 4 hours before omeprazole 20 mg (equivalent to 20 hours after the previous omeprazole dose).

Study GS-US-342-1709 also demonstrates that the nature of VEL exposure decrease was not uniform across the study population. Largest decreases were observed in subjects with highest exposure at reference, and those with low exposure at reference were generally unaffected by administration with a PPI. These data suggests that gastric pH is a contributor to the natural variability of VEL, and the range of exposure for HCV-infected subjects on PPIs is expected to be within that observed in Phase 3 ASTRAL studies. Accordingly, PPI doses comparable with omeprazole 20 mg can be administered with SOF/VEL when SOF/VEL is administered with food.

Table 1-4. Summary of Changes in SOF/VEL PK following administration with Representative H2RAs and PPIs

| | Dosing | SOF PK Parameters | | | GS-331007 PK<br>Parameters | | | VEL PK Parameters | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study | Scheme | AUC <sub>last</sub> | AUCinf | C <sub>max</sub> | AUC <sub>last</sub> | AUCinf | C <sub>max</sub> | AUC <sub>last</sub> | AUCinf | C <sub>max</sub> |
| GS-US-<br>342-1346<br>(N=60) | SOF/VEL<br>(fasted) with<br>simultaneous<br>FAM 40 mg | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ |
| | SOF/VEL<br>(fasted) with<br>12 hours<br>after FAM<br>40 mg | $\leftrightarrow$ | $\leftrightarrow$ | ↓23% | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ |
| | SOF/VEL<br>(fasted) with<br>simultaneous<br>OME 20 mg | ↓29% | ↓29% | ↓34% | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | ↓37% | ↓36% | ↓37% |
| | SOF/VEL<br>(fasted) 12<br>hours after<br>OME 20 mg | ↓44% | ↓44% | ↓45% | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | ↓56% | ↓55% | ↓57% |
| GS-US-<br>342-1709<br>(N=40) | SOF/VEL<br>(fed) 2 hours<br>After OME<br>20 mg | $\leftrightarrow$ | $\leftrightarrow$ | ↓16% | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | ↓38% | ↓38% | ↓48% |
| | SOF/VEL<br>(fed)<br>4 hours<br>Before OME<br>20 mg | $\leftrightarrow$ | $\leftrightarrow$ | ↓21% | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | ↓26% | ↓26% | ↓33% |
| | SOF/VEL<br>(fed) 4 hours<br>Before OME<br>40 mg | $\leftrightarrow$ | $\leftrightarrow$ | ↓30% | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | ↓53% | ↓53% | ↓56% |

FAM = famotidine; OME = omeprazole

The 90% CIs of the %GLSM ratios were within (↔), or extended below (↓) the predetermined PK alteration boundary of 70%.

# 1.3. Rationale for This Study

After transplantation, recurrence of HCV infection occurs in almost all subjects {Feray et al 1992, Wiesner et al 2003, Wright et al 1992} and is associated with cirrhosis, fibrosing cholestatic hepatitis, graft loss, liver re-transplantation, and death {Berenguer 2002, Berenguer et al 2000, Charlton et al 2014, Firpi et al 2009, Forman et al 2002, Gane 2008, Marks et al 2012, Prieto et al 1999, Wiesner et al 2003}. Recurrence of infection is immediate in recipients who are serum HCV RNA-positive at liver transplantation (LT).

Anti-viral therapies based on pegylated interferon-alpha (PEG) have been studied and may be indicated prior to liver transplantation (pre-emptive therapy) or later once chronic hepatitis has been confirmed and immunosuppression is relatively low {Calmus et al 2012, Crippin et al 2002, Forns et al 2003, Samuel et al 2003, Terrault 2008, Wang et al 2006. These regimens therapy have clear limitations: poor tolerance, poor efficacy and severe adverse reactions. More recently, anecdotal evidence has shown that treatment with protease inhibitors which have to be combined with pegylated interferon-alpha and ribavirin are being used as a last resort due to hard to manage drug-drug interactions with immunosuppression drugs and adverse events. SOF + RBV is currently approved in the US and Europe to be used in patients with HCV prior to transplantation to prevent post-transplant HCV reoccurrence (Gilead Sciences Inc 2013). The efficacy of this regimen is up to 70%, so this does offer an option over pegylated interferon regimens, but does not eliminate the use of pegylated interferon by practicing clinicians. Furthermore, this treatment regimen does not address patients with HCV reoccurrence who have already had their liver transplant. LDV/SOF + ribavirin for 12 weeks and LDV/SOF (without ribavirin) for 12 weeks (in patients without cirrhosis or 24 weeks (in patients with cirrhosis)) may be considered for patients who are ineligible or intolerant to ribavirin. Additionally, LDV/SOF + RBV is the only approved SOF-based, non-pegylated interferon regimen currently available for post-transplant patients. It is approved only in Europe for the treatment patients after liver transplant with genotypes 1, 4, 5, 6 HCV infections based on results from SOLAR-1 and SOLAR-2{Charlton et al 2015}. Though this regimen offers high efficacy, the limited genotype indication and requirement of ribavirin still leaves room for a non-RBV, non-interferon HCV regimen available to all patients with liver transplants and HCV infections, regardless of genotype.

This is a multicenter, open-label, Phase 2 study designed to evaluate SOF/VEL for 12 weeks in post liver transplant subjects with recurrent chronic HCV infection. Approximately 80 subjects with chronic HCV will be enrolled. Approximately 20% will have genotype 3 HCV infection and up to approximately 20% with Metavir stage 3 or 4 fibrosis/cirrhosis or corresponding fibrosis degree is approximately 20% at baseline will be enrolled.

This study will evaluate the safety and efficacy of SOF/VEL FDC for 12 weeks in subjects with recurring HCV infection (without cirrhosis or with compensated liver cirrhosis) following a liver transplant.

#### 1.4. Rationale for Dose Selection

Sofosbuvir 400 mg, once daily, when dosed in combination with RBV with or without PEG has demonstrated broad genotypic efficacy and favorable safety profile in over 1700 HCV-infected subjects across multiple patient populations in Phase 2 and 3 trials. This dose is the approved marketed dose of sofosbuvir for the treatment of HCV-infection and as such, has been selected for co-formulation with VEL into a fixed-dose combination tablet.

VEL 100 mg has been administered in combination with SOF 400 mg for 12 weeks to 237 HCV-infected subjects in Phase 2 studies. VEL 100 mg was selected for co-formulation with SOF and evaluation in this study based on the Phase 2 safety, PK and antiviral activity (studies GS-US-342-0102, GS-US-342-0109, and GS-US-337-0122 [Cohort 4]). The Phase 1
study GS-US-281-0102 established the anti-HCV activity of VEL and indicated that the exposures achieved following administration of doses > 25 mg provide at least 80% of maximal antiviral response in all HCV genotypes.

The favorable safety and efficacy profiles of SOF 400 mg and VEL 100 mg support further evaluation of this combination and doses in clinical development.

## 1.5. Risk/Benefit Assessment for the Study

This study will provide information on the safety and efficacy of SOF/VEL, a potent HCV nucleotide inhibitor and a potent HCV NS5A inhibitor. This combination has the potential to be the first once-daily, PEG-free, RBV-free, pangenotypic regimen for the treatment of chronic HCV infection in patients who have received a liver transplant.

The potential benefits of SOF/VEL over the current standard of care for the treatment of chronic HCV are:

- A once-daily, single tablet, single duration, pangenotypic therapy for HCV recurrence in patients with liver transplants could offer PEG-free treatment options to patients with genotypes that currently do not have approved PEG-free regimens
- The once-daily, single tablet, single duration, pangenotypic HCV reoccurrence regimen would offer a simplified algorithm for treatment of HCV recurrence in all patients with liver transplants, regardless of genotype
- A reduction in the AEs currently associated with the use of PEG (particularly for post-transplant patients with genotypes that do not have approved PEG-free regimens) and RBV (for all post-transplant patients, regardless of genotype).
- A reduction in the significant drug-drug interactions that are common amongst patients with liver transplants on complex immunosuppressive regimens.
- A short duration of therapy which should lead to better outcomes through improved adherence.

The safety profile of SOF in clinical studies includes over 1700 chronic HCV-infected subjects that have been administered  $\geq$  12 weeks of SOF and RBV+/-PEG-IFN. No clinical safety issues specifically related to SOF have been identified to date.

The safety profile of SOF + VEL 25mg or VEL 100mg administered for 8 or 12 weeks has been established in over 800 patients in Phase 2 studies. The safety profile of the proposed therapeutic regimen of SOF 400 mg and VEL 100 mg administered for 12 weeks has been established in 237 subjects enrolled in Phase 2 studies. No clinical safety issues specifically related to VEL or SOF + VEL have been identified to date. No clinical safety issues specifically related to the NS5A inhibitor class including daclatasvir (DCV) and LDV have been identified to date {Afdhal et al 2014a, Afdhal et al 2014b, Kowdley et al 2014}.

The safety profile of SOF/VEL has been studied in 4 Phase 3 trials (ASTRAL 1-4) in 1302 patients. Twelve weeks of SOF/VEL was generally well tolerated, and lead to a similar incidence of AEs and SAEs compared to placebo in patients with GT 1, 2, 4, 5, or 6 HCV (See Section 1.2.2.2.1.1). When 12 weeks of SOF/VEL was compared to SOF + RBV for 12 weeks in patients with GT2 or 3 HCV, therapy with SOF/VEL was again well tolerated with few differences in AEs or SAEs, minus the avoidance of RBV associated toxicities (See Sections 1.2.2.2.2 and 1.2.2.1.3). Patients who received SOF/VEL for either 12 or 24 weeks with decompensated cirrhosis experienced AEs and SAEs typical for patients with decompensated cirrhosis in no pattern that could be attributed to study drug (See Section 1.2.2.1.4). Patients with decompensated cirrhosis who received SOF/VEL + RBV for 12 weeks also experienced AEs and SAEs consistent with underlying liver disease as well as toxicities expected with RBV treatment (See Section 1.2.2.1.4).

In summary, there is no approved Peg-IFN-free or RBV-free treatment available for patients with liver transplants and chronic HCV recurrence. If high rates of SVR can be obtained with a short, IFN-free, RBV-free, pangenotypic regimen, the anticipated improvements in safety and tolerability would offer a favorable risk-benefit ratio for such patients.

## 1.6. Compliance

This study will be conducted in compliance with this protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements.

## 2. OBJECTIVES

The primary objectives of this study are:

- To evaluate the efficacy of study treatment with sofosbuvir (SOF)/velpatasvir (VEL) FDC for 12 weeks as measured by the proportion of subjects with sustained viral response 12 weeks after cessation of study treatment regimen (SVR12)
- To evaluate the safety and tolerability of the study treatment regimen

The secondary objectives of this study are:

- To determine the proportion of subjects who attain SVR at 4 weeks after cessation of the study treatment regimen (SVR4)
- To evaluate the kinetics of circulating HCV RNA during the study treatment and after cessation of the study treatment regimen
- To evaluate the emergence of viral resistance to SOF and VEL during study treatment and after cessation of study treatment regimen

The exploratory objective of the pharmacogenomics substudy is:



## 3. STUDY DESIGN

## 3.1. Treatment Plan and Regimen

This is a multicenter, open-label study that will evaluate the safety, tolerability and efficacy of SOF/VEL FDC administered for 12 weeks in subjects with chronic HCV post-liver transplant.

Approximately 80 subjects with recurrent HCV post-liver transplant will be enrolled and treated with SOF/VEL FDC tablet once daily for 12 weeks.

The enrollment target for subjects with GT 3 HCV infection is approximately 20%. The enrollment target for subjects with Metavir stage 3 or 4 fibrosis/cirrhosis or corresponding fibrosis degree is approximately 20%.

The total time to complete all study visits is approximately 28 weeks (30 weeks for those requiring liver biopsy or additional HCV genotype testing at screening):

- 28 day (4 week) screening period (can be extended up to 42 days if liver biopsy, additional HCV genotype testing is required, or for extenuating circumstances)
- 12 week study treatment period
- Up to 12 week post study treatment period

#### 3.2. Visit Schedule

All subjects will complete screening, on treatment, and post-treatment assessments.

Screening assessments will be completed within 28 days of the Baseline/Day 1 visit. The screening window can be extended to 42 days for subjects requiring liver biopsy, additional HCV genotype testing, or for extenuating circumstances.

All subjects will complete the following study visits: Screening, Baseline/Day 1, on treatment visits at the end of Weeks 2, 4, 8 and 12. All subjects will complete the post-treatment Week 4 visit. Subjects with HCV RNA <LLOQ at the post-treatment Week 4 visit will complete post-treatment Week 12 visit. Subjects with HCV RNA ≥LLOQ at post-treatment Week 4 or post-treatment Week 12s visit will be asked to return for confirmatory visit.

The assessments performed at each visit are described in Section 6 and Appendix 2.

## 3.3. HCV Virologic Response-Based Stopping Criteria

The following on-treatment HCV virologic response-based treatment stopping criteria will be utilized for all subjects:

• Confirmed HCV RNA ≥LLOQ after 2 consecutive HCV RNA <LLOQ

- Confirmed >1 log<sub>10</sub> increase from nadir
- HCV RNA ≥LLOQ through 12 weeks of treatment

Confirmation should be performed as soon as possible but within 2 weeks after determination of initial observation indicating virologic failure.

If HCV viral relapse is detected at post-treatment Week 4 or 12 visits, subjects will be asked to return for a confirmatory visit.

## 3.4. Stopping Rules for Individual Subjects

Subjects who meet any of the following criteria should be discontinued from the study and complete an Early Termination Visit and return for Post-treatment Follow-up visits:

- Elevation of ALT and/or AST that is greater than the ULN and > 5x baseline or nadir confirmed by immediate repeat testing unless laboratory results are assessed by both the investigator and Gilead Medical Monitor as having an explanation other than drug induced liver injury and it is deemed in the best interest of the subject to continue HCV treatment
- Confirmed elevation of ALT >15 x ULN (unrelated to any interventional procedures)
- Confirmed total bilirubin >10 x ULN (unrelated to any interventional procedures)
- Confirmed total bilirubin >3x baseline or 3x nadir (unrelated to any interventional procedures)
- Any Grade 3 or greater rash associated with constitutional symptoms
- Any non-laboratory Grade 4 events assessed as related to administration of SOF/VEL
- Worsening of disease state as evidenced by progressing hepatic decompensation and/or progression of Child-Pugh Score (CPT) to ≥ 10
- Steroid-resistant acute allograft rejection

The Gilead Medical Monitor should be consulted prior to discontinuation of SOF/VEL unless the investigator believes that immediate action is warranted to ensure the continued safety of the subject.

Any questions regarding toxicity management should be directed to Gilead Medical Monitor.

#### 3.5. Discontinuations

If the subject meets the Virologic Response-Based Criteria (Section 3.3), they should complete an Early Termination Visit as soon as possible after SOF/VEL is discontinued and complete post-treatment visits up to 30 days after the last dose of SOF/VEL to assess for safety.

If the subject meets the Stopping Rules for Individual Subjects (Section 3.4) or other criteria for discontinuation of study treatment (Section 3.7), prior to completion of SOF/VEL dosing period, the subject should complete an Early Termination Visit as soon as possible after SOF/VEL is discontinued and complete the post-treatment assessments as described in Section 6.3 and in Study Procedures Appendix 2.

Subjects discontinuing treatment prior to completion of dosing period for reasons other than those described in Sections 3.3, 3.4 and 3.7 should complete an Early Termination Visit as soon as possible after SOF/VEL is discontinued. The subject should also complete the post-treatment assessments as described in Section 6.3 and in Study Procedures Appendix 2.

## 3.6. Assessments for Premature Discontinuation from Study

If a subject discontinues SOF/VEL dosing (for example, as a result of an adverse event [AE]), every attempt should be made to keep the subject in the study and continue to perform the required study-related post-treatment assessments and procedures (see Section 6.3). If this is not possible or acceptable to the subject or investigator, the subject may be withdrawn from the study.

## 3.7. Criteria for Discontinuation of Study Treatment

When medically feasible, the Medical Monitor must be consulted prior to subject discontinuation.

Study drug must be discontinued in the following instances:

- Intercurrent illness that would, in the judgment of the investigator, affect assessments of clinical status to a significant degree
- Unacceptable toxicity, as defined in the toxicity management section of the protocol (Section 7.5), or toxicity that, in the judgment of the investigator, compromises the ability to continue study-specific procedures or is considered to not be in the subject's best interest
- Subject requests to discontinue for any reason; it is important to determine whether the withdrawal of consent is primarily due to an AE, lack of efficacy or other reason
- Subject non-compliance
- Pregnancy
- Discontinuation of the study at the request of Gilead, regulatory agency or an IRB/IEC

#### 3.8. **Biomarker Testing**

#### 3.8.1. Biomarker Samples for Optional Future Research



#### 3.8.2. Biomarker Samples for Optional Pharmacogenomics Research

PPD



## 4. SUBJECT POPULATION

## 4.1. Number of Subjects and Subject Selection

Approximately 80 chronic HCV infected subjects who had a liver transplant will be enrolled in this study. Patients both with cirrhosis (if compensated) and without cirrhosis and with treatment experienced (if non-NS5A) or treatment naïve will be eligiable.

In order to manage the total study enrollment, Gilead Sciences, Inc., at its discretion, may suspend screening and/or enrollment at any site or study-wide at any time.

## 4.2. Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

- 1) Willing and able to provide written informed consent
- 2) Males and females, age  $\geq$  18 years old
- 3) Chronic HCV infection (≥6 months) documented pretransplantation by prior medical history or liver biopsy
- 4) HCV RNA  $\geq 10^4$  IU/mL at screening
- 5) No clinical signs of rejection for 3 months prior to the Screening visit
- 6) Primary or secondary (re-transplant), liver alone or liver and kidney transplant recipient from deceased or living donor (regardless of the HCV status of the liver donor)
- 7) Liver transplant  $\geq 3$  months prior to screening
- 8) A body mass index (BMI) of  $\geq 18 \text{ kg/m}^2$
- 9) Subjects must have a determination of treatment experience (treatment naïve v. treatment experienced). Treatment naïve is defined as having never been exposed to an approved or experimental HCV-specific direct acting antiviral agents or prior treatment of HCV with interferon or ribavirin. All other patients will be considered treatment experienced
  - a) If treatment experienced, the subject's medical records must include details of prior treatment regimen(s). Any prior use of SOF or other nucleotide analogue HCV NS5B inhibitor should be documented. Previous use of an NS5A inhibitor is not allowed.

- 10) Subjects must have appropriate testing for determination of cirrhosis status.
  - a) Presence of cirrhosis is defined as any one of the following:
    - i) Fibrotest® score > 0.75 AND an AST platelet ration index (APRI) > 2 performed during Screening
    - ii) Fibroscan with a result of > 12.5 kPa within  $\le 6$  months of Baseline/Day 1
    - iii) Liver biopsy showing cirrhosis (e.g., Metavir score = 4 or Ishak score  $\geq 5$ )
  - b) Absence of cirrhosis is defined as any one of the following:
    - i) Fibrotest score  $\leq 0.48$  AND APRI  $\leq 1$  performed during Screening
    - ii) Fibroscan with a result of  $\leq 12.5$  kPa within  $\leq 6$  months of Baseline/Day 1
    - iii) Liver biopsy performed within 2 years of Screening showing absence of cirrhosis

In the absence of a definitive diagnosis of presence or absence of cirrhosis by Fibrotest /APRI using the above criteria, a liver biopsy or fibroscan is required. A diagnosis of cirrhosis will supersede a diagnosis of non-cirrhosis and be considered definitive.

- 11) Liver imaging within 6 months of Baseline/Day 1 is required in cirrhotic subjects only to exclude hepatocellular carcinoma (HCC)
- 12) A negative serum pregnancy test is required for female subjects (unless permanently sterile or greater than two years post-menopausal)
- 13) Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in Appendix 6
- 14) Lactating females must agree to discontinue nursing before the study drug is administered
- 15) Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments

#### 4.3. Exclusion Criteria

Subjects who meet *any* of the following exclusion criteria are not to be enrolled in this study:

- 1) Multi-organ transplant that includes heart or lung recipient (patients who have their liver transplant as part of a liver-kidney dual transplant are eligible to enroll)
- 2) Subjects with de novo or recurrent Hepatocellular Carcinoma (HCC) posttransplant

- 3) Current use of corticosteroids at any dose >5mg of prednisone/day (or equivalent dose of corticosteroid)
- 4) Child-Pugh-Turcotte (CPT) Score >7 at Screening
- 5) Recipient of ABO incompatible organ
- 6) Histological evidence of unresolved rejection
- 7) Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV) at Screening
- 8) Current, uncontrolled ascites, variceal hemorrhage, hepatic encephalopathy, hepatorenal syndrome, hepatopulmonary syndrome, or other signs of decompensated cirrhosis
- 9) Serum creatinine >2.5x upper limit of normal (ULN) or stage 4 chronic kidney disease (CrCl <30ml/min)
- 10) Screening ECG with clinically significant abnormalities
- 11) Subjects with the following laboratory results at Screening are excluded unless enrollment is approved by the sponsor medical monitor
  - ALT, AST or alkaline phosphatase >10 x ULN
  - Direct bilirubin >4 x ULN
  - WBC < 2.000/mm<sup>3\*</sup>
  - ANC <1,000cells/mm<sup>3\*</sup>
  - Platelets <50,000/mm<sup>3\*</sup>
  - HbA1C >8.5%
  - Hemoglobin <9g/dL\*
  - \*Use of GM-CSF, epoetin alfa or other therapeutic agents to increase cell counts for the purposes of meeting eligibility criteria is prohibited.
- 12) Use of GM-CSF, epoetin alfa or other therapeutic agents within 2 weeks of Screening
- 13) History of other clinically relevant chronic liver disease (e.g., hemochromatosis, autoimmune hepatitis, Wilson's disease,  $\alpha$ -1-antitrypsin deficiency, alcoholic liver disease, non-alcoholic steatohepatitis, or toxin exposure)
- 14) Recent (within 4 weeks of Screening) episode or infection requiring systemic antibiotics

- 15) Use or planned use of T-cell depleting/masking antibodies, systemic antineoplastic agents, cyclosporine >300mg/day,or use of any prohibited medications listed in Section 5.4 within 28 days of the Baseline/Day 1 visit
- 16) Prior exposure to any HCV NS5A inhibitor
- 17) History or current evidence of immunologic disorder, hemoglobinopathy, pulmonary or cardiac disease, porphyria, seizure disorder, poorly controlled diabetes, pancreatitis with elevated lipase, cancer, or a history of malignancy (with exception of certain resolved skin cancers or pre-transplant hepatocellular carcinoma; patients who received liver transplants for hepatocellular carcinoma must be 5 years post-transplant with no evidence of recurrence at Screening) that in the opinion of the investigator makes the subject unsuitable for the study
- 18) Treatment for HCV infection with experimental or approved regimens within 3 months of Baseline/Day 1.
- 19) Participation in a clinical study with an investigational drug, or biologic within 3 months prior to Baseline/Day 1
- 20) Clinically relevant alcohol or drug abuse within 12 months of Screening. A positive drug screen will exclude subjects unless it can be explained by prescribed medications; the diagnosis and prescription must be approved by the investigator
- 21) History or difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
- 22) Known hypersensitivity to SOF (and the metabolites), and/or VEL

### 5. INVESTIGATIONAL MEDICINAL PRODUCTS

## 5.1. Enrollment and Study Drug Supply

This is an open-label study. An Interactive Web Response System (IWRS) will be employed to manage subject enrollment and the study drug dispensing as well as re-supply of study drug.

## 5.2. Description and Handling of SOF/VEL FDC

#### **5.2.1.** Formulation

The SOF/VEL (400/100 mg) tablets are pink, diamond-shaped, film-coated tablets, debossed with "GSI" on one side and "7916" on the other side. In addition to the active ingredients, the SOF/VEL tablets contain copovidone, microcrystalline cellulose, croscarmellose sodium, magnesium stearate, polyvinyl alcohol, titanium dioxide, polyethylene glycol, talc, and iron oxide red.

## 5.2.2. Packaging and Labeling

SOF/VEL (400/100 mg) tablets are packaged in white, high density polyethylene (HDPE) bottles. Each bottle contains 28 tablets and polyester packing material. Each bottle is enclosed with a white, continuous thread, child-resistant screw cap with an induction-sealed, aluminum-faced liner.

SOF/VEL bottles to be distributed to centers in participating countries shall be labeled to meet all applicable requirements of the US Food and Drug Administration (FDA), EU Guideline to Good Manufacturing Practices – Annex 13 (Investigational Medicinal Products), and/or other local regulations.

#### 5.2.3. Storage and Handling

SOF/VEL tablets should be stored at controlled room temperature until required for administration. Controlled room temperature is defined as 25°C (77 °F); excursions are permitted between 15°C and 30°C (59°F to 86°F).

All drug products should be stored in a securely locked area, accessible only to authorized site personnel. To ensure the stability of the study drug and to ensure proper product identification, the drug product should not be stored in a container other than the container in which they are supplied. Consideration should be given to handling, preparation, and disposal through measures that minimize drug contact with the body. Appropriate precautions should be followed to avoid direct eye contact or exposure through inhalation when handling SOF/VEL tablets.

Sufficient quantities of SOF/VEL tablets to complete the entire study will be shipped to the investigator or qualified designee from Gilead Supply Management Team (or its designee).

## 5.3. Dosage and Administration

SOF/VEL tablet is to be administered once daily with or without food. Each subject must be given instructions to maintain approximately the same daily dosing interval between study drug doses.

For a missed dose of study medication, subjects must be instructed to take the missed dose of study medication as soon as possible during the same day. Subjects should be cautioned never to double the next dose with a missed dose of study drug under any circumstances.

#### 5.4. Prior and Concomitant Medications

Concomitant medications taken within 30 days of Screening, up to and including the date of the visit four weeks after discontinuation of study drug, need to be recorded in the source documents and eCRFs. All concomitant medications should be recorded in the source documents (including all blood products).

For subjects on a calcineurin inhibitor (e.g., tacrolimus, sirolimus, everolimus) for post-transplant immunosuppression, levels should be collected as per the standard schedule (or as clinically indicated) for dose management at the clinical site, and processed at the local laboratory. Management of the immunosuppression is not part of the clinical protocol, but levels and resulting dose adjustments will be recorded to assess whether the regimens required adjustment in correlation with resolution of the HCV infection.

The following medications are prohibited from 28 days prior to the Baseline/Day 1 visit through the end of study drug dosing:

- Use of corticosteroids at any dose > 5mg of prednisone/day (or equivalent dose of corticosteroid) for maintenance of immunosuppression is prohibited. However, use of steroids for the short term treatment of Acute Cellular Rejection (ACR) is up to the discretion of the Investigator.
- Investigational agents or devices for any indication

Concomitant use of certain medications or herbal/natural supplements (inducers of drug transporters i.e. P-gp) with study drug may result in pharmacokinetic interactions resulting in increases or decreases in exposure of study drug or these medication. The use of the following agents is prohibited from 28 days prior to Baseline/Day 1 through the end of study drug dosing. The use of amiodarone is prohibited from 60 days prior to Baseline/Day 1 through the end of study drug dosing.

Examples of representative medications which are prohibited or are to be used with caution are listed below:

Table 5-1. List of Disallowed/ Use with Caution Medications

| Drug Class | Agents Disallowed | <b>Use with Caution</b> |
|---|---|---|
| Acid Reducing Agents <sup>a</sup> | | Proton Pump Inhibitors, H2-Receptor<br>Antagonists, Antacids, |
| Anticonvulsants <sup>b</sup> | Phenobarbital, Phenytoin,<br>Carbamazepine, Oxcarbazepine | |
| Antimycobacterials <sup>b</sup> | Rifabutin, Rifapentine, Rifampin | |
| Cardiac Medications <sup>c</sup> | Amiodarone <sup>f</sup> | Diltiazem, Verapamil, Dronedarone,<br>Quinidine, Ranolazine, Bosentan,<br>Olmesartan, Valsartan, Digoxin <sup>d</sup> |
| Herbal/Natural<br>Supplements <sup>b</sup> | St. John's Wort, Echinacea. Milk thistle (i.e. silymarin), Chinese herb sho-saikoto (or Xiao-Shai-Hu-Tang) | |
| HMG-CoA Reductase<br>Inhibitors <sup>e</sup> | | Rosuvastatin (≤10 mg/day) |
| Other | Modafinil <sup>b</sup> , Sulfasalazine <sup>c</sup> , Methotrexate <sup>c</sup> | |

a Proton pump inhibitor (PPI) doses comparable with omeprazole 20 mg can be administered with SOF/VEL when SOF/VEL is administered with food. H2-receptor antagonists must not exceed a dose of 40 mg famotidine or equivalent and can be taken simultaneously with SOF/VEL and/or staggered by 12 hours. Antacids that directly neutralize stomach acid (i.e. Tums, Maalox) may not be taken within 4 hours (before or after) of SOF/GS-5816 administration.

- b May result in a decrease in the concentration of study drugs.
- c May result in an increase in the concentration of study drugs and/or concomitant medications
- d Monitor for signs and symptoms of digoxin toxicity.
- e Use with SOF/VEL may result in an increase in the concentration of HMG-CoA reductase inhibitor rosuvastatin.. Monitor for signs and symptoms of muscle weakness or myopathy, including rhabdomyolysis.
- f May result in symptomatic bradycardia. Mechanism is not currently known. The use of amiodarone is prohibited from **60 days prior to Baseline/Day 1** through the end of treatment

Medications for disease conditions **excluded** from the protocol (e.g., HIV-1 infection, active cancer) are not listed under this Concomitant Medication section and are disallowed in the study.

Subjects may not take any approved HCV medications during their participation in the study period.

Should subjects have a need to initiate treatment with any excluded concomitant medication, the Medical Monitor must be consulted prior to initiation of the new medication. In instances where an excluded medication is initiated prior to discussion with the Sponsor, the Investigator must notify Gilead as soon as he/she is aware of the use of the excluded medication.

### 5.4.1. Colony Stimulating Agents

Potential subjects may not be treated with colony stimulating agents (CSA) during Screening to elevate hematology laboratory parameters to facilitate entry into the study. Use during the study is allowed as clinically indicated. Use should be captured as a concomitant medication.

## 5.5. Management of Rejection

The diagnosis of ACR, based on liver biopsy, and the decision to treat are important concerns due to the potential interactions between immunosuppression and the success of HCV treatment. It is expected that this will not be a common occurrence in this study, given that subjects must be stable and at least 6 months from transplant at study entry. Sites will be asked to follow their institutional guidelines for the management of organ rejection, but to also give consideration to the following issues as related to this study protocol. (This information is provided for guidance and consistency across subjects, but variations will not be considered protocol violations if the treatment is consistent with the guidelines of the institution).

- It is important to use standard criteria for diagnosis of rejection, to avoid over-treatment of milder grades of rejection with corticosteroids whenever possible, and to standardize the exposure to corticosteroids when treatment for rejection is necessary
- Episodes of rejection will be recorded on the CRF and severity will be graded (grading by Banff criteria, Appendix 5)
- It is preferred that mild ACR is to be treated with upward adjustment of maintenance immunosuppression rather than the addition of corticosteroids
- Cases of moderate or severe ACR may require treatment with corticosteroids
- Cases of presumptive rejection should be confirmed by liver biopsy (as per standard practice) if more than one dose of corticosteroid is required
- Subjects with steroid-resistant ACR should be discontinued from the study so that management of their organ rejection can be the primary focus of treatment.

## 5.6. Study Drug Accountability

The investigator is responsible for ensuring adequate accountability of all used and unused study drug (SOF/VEL FDC). This includes acknowledgement of receipt of each shipment of study drugs (quantity and condition). All used and unused study drugs dispensed to subjects must be returned to the site.

SOF/VEL FDC accountability records will be provided to each study site:

- Record the date received and quantity of study drug bottles
- Record the date, subject number, subject initials, the study drug bottle number dispensed
- Record the date, quantity of used and unused study drug returned, along with the initials of the person recording the information.

• At the Baseline/Day 1 visit, subjects will be dispensed 2 bottles of SOF/VEL so that they have sufficient tablets to cover the 3 day time window around the Week 4 and Week 8 visit. Subjects must be instructed to bring back the study drug in the original container at every post Day 1 study visit through the end of study treatment. The extra bottle dispensed at Baseline/Day 1 visit must be brought back to each on-treatment visit for accountability purposes and will be re-dispensed to the subject except at Week 12 or EOT visit.

## 5.6.1. Study Drug Return and Disposal

Please refer to Section 9.1.7 for information pertaining to study drug return and disposal.

## 6. STUDY PROCEDURES

The study procedures to be conducted for each subject enrolled in the study are presented in tabular form in Appendix 2 and described in the text that follows. All subjects will complete the following study visits: Screening, Baseline/Day 1, on treatment visits at the end of Weeks 2, 4, 8 and 12. All subjects will complete the post-treatment Week 4 visit. Subjects with HCV RNA <LLOQ at the post-treatment Week 4 visit will complete post-treatment Week 12 visit. Subjects with HCV RNA ≥LLOQ at post-treatment Week 4 or post-treatment Week 12s visit will be asked to return for confirmatory visit. Viral breakthrough or relapse must be confirmed.

Information on the specific laboratory parameters to be measured and clinical assessment to be performed are provided in Section 6.5.

The investigator must document any deviation from protocol procedures and notify the sponsor or contract research organization (CRO).

### 6.1. Screening Assessments

## 6.1.1. Screening Visit (Day 28 to Day 0)

Subjects will be screened within 28 days of Baseline/Day 1 visit. The screening window can be extended to 42 days for subjects requiring liver biopsy, additional HCV genotype testing or for extenuating circumstances.

The following will be performed and documented:

Obtain written informed consent



- Determine inclusion and exclusion eligibility
- Obtain medical history, including
  - Hepatitis C history
  - Liver transplant history
  - Liver biopsy results (if applicable)

- Determine cirrhosis status as defined in Section 4.1
  - If the presence of cirrhosis is determined, then appropriate diagnostic imaging (CT or Ultrasound) should be performed or confirmed to have been performed within 6 months of screening to exclude the presence of hepatocellular carcinoma (HCC)
- Determine treatment experience status as defined in Section 4.1
  - If treatment experienced, record the duration(s) and type(s) of the prior treatment administered.
  - If treatment experienced, record whether or not any past treatment regimens contained SOF or other nucleotide analogue HCV NS5B inhibitors.
- Complete physical examination including, vital signs (temperature, blood pressure, pulse, respiratory rate), body weight, and height
- Obtain details of concomitant medications
- Perform 12-lead ECG
- Fibrosis Assessment
- Calculate CPT score
- Obtain blood samples for tests as listed in Section 6.6.2:
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Determination of HCV viral genotype and subtype
  - HCV antibody, HIV, and HBV surface antigen (HBV serology)
  - $HbA_{1c}$
  - IL28B
  - Serum β-hCG pregnancy test for females of childbearing potential only

- Obtain urine sample for:
  - Urinalysis
  - Serum pregnancy test for females of childbearing potential
  - Urine drug screen
- Record any serious adverse events and all adverse events related to protocol mandated procedures occurring after signing of the consent form.
- Retests of Screening labs are permitted only if there is reason to believe the retest value will
  be within accepted parameters, for example, if the initial exclusionary value was either due to
  a sample processing error or due to an extenuating circumstance such as intercurrent illness.
- Subjects meeting all of the inclusion criteria and none of the exclusion criteria will return to the clinic for the Baseline/Day 1 Visit assessments and enrollment into the study.

From the time of obtaining informed consent through the first administration of investigational medicinal product, record all serious adverse events (SAEs), as well as any adverse events related to protocol-mandated procedures on the adverse events case report form (eCRF). All other untoward medical occurrences observed during the screening period, including exacerbation or changes in medical history are to be captured on the medical history eCRF. See Section 7 Adverse Events and Toxicity Management for additional details.

#### **6.2.** Treatment Assessments

## 6.2.1. Baseline/Day 1 Visit

The following baseline tests and procedures must be completed prior to enrollment and dosing/dispensing of study drug:

- Confirm eligibility (Reference Sections 4.2 & 4.3)
- Perform complete physical examination, including body weight
- Obtain vital signs (resting blood pressure, pulse, respiratory rate and temperature)
- Assessment of AEs and concomitant medications
- Conduct pregnancy prevention counseling
- Obtain blood samples for:
  - Hematology

- Chemistry
- Coagulation tests
- HCV RNA
- Viral sequencing
- Obtain blood sample for Pharmacogenomics testing (for subjects who have consented)



- Obtain urine samples for the following procedures:
  - Urinalysis
  - Pregnancy test for females of child bearing potential only
- Study Drug Administration
  - Dispense study drug as directed by the IWRS
  - Instruct the subject on the packaging, storage and administration of the study drug
  - Observe the subject taking the first dose of study drug and record the time of first dose and whether it was taken with or without food.

## 6.2.2. Week 2 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Week 2:

- Obtain vital signs (resting blood pressure, pulse, respiratory rate and temperature)
- Assessment of AEs and concomitant medications
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - HCV RNA
  - Viral sequencing
  - PK sample
- Assess adherence with study drug dosing regimen including pill count

## 6.2.3. Weeks 4 and 8 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Weeks 4 and 8:

- Obtain vital signs (resting blood pressure, pulse, respiratory rate and temperature)
- Assessment of AEs and concomitant medications
- Conduct pregnancy prevention counseling
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - HCV RNA
  - Viral sequencing
  - PK sample
- Obtain urine sample for pregnancy test (for females of child bearing potential only)
- Assess adherence with study drug dosing regimen including pill count
- Dispense study drugs as directed by the IWRS

## 6.2.4. Week 12 (± 3 days) or Early Termination (ET)

The following procedures/assessments are to be completed at the end of Week 12 or ET:

- Perform complete physical examination, including weight.
- Obtain vital signs (resting blood pressure, pulse, respiratory rate and temperature)
- Calculate CPT score
- Assessment of AEs and concomitant medications
- Pregnancy prevention counseling
- Obtain blood samples for:
  - Hematology
  - Coagulation tests

- Chemistry
- HCV RNA
- Viral sequencing
- PK sample



- Obtain urine samples for
  - Urinalysis
  - Pregnancy test for females of child bearing potential only
- Assess adherence with study drug dosing regimen including pill count. Study drug should be returned at this visit

#### 6.2.5. Unscheduled Visit

A subject should attend an unscheduled visit if requested by the sponsor or the investigator. The assessments are at the investigator's discretion. At all unscheduled visits initiated for the purpose of confirming HCV virologic failure, a sample for viral HCV RNA Sequencing/Phenotyping must be collected.

The Sponsor (e.g. Medical Monitor) and CRO must be informed, as soon as possible, when a subject comes off treatment due to an AE.

#### 6.3. Post-treatment Assessments

The post-treatment Week 4 and 12 visits should be timed from the date of last administration of study drug. All subjects must complete the post-treatment Week 4 visit. All subjects who achieve SVR4 will attend the Week 12 visit. The end of study will occur at the post-treatment Week 4 visit in the case of subjects who do not achieve SVR4, and the post-treatment Week 12 visit in the case of patients who do achieve SVR4.

## 6.3.1. Post-treatment Week 4 ( $\pm 5$ days)

The following procedures/assessments are to be completed for all subjects, 4 weeks after taking the last dose of study drug:

- Perform complete physical examination
- Obtain vital signs (resting blood pressure, pulse, respiratory rate and temperature)
- Calculate CPT score

- Assessment of AEs and concomitant medications
- Pregnancy Prevention Counseling
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - HCV RNA
  - Viral sequencing
- Obtain urine sample for pregnancy test (for females of child bearing potential only)

## 6.3.2. Post-treatment Week 12 ( $\pm$ 5 days)

The following procedures/assessments are to be completed for all subjects who achieve SVR4, 12 weeks after taking the last dose of study drug:

- Perform complete physical examination
- Obtain vital signs (resting blood pressure, pulse, respiratory rate and temperature)
- Calculate CPT score
- Assessment of AEs and concomitant medications
- Obtain blood samples for:
  - Hematology
  - Chemistry
  - HCV RNA
  - Viral sequencing

## 6.4. Confirmatory Visit

Subjects with HCV RNA ≥LLOQ at post-treatment week 12 visit will be asked to return for confirmatory visit. A sample for viral HCV RNA sequencing/phenotyping will be collected.

## 6.5. End of Study

Discontinuation from study drug dosing and discontinuation from the overall study, including the Post-treatment period, will be recorded as two separate events.

The end of study will occur at the post-treatment Week 4 visit in the case of subjects who do not achieve SVR4, and the post-treatment Week 12 visit in the case of patients who do achieve SVR4.

## 6.6. Procedures and Specifications

## 6.6.1. Clinical Laboratory Analytes

<u>Hematology</u>: Hematocrit, Hemoglobin (Hb), Platelet count, Red blood cell count (RBC), White blood cell count (WBC) with differential (absolute and percentage) including Lymphocytes, Monocytes, Neutrophils, Eosinophils, Basophils, Reticulocyte count and mean cellular volume (MCV).

Coagulation: INR, Prothrombin time (PT), Activated partial thromboplastin time (APTT).

<u>Chemistry:</u> Alanine aminotransferase (ALT/SGPT), Aspartate aminotransferase (AST/SGOT), Albumin, Alkaline phosphatase, Bicarbonate, Creatinine, Creatine kinase (CK), Total Bilirubin (reflex to Direct Bilirubin), Glucose, Lipase, Potassium, Phosphate, Sodium, Uric Acid; FibroTest®/APRI calculation, and Direct Bilirubin at Screening only.

<u>Virological Tests</u>: Serologies for HCV and HBV, Serology and/or antigen testing for HIV including reflex testing, as necessary, HCV RNA will be measured using the COBAS<sup>®</sup> Ampliprep/COBAS<sup>®</sup> TaqMan<sup>®</sup> HCV Quantitative Test, v2.0. HCV genotype and subtype will be determined using the Siemens VERSANT<sup>®</sup> HCV genotype INNO-LiPA 2.0 Assay. The Abbott RealTime HCV genotype II assay is unable to result HCV genotype 6; these subjects will be identified as "Unable to genotype" on the laboratory report as well as those with mixed genotype will be considered indeterminate. Gilead reserves the right to use alternate assays for HCV RNA, and HCV genotype should the above assays become unavailable or the results are indeterminate.

IL28B genotype will be determined by polymerase chain reaction (PCR) amplification of the SNP, rs12979860, with sequence specific forward and reverse primers and allele specific fluorescently labeled TaqMan<sup>®</sup> MGB probes. Gilead reserves the rights to use an alternate assay for IL28B determination should the above assay become unavailable.

<u>Pregnancy Tests</u>: Serum β-hCG or Urine β-hCG (if positive, requires immediate confirmation with Serum β-hCG).

<u>Additional Tests</u>: Urine Drug screen (for Amphetamines, Cocaine, Methadone, Opiates) and Hemoglobin A1c (HbA1c)

#### **Urine Collection**

<u>Urinalysis:</u> Appearance, Blood, Color, Glucose, Leukocyte esterase, pH, Protein, Urobilinogen. Reflex to microscopic urinalysis if dipstick result is abnormal. At each visit this is tested, it will be recorded whether female subjects of childbearing potential are currently menstruating.

## 6.6.2. Medical History

Medical history including details regarding illnesses and allergies, date(s) of onset, and whether condition(s) is currently ongoing, and medication history, including prior HCV treatment history (only applicable for treatment experienced subjects), will be collected on all subjects during screening. Obtain HCV treatment history as per Section 4.1.

## 6.6.3. Complete Physical Examination

A complete physical examination must include source documentation of general appearance, and the following body systems: Head, neck and thyroid; eyes, ears, nose, throat, mouth and tongue; chest (excluding breasts); respiratory; cardiovascular; lymph nodes, abdomen; skin, hair, nails; musculoskeletal; neurological.

## 6.6.4. Vital Signs

Assessment of vital signs will include measurement of resting blood pressure, pulse, respiratory rate, and temperature.

Blood pressure will be measured using the following standardized process:

- Subject should sit for  $\geq 5$  minutes with feet flat on the floor and measurement arm supported so that the midpoint of the manometer cuff is at heart level;
- Use a mercury sphygmomanometer or automatic blood pressure device with an appropriately sized cuff with the bladder centered over the brachial artery;
- Measure and record the blood pressure to the nearest 2 mmHg mark on the manometer or to the nearest whole number on an automatic device.

#### 6.6.5. Creatinine Clearance

Creatinine clearance will be calculated at all visits where blood is drawn for creatine. Creatinine clearance is calculated by the Cockcroft-Gault equation {Cockcroft et al 1976} using actual body weight (BW).

Male: 
$$CL_{cr} (mL/min) = [140 - age (years)] \times BW(kg)$$
  
 $72 \times S_{cr}$ 

Female: 
$$CL_{cr}$$
 (mL/min) = [140 - age (years)] × BW(kg) × 0.85  
72 ×  $S_{cr}$ 

 $S_{cr}$  = serum creatinine (mg/dL)

## 6.6.6. Child-Pugh Score

Child-Pugh score should be assessed at Screening, Week 12, post-treatment Week 4 and post-treatment Week 12. Please refer to Appendix 4 for more information regarding the Child-Pugh classification.

#### 6.6.7. 12-Lead ECG

Subjects will be required to rest in a supine position for  $\geq 5$  minutes prior to making a recording.

The investigator (or qualified designee) should review the ECG traces recorded in real time for clinically significant abnormalities. On treatment ECGs should be compared to the subject's baseline as part of routine safety monitoring.

## 6.6.8. HCV Viral RNA Sequencing/ Phenotyping (Archive)

Plasma samples will be collected at Baseline/Day 1 and each subsequent visit for HCV viral sequence analysis. At any unscheduled visit initiated for the purpose of confirming HCV virologic breakthrough, HCV viral sequence/phenotype plasma sample must also be collected. Unused samples may be archived.

Details regarding the collection, processing, and shipping of samples will be included in the lab manual.

## 6.6.9. Single Pharmacokinetic (PK) Sample

Single PK blood samples will be collected for all subjects at each on-treatment visit and archived for PK analysis of SOF (and metabolites) and VEL.

Details regarding the collection, processing, and shipping of samples will be included in the lab manual.

## 6.6.10. Pharmacogenomics Testing

An additional and distinct informed consent document will be provided to allow the Sponsor to obtain and test a subject's blood sample taken on Baseline/Day 1 for pharmacogenomics discovery research. If not obtained at Baseline/Day 1, the sample may be drawn at any time during the study. PPD

## 6.6.11. Sample Storage

## PPD

The stored blood samples may be used by the Sponsor or its research partners for HCV genotyping/phenotyping assays (as applicable) or their development, for retesting the amount of HCV in the blood, for measurement of antiviral drug levels in the blood, for future

testing to learn more about how the study drug has worked against HCV, to determine the durability of response, to identify changes in resistance conferring mutations, analysis of tumor biomarkers, or clinical laboratory testing to provide additional clinical data. No human genetic testing will be performed on these samples. At the conclusion of this study, these samples may be retained in storage by Gilead Sciences, Inc. for a period up to 15 years.

## 6.6.12. Pregnancy Testing

All females of childbearing potential will have urine pregnancy testing every 4 weeks during the dosing period and 30 days after last dose of study drug.

If a positive urine pregnancy test is reported, an immediate confirmation with Serum  $\beta$ -hCG is required.

## 7. ADVERSE EVENTS AND TOXICITY MANAGEMENT

# 7.1. Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events

### 7.1.1. Adverse Events

An adverse event (AE) is any untoward medical occurrence in a clinical study subject administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs may also include pre- or post-treatment complications that occur as a result of protocol specified procedures, lack of efficacy, overdose, drug abuse/misuse reports, or occupational exposure. Preexisting events that increase in severity or change in nature during or as a consequence of participation in the clinical study will also be considered AEs.

An AE does not include the following:

- Medical or surgical procedures such as surgery, endoscopy, tooth extraction, and transfusion. The condition that led to the procedure may be an adverse event and must be reported.
- Pre-existing diseases, conditions, or laboratory abnormalities present or detected before the screening visit that do not worsen
- Situations where an untoward medical occurrence has not occurred (e.g., hospitalization for elective surgery, social and/or convenience admissions)
- Overdose without clinical sequelae (see Section 7.6.1)
- Any medical condition or clinically significant laboratory abnormality with an onset date before the consent form is signed and not related to a protocol-associated procedure is not an AE. It is considered to be pre-existing and should be documented on the medical history CRF.

#### 7.1.2. Serious Adverse Events

A serious adverse event (SAE) is defined as an event that, at any dose, results in the following:

- Death
- Life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)

- In-patient hospitalization or prolongation of existing hospitalization (excluding those for study therapy or placement of an indwelling catheter, unless associated with other SAEs)
- Persistent or significant disability/incapacity
- A congenital anomaly/birth defect in the offspring of the subject who received investigational medicinal product
- A medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. Medical and scientific judgment must be exercised to determine whether such an event is a reportable under expedited reporting rules. Examples of medically important events include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; and development of drug dependency or drug abuse. For the avoidance of doubt, infections resulting from contaminated medicinal product will be considered a medically important event and subject to expedited reporting requirements.

# 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities without clinical significance are not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, and urinalysis) that require medical or surgical intervention or lead to IMP interruption, modification, or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE or SAE as described in Sections 7.1.1 and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (eg, anemia), not the laboratory result (ie, decreased hemoglobin).

For specific information on handling of clinical laboratory abnormalities in this study, please refer to Section 3.4.

#### 7.2. Assessment of Adverse Events and Serious Adverse Events

The investigator or qualified subinvestigator is responsible for assessing AEs and SAEs for causality and severity, and for final review and confirmation of accuracy of event information and assessments.

## 7.2.1. Assessment of Causality for Study Drugs and Procedures

The investigator or qualified subinvestigator is responsible for assessing the relationship to study drug using clinical judgment and the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the study drug. For SAEs, an alternative causality must be provided (eg, pre-existing condition, underlying disease, intercurrent illness, or concomitant medication).
- Yes: There is reasonable possibility that the event may have been caused by the study drug.

It should be emphasized that ineffective treatment should not be considered as causally related in the context of adverse event reporting.

The relationship to study procedures (eg, invasive procedures such as venipuncture or biopsy) should be assessed using the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the study procedure.
- Yes: The adverse event occurred as a result of protocol procedures, (eg., venipuncture)

## 7.2.2. Assessment of Severity

The severity grading of AEs will be assessed as Grade 1, 2, 3 or 4 using the GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities (Appendix 3). For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.

# 7.3. Investigator Requirements and Instructions for Reporting Adverse Events and Serious Adverse Events to Gilead

Requirements for collection prior to study drug initiation:

After informed consent, but prior to initiation of study medication, the following types of events should be reported on the case report form (eCRF): all SAEs and adverse events related to protocol-mandated procedures.

#### Adverse Events

- Following initiation of study medication, all AEs, regardless of cause or relationship, until 30 days after last administration of study drug must be collected/ reported to the eCRF database as instructed.
- All AEs should be followed up until resolution or until the adverse event is stable, if possible.
   Gilead Sciences may request that certain AEs be followed beyond the protocol defined follow up period.

#### Serious Adverse Events

- All SAEs, regardless of cause or relationship, that occurs after the subject first consents to
  participate in the study (ie, signing the informed consent) and throughout the duration of the
  study, including the protocol-required post-treatment follow-up period, must be reported to
  the eCRF database and Gilead Drug Safety and Public Health (DSPH) as instructed. This
  also includes any SAEs resulting from protocol-associated procedures performed after
  informed consent is signed.
- Any SAEs and deaths that occur after the post-treatment follow-up visit and within 30 days of the last dose of study drug, regardless of causality, should also be reported.

Investigators are not obligated to actively seek SAEs after the protocol defined follow up period; however, if the investigator learns of any SAEs that occur after study participation has concluded and the event is deemed relevant to the use of study drug, he/she should promptly document and report the event to Gilead DSPH.

• All AEs and SAEs will be recorded in the eCRF database within the timelines outlined in the eCRF completion guideline.

## Electronic Serious Adverse Event (eSAE) Reporting Process

- Site personnel record all SAE data in the eCRF database and from there transmit the SAE information to Gilead DSPH within 24 hours of the investigator's knowledge of the event. Detailed instructions can be found in the eCRF completion guidelines.
- If for any reason it is not possible to record the SAE information electronically, ie, the eCRF database is not functioning, record the SAE on the paper serious adverse event reporting form and submit within 24 hours to:

Gilead DSPH Email: Safety FC@gilead.com

Fax: +1 650-522-5477

- As soon as it is possible to do so, any SAE reported via paper must be transcribed into the eCRF Database according to instructions in the eCRF completion guidelines.
- If an SAE has been reported via a paper form because the eCRF database has been locked, no further action is necessary.
- For fatal or life-threatening events, copies of hospital case reports, autopsy reports, and other documents are also to be submitted by e-mail or fax when requested and applicable.
   Transmission of such documents should occur without personal subject identification, maintaining the traceability of a document to the subject identifiers.

- Additional information may be requested to ensure the timely completion of accurate safety reports.
- Any medications necessary for treatment of the SAE must be recorded onto the concomitant medication section of the subject's eCRF and the event description section of the SAE form.

## 7.4. Gilead Reporting Requirements

Depending on relevant local legislation or regulations, including the applicable US FDA Code of Federal Regulations, the EU Clinical Trials Directive (2001/20/EC) and relevant updates, and other country-specific legislation or regulations, Gilead may be required to expedite to worldwide regulatory agencies reports of SAEs, serious adverse drug reactions (SADRs), or suspected unexpected serious adverse reactions (SUSARs). In accordance with the EU Clinical Trials Directive (2001/20/EC), Gilead or a specified designee will notify worldwide regulatory agencies and the relevant IEC in concerned Member States of applicable SUSARs as outlined in current regulations.

Assessment of expectedness for SAEs will be determined by Gilead using reference safety information specified in the investigator's brochure or relevant local label as applicable.

All investigators will receive a safety letter notifying them of relevant SUSAR reports associated with any study IMP. The investigator should notify the IRB or IEC of SUSAR reports as soon as is practical, where this is required by local regulatory agencies, and in accordance with the local institutional policy.

## 7.5. Toxicity Management

## 7.5.1. Subject Stopping Rules

See Section 3.4 for individual subject stopping rules.

#### 7.6. Special Situations Reports

## 7.6.1. Definitions of Special Situations

Special situation reports include all reports of medication error, abuse, misuse, overdose, reports of adverse events associated with product complaints, and pregnancy reports regardless of an associated AE.

Medication error is any unintentional error in the prescribing, dispensing, or administration of a medicinal product while in the control of the health care provider, subject, or consumer.

Abuse is defined as persistent or sporadic intentional excessive use of a medicinal product by a subject.

Misuse is defined as any intentional and inappropriate use of a medicinal product that is not in accordance with the protocol instructions or the local prescribing information.

An overdose is defined as an accidental or intentional administration of a quantity of a medicinal product given per administration or cumulatively which is above the maximum recommended dose as per protocol or in the product labelling (as it applies to the daily dose of the subject in question). In cases of a discrepancy in drug accountability, overdose will be established only when it is clear that the subject has taken the excess dose(s). Overdose cannot be established when the subject cannot account for the discrepancy except in cases in which the investigator has reason to suspect that the subject has taken the additional dose(s).

Product complaint is defined as complaints arising from potential deviations in the manufacture, packaging, or distribution of the medicinal product.

## 7.6.2. Instructions for Reporting Special Situations

## 7.6.2.1. Instructions for Reporting Pregnancies

The investigator should report pregnancies in female study subjects that are identified after initiation of study medication and throughout the study, including the post study drug follow-up period, to the Gilead DSPH using the pregnancy report form within 24 hours of becoming aware of the pregnancy.

Refer to Section 7.3 and the eCRF completion guidelines for full instructions on the mechanism of pregnancy reporting.

The pregnancy itself is not considered an AE nor is an induced elective abortion to terminate a pregnancy without medical reasons.

Any premature termination of pregnancy (eg, a spontaneous abortion, an induced therapeutic abortion due to complications or other medical reasons) must be reported within 24 hours as an SAE. The underlying medical reason for this procedure should be recorded as the AE term.

A spontaneous abortion is always considered to be an SAE and will be reported as described in Sections 7.1.1 and 7.1.2. Furthermore, any SAE occurring as an adverse pregnancy outcome post study must be reported to Gilead DSPH.

The subject should receive appropriate monitoring and care until the conclusion of the pregnancy. The outcome should be reported to Gilead DSPH using the pregnancy outcome report form. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH. Gilead DSPH contact information is as follows:

Email: Safety FC@gilead.com and Fax: +1 (650) 522-5477.

Pregnancies of female partners of male study subjects exposed to Gilead or other study drugs must also be reported and relevant information should be submitted to Gilead DSPH using the pregnancy and pregnancy outcome forms within 24 hours. Monitoring of the subject should continue until the conclusion of the pregnancy. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH, fax number +1 650 522-5477 or email Safety FC@gilead.com.

Refer to Appendix 6 for Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements.

## 7.6.2.2. Reporting Other Special Situations

All other special situation reports must be reported on the special situations report form and forwarded to Gilead DSPH within 24 hours of the investigator becoming aware of the situation. These reports must consist of situations that involve study drug and/or Gilead concomitant medications, but do not apply to non-Gilead concomitant medications.

Special situations involving non-Gilead concomitant medications does not need to be reported on the special situations report form; however, for special situations that result in AEs due to a non-Gilead concomitant medication, the AE should be reported on the AE form.

Any inappropriate use of concomitant medications prohibited by this protocol should not be reported as "misuse," but may be more appropriately documented as a protocol deviation.

Refer to Section 7.6 and the eCRF completion guidelines for full instructions on the mechanism of special situations reporting.

All clinical sequelae in relation to these special situation reports will be reported as AEs or SAEs at the same time using the AE eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management, and outcome will be reported, when available.

## 8. STATISTICAL CONSIDERATIONS

## 8.1. Analysis Objectives and Endpoints

## 8.1.1. Analysis Objectives

The primary objectives of this study are as follows:

- To evaluate the efficacy of study treatment with sofosbuvir (SOF)/velpatasvir (VEL) for 12 weeks as measured by the proportion of subjects with sustained viral response 12 weeks after cessation of study treatment regimen (SVR12)
- To evaluate the safety and tolerability of the study treatment regimen

The secondary objectives of this study are as follows:

- To determine the proportion of subjects who attain SVR at 4 weeks after cessation of the study treatment regimen (SVR4)
- To evaluate the kinetics of circulating HCV RNA during the study treatment and after cessation of the study treatment regimen
- To evaluate the emergence of viral resistance to SOF and VEL during study treatment and after cessation of study treatment regimen

The exploratory objective of this study is as follows:



## 8.1.2. Primary Endpoint

The primary efficacy endpoint is SVR12 (HCV RNA < LLOQ 12 weeks after cessation of study treatment regimen) in the Full Analysis Set (FAS).

The primary safety endpoint is any AE that led to permanent discontinuation of study drug.

#### 8.1.3. Secondary Endpoints

The secondary efficacy endpoints include the proportion of subjects who attain sustained virologic response at 4 weeks after cessation of the study treatment regimen (SVR4); the proportion of subjects who have HCV RNA < LLOQ by visit while on study treatment; absolute and change from baseline/Day 1 in HCV RNA through Week 12; and the proportion of subjects with virologic failure.
#### 8.1.4. Other Endpoints of Interest

Additional efficacy evaluations may include ALT normalization.

#### 8.2. Analysis Conventions

All individual subject data will be listed as measured. All statistical summaries and analyses will be performed using SAS<sup>®</sup> software (SAS Institute, Cary, North Carolina, USA).

#### 8.2.1. Analysis Sets

# 8.2.1.1. Efficacy

The primary analysis set for efficacy analysis will be the FAS which include all enrolled subjects who received at least one dose of study drug.

#### 8.2.1.2. Safety

The primary analysis set for safety analyses will be the Safety Analysis Set which includes all subjects who took at least 1 dose of study drug.

Treatment-emergent data will be analyzed and defined as data collected from the first dose of the study drug through the last dose date of the study drug plus 30 days.

#### 8.2.1.3. Pharmacokinetics

The Pharmacokinetic (PK) Analysis Set include all subjects who took at least 1 dose of study drug and have at least 1 nonmissing postdose concentration value for the corresponding analyte in plasma. The analytes of interest may include SOF (and its metabolites GS-566500 and GS-331007), and VEL. The PK analysis set will be used for analyses of general PK

#### 8.3. Data Handling Conventions

Missing data can have an impact upon the interpretation of the trial data. Other than the endpoints discussed below, values for missing data will not be imputed.

For the analyses of categorical HCV RNA data, missing post-treatment HCV RNA data will have the missing data imputed. Missing on-treatment HCV RNA will have the missing data imputed up to the time of the last dose.

If a data point is missing and is preceded and followed in time by values that are "< LLOQ target not detected (TND)," then the missing data point will be set to "< LLOQ TND." If a data point is missing and preceded and followed by values that are "< LLOQ detected," or proceeded by "< LLOQ TND" and followed by "< LLOQ TND," or proceeded by "< LLOQ TND" and followed by "< LLOQ detected," then the missing value will be set to "< LLOQ detected." In these situations the data point will be termed a bracketed success; otherwise, the data point will be termed a bracketed failure (ie,  $\geq$  LLOQ detected). If a data point is missing and is not bracketed, the missing data point will also be termed a failure (ie,  $\geq$  LLOQ detected).

Where appropriate, safety data for subjects that did not complete the study will be included in summary statistics. For example,

- If a subject took at least 1 dose of study drug, the subject will be included in a summary of AEs according to the treatment received; otherwise, if the subject is not dosed, then they will be excluded from the summary.
- If safety laboratory results for a subject are missing for any reason at a time point, the subject will be excluded from the calculation of summary statistics for that time point. If the subject is missing a pre-dose value, then the subject will be excluded from the calculation of summary statistics for the predose value and the change from predose values.

Values for missing safety laboratory data will not be imputed; however, a missing Baseline/Day 1 result will be replaced with a screening result, if available. If no pretreatment laboratory value is available, the Baseline/Day 1 value will be assumed to be normal (i.e., no grade [Grade 0]) for the summary of graded laboratory abnormalities.

Values for missing vital signs data will not be imputed; however, a missing Baseline/Day 1 result will be replaced with a screening result, if available.

HCV RNA values below the LLOQ for the assay will be set to the lower limit minus 1 for calculation of summary statistics for the actual HCV RNA values and the change from Baseline/Day 1 values by study visit. The reported values will be provided in the HCV RNA listing.

For selected analyses of early time point data, HCV RNA data (IU/mL) may be transformed to the logarithmic (base 10) scale (log<sub>10</sub> IU/mL).

# 8.4. Demographic Data and Baseline Characteristics

Demographic and baseline measurements will be summarized using standard descriptive methods.

Demographic summaries will include age, sex, self-identified race and ethnicity.

Baseline characteristic data will include body mass index, absence or presence of cirrhosis, baseline HCV RNA level (log<sub>10</sub> IU/mL), HCV genotype, IL28B genotype, and additional endpoints as necessary.

#### 8.5. Efficacy Analysis

#### 8.5.1. Primary Analysis

The primary efficacy endpoint for this study will be the proportion of subjects with SVR12, defined as HCV RNA < LLOQ 12 weeks after cessation of the study treatment regimen) in the FAS population. Point estimate and 95% confidence interval (using the Clopper-Pearson method) of SVR12 will be computed.

# 8.5.2. Secondary Analyses

The proportion of subjects with HCV RNA below LLOQ over time (including SVR endpoints) will be presented in tabular and graphical form.

Descriptive summaries and listings will be provided for additional efficacy evaluations including serum HCV RNA values and change from baseline through Week 12, the proportion of subjects who experience virologic failure and ALT normalization.



Details on efficacy analyses will be described in the statistical analysis plan.

# 8.6. Safety Analysis

Safety will be evaluated by assessment of clinical laboratory tests, physical examinations, vital signs measurements and AEs will be documented at various time points during the study.

All safety data collected on or after the first dose of study drug administration up to 30 days after the last dose of study drug will be summarized.

# 8.6.1. Extent of Exposure

A subject's extent of exposure to study drug will be generated from the study drug administration page of the CRF. Exposure data will be summarized.

#### 8.6.2. Adverse Events

Clinical and laboratory adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), High-Level Group Term (HLGT), High-Level Term (HLT), Preferred Term (PT), and Lower-Level Term (LLT) will be attached to the clinical database.

Events will be summarized on the basis of the date of onset for the event. A treatment-emergent AE will be defined as any AE with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of the study drug; or any AE leading to premature discontinuation of the study drug.

Summaries (number and percentage of subjects) of treatment-emergent AEs (by SOC and PT) will be provided for:

All AEs

- AEs of Grade 3 or above
- AEs of Grade 2 or above
- All treatment-related AEs
- Treatment-related AEs of Grade 3 or above
- Treatment-related AEs of Grade 2 or above
- All SAEs
- All treatment-related SAEs
- All AEs leading to premature discontinuation of the study drug

All AEs collected during the study will be presented in data listings.

# 8.6.3. Laboratory Evaluations

Selected laboratory data will be summarized (n, mean, SD, median, Q1, Q3, minimum, and maximum) by study visit along with corresponding change from Baseline/Day 1.

Graded laboratory abnormalities will be defined using the laboratory toxicity grading scheme defined in Appendix 3 of this protocol. The incidence of treatment-emergent laboratory abnormalities, defined as values that increase by at least one toxicity grade from Baseline/Day 1 at any time post-baseline up to the date of last dose of study drug plus 30 days will be summarized.

Values for missing laboratory data will not be imputed; however, a missing Baseline/Day 1 data will be replaced with a screening result, if available. If no pre-treatment laboratory value is available, the Baseline/Day 1 value will be assumed to be normal (i.e., no grade [Grade 0] for the summary of graded laboratory [abnormalities]. If Baseline/Day 1 data are missing, then any post-baseline graded abnormality (ie, at least Grade 1) will be considered treatment emergent.

All laboratory abnormalities will be included in the listings of laboratory data.

# 8.6.4. Other Safety Evaluations

Individual data and change from baseline for vital signs measurements will be listed by subject and summarize by descriptive statistical summaries (n, mean, SD, median, Q1, Q3, minimum, and maximum).

# 8.7. Pharmacokinetic Analysis

Concentrations of SOF (and its metabolites GS-566500 and GS-331007) and VEL (GS-5816) in plasma may be determined using validated bioanalytical assays and listed.

# 8.8. Sample Size

Due to the exploratory nature of this study, no formal power calculations were used to determine sample size. The sample size is selected for practical reasons.

With a sample size of 80, a two-sided 95% exact confidence interval will extend at most 23% in length.

# 9. **RESPONSIBILITIES**

# 9.1. Investigator Responsibilities

#### 9.1.1. Good Clinical Practice

The investigator will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki (as amended in Edinburgh, Tokyo, Venice, Hong Kong, South Africa, Washington DC, Seoul and Brazil), International Conference on Harmonisation (ICH) guidelines, or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the study subject. These standards are consistent with the European Union Clinical Trials Directive 2001/20/EC and Good Clinical Practice Directive 2005/28/EC.

The investigator and all applicable subinvestigators will comply with 21 CFR, Part 54, 1998, providing documentation of their financial interest or arrangements with Gilead, or proprietary interests in the investigational drug under study. This documentation must be provided prior to the investigator's (and any subinvestigator's) participation in the study. The investigator and subinvestigator agree to notify Gilead of any change in reportable interests during the study and for 1 year following completion of the study. Study completion is defined as the date when the last subject completes the protocol-defined activities.

# 9.1.2. Independent Ethics Committee (IEC) Review and Approval

The investigator (or sponsor as appropriate according to local regulations) will submit this protocol, informed consent form, and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent) to an IEC. The investigator will not begin any study subject activities until approval from the IEC has been documented and provided as a letter to the investigator.

Before implementation, the investigator will submit to and receive documented approval from the IEC any modifications made to the protocol or any accompanying material to be provided to the subject after initial IEC approval, with the exception of those necessary to reduce immediate risk to study subjects.

#### 9.1.3. Informed Consent

The investigator is responsible for obtaining written informed consent from each individual participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study and before undertaking any study-related procedures. The investigator must use the most current IEC-approved consent form for documenting written informed consent. Each informed consent will be appropriately signed and dated by the subject and the person obtaining consent, and also by an impartial witness if required by IEC or local requirements. The consent form will inform subjects about pharmacogenomics testing and sample retention, and their right to receive clinically relevant pharmacogenomics analysis results.

# 9.1.4. Confidentiality

The investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only subject initials, date of birth, another unique identifier (as allowed by local law) and an identification code will be recorded on any form or biological sample submitted to the Sponsor, IEC or laboratory. Laboratory specimens must be uniquely labeled to protect subject identity while allowing the results to be recorded to the proper subject or in accordance with local regulations. NOTE: The investigator must keep a screening log showing codes, names, and addresses for all subjects screened and for all subjects enrolled in the trial. Subject data will be processed in accordance with all applicable regulations.

The investigator agrees that all information received from Gilead, including but not limited to the investigator brochure, this protocol, eCRF, the study drug, and any other study information, remain the sole and exclusive property of Gilead during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from Gilead. The investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

# 9.1.5. Study Files and Retention of Records

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following two categories: (1) investigator's study file, and (2) subject clinical source documents.

The investigator's study file will contain the protocol/amendments, eCRF and query forms, IRB [or] IEC and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data should include sequential notes containing at least the following information for each subject:

- Subject identification (name, date of birth, gender);
- Documentation that subject meets eligibility criteria, ie, history, physical examination, and confirmation of diagnosis (to support inclusion and exclusion criteria);
- Documentation of the reason(s) a consented subject is not enrolled
- Participation in study (including study number);
- Study discussed and date of informed consent;
- Dates of all visits;

- Documentation that protocol specific procedures were performed;
- Results of efficacy parameters, as required by the protocol;
- Start and end date (including dose regimen) of study drug, including dates of dispensing and return;
- Record of all adverse events and other safety parameters (start and end date, and including causality and severity);
- Concomitant medication (including start and end date, dose if relevant; dose changes);
- Date of study completion and reason for early discontinuation, if it occurs.

All clinical study documents must be retained by the investigator until at least 2 years or according to local laws, whichever is longer, after the last approval of a marketing application in an ICH region (ie, United States, Europe, or Japan) and until there are no pending or planned marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if specified by regulatory requirements, by local regulations, or by an agreement with Gilead. The investigator must notify Gilead before destroying any clinical study records.

Should the investigator wish to assign the study records to another party or move them to another location, Gilead must be notified in advance.

If the investigator cannot provide for this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the investigator and Gilead to store these records securely away from the site so that they can be returned sealed to the investigator in case of an inspection. When source documents are required for the continued care of the subject, appropriate copies should be made for storage away from the site.

Biological samples at the conclusion of this study may be retained in storage by the Sponsor for a period up to 15 years for purposes of this study.

#### 9.1.6. Case Report Forms

For each subject consented, an eCRF will be completed by an authorized study staff member whose training for this function is documented according to study procedures. The eCRF should be completed on the day of the subject visit to enable the sponsor to perform central monitoring of safety data. The Eligibility Criteria eCRF should be completed only after all data related to eligibility have been received. Subsequent to data entry, a study monitor will perform source data verification within the electronic data capture (EDC) system. Original entries as well as any changes to data fields will be stored in the audit trail of the system. Prior to database lock (or any interim time points as described in the clinical data management plan), the investigator will use his/her log in credentials to confirm that the forms have been reviewed, and that the entries

accurately reflect the information in the source documents. The eCRF capture the data required per the protocol schedule of events and procedures. System-generated or manual queries will be issued to the investigative site staff as data discrepancies are identified by the monitor or internal Gilead staff, who routinely review the data for completeness, correctness, and consistency. The site coordinator is responsible for responding to the queries in a timely manner, within the system, either by confirming the data as correct or updating the original entry, and providing the reason for the update (e.g. data entry error). At the conclusion of the trial, Gilead will provide the site with a read-only archive copy of the data entered by that site. This archive must be stored in accordance with the records retention requirements outlined in Section 9.1.5

# 9.1.7. Study Drug Return and Disposal

Gilead recommends that used and unused study drugs be returned to the shipping facility from which it came for eventual destruction. The study monitor will provide instructions for return. If return is not possible, the study monitor will evaluate each study center's study drug disposal procedures and provide appropriate instruction for destruction of unused study drugs. If the site has an appropriate standard operating procedure (SOP) for drug destruction as determined by Gilead QA, the site may destroy used (empty or partially empty) and unused study drugs in accordance with that site's approved SOP. A copy of the site's approved SOP will be obtained for central files.

If study drug is destroyed on site, the investigator must maintain accurate records for all study drug destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and the person who disposed of the study drug. Upon study completion, copies of the study drug accountability records must be filed at the site. Another copy will be returned to Gilead.

The site monitor will review study drug supplies and associated records at periodic intervals.

# 9.1.8. Inspections

The investigator will make available all source documents and other records for this trial to Gilead's appointed study monitors, to IRB/IECs, or to regulatory authority or health authority inspectors.

# 9.1.9. Protocol Compliance

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.

# 9.2. Sponsor Responsibilities

#### 9.2.1. Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by Gilead. All substantial protocol modifications will be reviewed and approved by

the local competent authority in accordance with local requirements prior to implementation of any changes. In addition, the investigator must submit all protocol modifications to the IRB/IEC in accordance with local requirements and receive documented IRB/IEC approval before modifications can be implemented.

# 9.2.2. Study Report and Publications

A clinical study report (CSR) will be prepared and provided to the regulatory agency(ies). Gilead will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

Investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

- the results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form or
- the study has been completed at all study sites for at least 2 years

The investigator will submit to Gilead any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation.

No such communication, presentation, or publication will include Gilead's confidential information (see Section 9.1.4).

The investigator will comply with Gilead's request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

# 9.3. Joint Investigator/Sponsor Responsibilities

#### 9.3.1. Payment Reporting

Investigators and their study staff may be asked to provide services performed under this protocol, e.g. attendance at Investigator's Meetings. If required under the applicable statutory and regulatory requirements, Gilead will capture and disclose to Federal and State agencies any expenses paid or reimbursed for such services, including any clinical trial payments, meal, travel expenses or reimbursements, consulting fees, and any other transfer of value.

# 9.3.2. Access to Information for Monitoring

In accordance with regulations and guidelines, the study monitor must have direct access to the investigator's source documentation in order to verify the accuracy of the data recorded in the eCRF.

The monitor is responsible for routine review of the eCRF at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records needed to verify the entries on the eCRF. The investigator agrees to cooperate with the monitor to ensure that any problems detected through any type of monitoring (central, on site) are resolved.

# 9.3.3. Access to Information for Auditing or Inspections

Representatives of regulatory authorities or of Gilead may conduct inspections or audits of the clinical study. If the investigator is notified of an inspection by a regulatory authority the investigator agrees to notify the Gilead medical monitor immediately. The investigator agrees to provide to representatives of a regulatory agency or Gilead access to records, facilities, and personnel for the effective conduct of any inspection or audit.

#### 9.3.4. Study Discontinuation

The sponsor reserves the right to terminate the study at any time. Should this be necessary, the sponsor will arrange discontinuation procedures and notify the appropriate regulatory authority(ies), IRBs, and/or IECs. In terminating the study, Gilead will assure that adequate consideration is given to the protection of the subjects' interests.

# 10. REFERENCES

- Afdhal N, Reddy KR, Nelson DR, Lawitz E, Gordon SC, Schiff E, et al. Ledipasvir and sofosbuvir for previously treated HCV genotype 1 infection. N Engl J Med 2014a;370 (16):1483-93.
- Afdhal N, Zeuzem S, Kwo P, Chojkier M, Gitlin N, Puoti M, et al. Ledipasvir and sofosbuvir for untreated HCV genotype 1 infection. N Engl J Med 2014b;370 (20):1889-98.
- Andrews E, Damle BD, Fang A, Foster G, Crownover P, LaBadie R, et al. Pharmacokinetics and tolerability of voriconazole and a combination oral contraceptive co-administered in healthy female subjects. Br J Clin Pharmacol 2008;65 (4):531-9.
- Barditch-Crovo P, Trapnell CB, Ette E, Zacur HA, Coresh J, Rocco LE, et al. The effects of rifampin and rifabutin on the pharmacokinetics and pharmacodynamics of a combination oral contraceptive. Clin Pharmacol Ther 1999;65 (4):428-38.
- Berenguer M. Natural history of recurrent hepatitis C. Liver Transpl 2002;8 (10 Suppl 1):S14-8.
- Berenguer M, Ferrell L, Watson J, Prieto M, Kim M, Rayon M, et al. HCV-related fibrosis progression following liver transplantation: increase in recent years. J Hepatol 2000;32 (4):673-84.
- Biggins SW, Bambha KM, Terrault NA, Inadomi J, Shiboski S, Dodge JL, et al. Projected future increase in aging hepatitis C virus-infected liver transplant candidates: a potential effect of hepatocellular carcinoma. Liver Transpl 2012;18 (12):1471-8.
- Calmus Y, Duvoux C, Pageaux G, Wolf P, Rostaing L, Vanlemmens C, et al. Treatment of recurrent HCV infection following liver transplantation: results of a multicenter, randomized, versus placebo, trial of ribavirin alone as maintenance therapy after one year of PegIFNalpha-2a plus ribavirin. J Hepatol 2012;57 (3):564-71.
- Campos-Varela I, Lai JC, Verna EC, O'Leary JG, Todd Stravitz R, Forman LM, et al. Hepatitis C genotype influences post-liver transplant outcomes. Transplantation 2015;99 (4):835-40.
- Carrion JA, Navasa M, Garcia-Retortillo M, Garcia-Pagan JC, Crespo G, Bruguera M, et al. Efficacy of antiviral therapy on hepatitis C recurrence after liver transplantation: a randomized controlled study. Gastroenterology 2007;132 (5):1746-56.
- Charlton M, Everson GT, Flamm SL, Kumar P, Landis C, Brown Jr RS, et al. Ledipasvir and Sofosbuvir Plus Ribavirin for Treatment of HCV Infection in Patients with Advanced Liver Disease. Gastroenterology 2015:649-59.
- Charlton M, Gane E, Manns MP, Brown RS, Jr., Curry MP, Kwo PY, et al. Sofosbuvir and Ribavirin for Treatment of Compensated Recurrent Hepatitis C Virus Infection After Liver Transplantation. Gastroenterology 2014.
- Charlton M, Ruppert K, Belle SH, Bass N, Schafer D, Wiesner RH, et al. Long-term results and modeling to predict outcomes in recipients with HCV infection: results of the NIDDK liver transplantation database. Liver Transpl 2004;10 (9):1120-30.
- Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41.
- Crespo G, Marino Z, Navasa M, Forns X. Viral hepatitis in liver transplantation. Gastroenterology 2012;142 (6):1373-83 e1.

- Crippin JS, McCashland T, Terrault N, Sheiner P, Charlton MR. A pilot study of the tolerability and efficacy of antiviral therapy in hepatitis C virus-infected patients awaiting liver transplantation. Liver Transpl 2002;8 (4):350-5.
- Feray C, Samuel D, Thiers V, Gigou M, Pichon F, Bismuth A, et al. Reinfection of liver graft by hepatitis C virus after liver transplantation. J Clin Invest 1992;89 (4):1361-5.
- Firpi RJ, Clark V, Soldevila-Pico C, Morelli G, Cabrera R, Levy C, et al. The natural history of hepatitis C cirrhosis after liver transplantation. Liver Transpl 2009;15 (9):1063-71.
- Forman LM, Lewis JD, Berlin JA, Feldman HI, Lucey MR. The association between hepatitis C infection and survival after orthotopic liver transplantation. Gastroenterology 2002;122 (4):889-96.
- Forns X, Garcia-Retortillo M, Serrano T, Feliu A, Suarez F, de la Mata M, et al. Antiviral therapy of patients with decompensated cirrhosis to prevent recurrence of hepatitis C after liver transplantation. J Hepatol 2003;39 (3):389-96.
- Gane EJ. The natural history of recurrent hepatitis C and what influences this. Liver Transpl 2008;14 Suppl 2:S36-44.
- Gilead Sciences Inc. SOVALDI® (sofosbuvir) tablets, for oral use. US Prescribing Information. Foster City, CA. December 2013:
- Gilead Sciences Inc. HARVONI® (ledipasvir and sofosbuvir) tablets, for oral use. US Prescribing Information. Foster City, CA. Revised November 2015:
- Gilead Sciences International Limited. HARVONI (ledipasvir/sofosbuvir) 90 mg/400 mg film-coated tablet. Summary of Product Characteristics. Cambridge, UK. 2014:
- Gower E, Estes C, Blach S, Razavi-Shearer K, Razavi H. Global epidemiology and genotype distribution of the hepatitis C virus infection. J Hepatol 2014.
- Janssen Pharmaceuticals Inc. INTELENCE® (etravirine) tablets for oral use. US Prescribing Information. 2008 Titusville NJ. Revised February 2013.
- Kim JM, Lee KW, Song GW, Jung BH, Lee HW, Yi NJ, et al. Outcomes for patients with HCV after liver transplantation in Korea: a multicenter study. Ann Surg Treat Res 2016;90 (1):36-42.
- Kowdley KV, Gordon SC, Reddy KR, Rossaro L, Bernstein DE, Lawitz E, et al. Ledipasvir and sofosbuvir for 8 or 12 weeks for chronic HCV without cirrhosis. N Engl J Med 2014;370 (20):1879-88.
- Lim SG. Chronic hepatitis C genotype 1 treatment roadmap for resource constrained settings. World J Gastroenterol 2015;21 (6):1972-81.
- Manns M, Samuel D, Gane EJ, Mutimer D, McCaughan G, Buti M, et al. Ledipasvir and sofosbuvir plus ribavirin in patients with genotype 1 or 4 hepatitis C virus infection and advanced liver disease: a multicentre, open-label, randomised, phase 2 trial. Lancet Infect Dis 2016.
- Marks KM, Jacobson IM. The first wave: HCV NS3 protease inhibitors telaprevir and boceprevir. Antivir Ther 2012;17 (6 Pt B):1119-31.
- Prieto M, Berenguer M, Rayon JM, Cordoba J, Arguello L, Carrasco D, et al. High incidence of allograft cirrhosis in hepatitis C virus genotype 1b infection following transplantation: relationship with rejection episodes. Hepatology 1999;29 (1):250-6.
- Quest Diagnostics. FSH and LH Reference Ranges. 2013a:
- Quest Diagnostics. Progesterone, LC/MS/MS Reference Ranges. 2013b:

- Samuel D, Bizollon T, Feray C, Roche B, Ahmed SN, Lemonnier C, et al. Interferon-alpha 2b plus ribavirin in patients with chronic hepatitis C after liver transplantation: a randomized study. Gastroenterology 2003;124 (3):642-50.
- Terrault NA. Hepatitis C therapy before and after liver transplantation. Liver Transpl 2008;14 Suppl 2:S58-66.
- Wang CS, Ko HH, Yoshida EM, Marra CA, Richardson K. Interferon-based combination antiviral therapy for hepatitis C virus after liver transplantation: a review and quantitative analysis. Am J Transplant 2006;6 (7):1586-99.
- Wiesner RH, Sorrell M, Villamil F. Report of the first International Liver Transplantation Society expert panel consensus conference on liver transplantation and hepatitis C. Liver Transpl 2003;9 (11):S1-9.
- World Health Organization (WHO). Hepatitis C Fact sheet N°164. Available at: http://www.who.int/mediacentre/factsheets/fs164/en/#. Accessed: 20 March. 2014.
- Wright TL, Donegan E, Hsu HH, Ferrell L, Lake JR, Kim M, et al. Recurrent and acquired hepatitis C viral infection in liver transplant recipients. Gastroenterology 1992;103 (1):317-22.
- Zekry A, Whiting P, Crawford DH, Angus PW, Jeffrey GP, Padbury RT, et al. Liver transplantation for HCV-associated liver cirrhosis: predictors of outcomes in a population with significant genotype 3 and 4 distribution. Liver Transpl 2003;9 (4):339-47.

# 11. APPENDICES

| Appendix 1. | Investigator Signature Page |
|---|---|
| Appendix 2. | Study Procedures Table |
| Appendix 3. | GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities |
| Appendix 4. | Child-Pugh-Turcotte Classification of the severity of cirrhosisa |
| Appendix 5. | Banff Criteria* |
| Appendix 6. | Pregnancy Precautions, Definition for Female of Childbearing Potential, and |
| | Contraceptive Requirements |

Appendix 1.

**Investigator Signature Page** 

# GILEAD SCIENCES, INC. 333 LAKESIDE DRIVE FOSTER CITY, CA 94404, USA

# STUDY ACKNOWLEDGEMENT

A Phase 2. Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of

| Sofosbuvir/Velpatasvir Fixed Dose Combination<br>have received a Li | |
|---|---|
| GS-US-342-2104, Origin | nal 19 February 2016 |
| This protocol has been approved by Gilead Science this approval. Drian Mc Walb Brian McNabb, MD | PPD |
| | Signature |
| 19- Feb- 2016 Date | |
| INVESTIGATOR | STATEMENT |
| I have read the protocol, including all appendices, a details for me and my staff to conduct this study as outlined herein and will make a reasonable effort to designated. I will provide all study personnel under my supervisinformation provided by Gilead Sciences, Inc. I will that they are fully informed about the drugs and the | described. I will conduct this study as complete the study within the time sion copies of the protocol and access to all discuss this material with them to ensure study. |
| Principal Investigator Name (Printed) | Signature |
| Date | Site Number |

**Appendix 2. Study Procedures Table** 

| | | | | On-treatm | nent Week | | Post-treat | ment Week |
|---|---|---|---|---|---|---|---|---|
| | Screen | Baseline/Day 1 <sup>b</sup> | 2 | 4 | 8 | 12/ET | 4 | 12 |
| Clinical Assessments | • | | | • | | | | |
| Informed Consent | X | | | | | | | |
| Determine Eligibility | X | X | | | | | | |
| Medical History | X | | | | | | | |
| Physical Examination | X | X | | | | X | X | X |
| Height | X | | | | | | | |
| Weight | X | X | | | | X | | |
| Vital Signs | X | X | X | X | X | X | X | X |
| 12-Lead ECG | X | | | | | | | |
| CPT score | X | | | | | X | X | X |
| Adverse Events and<br>Concomitant Medications | X | X | X | X | X | X | X | X |
| Pregnancy Prevention<br>Counseling | | X | | X | X | X | X | |
| Review of Study<br>Medication Compliance | | | X | X | X | X | | |
| Study Drug Dispensing <sup>a</sup> | | X | | X | X | | | |
| Laboratory Assessments | • | | | • | | • | • | • |
| Hematology, Chemistry <sup>g</sup> | X | X | X | X | X | X | X | X |
| Coagulation Tests | X | X | | | | X | | |
| Urinalysis | X | X | | | | X | | |
| HCV RNA <sup>c</sup> | X | X | X | X | X | X | X | $X^{f}$ |

| | | | | On-treatn | nent Week | | Post-treati | ment Week |
|---|---|---|---|---|---|---|---|---|
| | Screen | Baseline/Day 1 <sup>b</sup> | 2 | 4 | 8 | 12/ET | 4 | 12 |
| Viral Sequencing <sup>c</sup> | | X | X | X | X | X | X | X <sup>f</sup> |
| Single PK | | | X | X | X | X | | |
| Serum β-hCG or Urine<br>Pregnancy Test <sup>d</sup> | X | X | | X | X | X | X | |
| Urine Drug Screen | X | | | | | | | |
| HCV Genotyping, IL28B | X | | | | | | | |
| HCV, HIV, HBV Serology | X | | | | | | | |
| HbA1c, Fibrotest® | X | | | | | | | |
| Archive Sample <sup>e</sup> | | X | | | | X | | |
| Pharmacogenomic Sample <sup>e</sup> | | X | | | | | | |

- a The IWRS will provide direction on the specifics of each subject's study drug dispensing
- b Baseline/Day 1 assessments must be performed prior to dosing
- c Viral sequencing samples for virologic sequencing required at baseline and after any visit where a previously undetectable HCV RNA becomes detectable
- d Serum β-hCG pregnancy test performed at screening and for confirmation of positive urine pregnancy test.
- Only for subjects who have provided consent for this sample and testing.
- f Only for subjects with HCV RNA ≥LLOQ at post-treatment week 12 visit will be asked to return after for a confirmatory visit where additional samples are collected.
- g CrCl will be calculated at all visits where a blood sample is drawn

**Appendix 3.** GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities

Antiviral Toxicity Grading Scale Version: 01 April 2015

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin<br>HIV POSITIVE<br>Adult and Pediatric ≥ 57 Days | 8.5 to 10.0 g/dL<br>85 to 100 g/L | 7.5 to < 8.5 g/dL<br>75 to < 85 g/L | 6.5 to < 7.5 g/dL<br>65 to < 75 g/L | < 6.5 g/dL<br>< 65 g/L |
| HIV NEGATIVE<br>Adult and Pediatric ≥ 57 Days | 10.0 to 10.9 g/dL<br>100 to 109 g/L<br>OR<br>Any decrease from Baseline<br>2.5 to < 3.5 g/dL<br>25 to < 35 g/L | 9.0 to < 10.0 g/dL $90 to < 100 g/L$ $OR$ Any decrease from Baseline $3.5 to < 4.5 g/dL$ $35 to < 45 g/L$ | $7.0 \text{ to} < 9.0 \text{ g/dL}$ $70 \text{ to} < 90 \text{ g/L}$ $OR$ Any decrease from Baseline $\geq 4.5 \text{ g/dL}$ $\geq 45 \text{ g/L}$ | < 7.0 g/dL<br>< 70 g/L |
| Infant, 36–56 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 8.5 to 9.4 g/dL<br>85 to 94 g/L | 7.0 to < 8.5 g/dL<br>70 to < 85 g/L | 6.0 to < 7.0 g/dL<br>60 to < 70 g/L | < 6.0 g/dL<br>< 60 g/L |
| Infant, 22–35 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 9.5 to 10.5 g/dL<br>95 to 105 g/L | 8.0 to < 9.5 g/dL<br>80 to < 95 g/L | 7.0 to < 8.0 g/dL<br>70 to < 80 g/L | < 7.0 g/dL<br>< 70 g/L |
| Infant, 1–21 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 12.0 to 13.0 g/dL<br>120 to 130 g/L | 10.0 to < 12.0 g/dL<br>100 to < 120 g/L | 9.0 to < 10.0 g/dL<br>90 to < 100 g/L | < 9.0 g/dL<br>< 90 g/L |
| Absolute Neutrophil Count (ANC) Adult and Pediatric, ≥ 7 Months# | 1000 to 1300/mm <sup>3</sup> 1.00 to 1.30 GI/L | 750 to < 1000/mm <sup>3</sup><br>0.75 to < 1.00 GI/L | 500 to < 750/mm <sup>3</sup><br>0.50 to < 0.75 GI/L | < 500/mm <sup>3</sup><br>< 0.50 GI/L |
| Absolute CD4+ Count<br>HIV NEGATIVE ONLY<br>Adult and Pediatric > 13 Years | 300 to 400/mm <sup>3</sup><br>300 to 400/μL | $200 \text{ to} < 300/\text{mm}^3$<br>$200 \text{ to} < 300/\mu\text{L}$ | 100 to < 200/mm <sup>3</sup><br>100 to < 200/μL | $< 100/mm^3$<br>$< 100/\mu L$ |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Absolute Lymphocyte Count<br>HIV NEGATIVE ONLY<br>Adult and Pediatric > 13 Years | 600 to 650/mm <sup>3</sup><br>0.60 to 0.65 GI/L | 500 to < 600/mm <sup>3</sup><br>0.50 to < 0.60 GI/L | 350 to < 500/mm <sup>3</sup><br>0.35 to < 0.50 GI/L | < 350/mm <sup>3</sup><br>< 0.35 GI/L |
| Platelets | 100,000 to < 125,000/mm <sup>3</sup><br>100 to < 125 GI/L | 50,000 to < 100,000/mm <sup>3</sup><br>50 to < 100 GI/L | 25,000 to < 50,000/mm <sup>3</sup><br>25 to < 50 GI/L | < 25,000/mm <sup>3</sup><br>< 25 GI/L |
| WBCs | 2000/mm <sup>3</sup> to 2500/mm <sup>3</sup> | 1,500 to < 2,000/mm <sup>3</sup> | 1000 to < 1,500/mm <sup>3</sup> | < 1000/mm <sup>3</sup> |
| | 2.00 GI/L to 2.50 GI/L | 1.50 to < 2.00 GI/L | 1.00 to < 1.50 GI/L | < 1.00 GI/L |
| Hypofibrinogenemia | 100 to 200 mg/dL | 75 to < 100 mg/dL | 50 to < 75 mg/dL | < 50 mg/dL |
| | 1.00 to 2.00 g/L | 0.75 to < 1.00 g/L | 0.50 to < 0.75 g/L | < 0.50 g/L |
| Hyperfibrinogenemia | > ULN to 600 mg/dL | > 600 mg/dL | _ | _ |
| | > ULN to 6.0 g/L | > 6.0 g/L | _ | _ |
| Fibrin Split Product | 20 to 40 μg/mL | > 40 to 50 μg/mL | > 50 to 60 μg/mL | > 60 μg/mL |
| | 20 to 40 mg/L | > 40 to 50 mg/L | > 50 to 60 mg/L | > 60 mg/L |
| Prothrombin Time (PT) | > 1.00 to 1.25 × ULN | > 1.25 to 1.50 × ULN | > 1.50 to 3.00 × ULN | > 3.00 × ULN |
| International Normalized Ratio of prothrombin time (INR) | 1.1 to 1.5 x ULN | >1.5 to 2.0 x ULN | >2.0 to 3.0 x ULN | >3.0 x ULN |
| Activated Partial<br>Thromboplastin Time (APTT) | > 1.00 to 1.66 × ULN | > 1.66 to 2.33 × ULN | > 2.33 to 3.00 × ULN | > 3.00 × ULN |
| Methemoglobin | 5.0 to 10.0% | > 10.0 to 15.0% | > 15.0 to 20.0% | > 20.0% |

<sup>#</sup> An overlap between the Grade 1 scale and the Lab's normal range for absolute neutrophils may result for pediatric subjects. Please follow the Gilead convention of grading any result within the LLN and ULN a 0.

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 to <lln l<="" meq="" td=""><td>125 to &lt; 130 mEq/L</td><td>121 to &lt; 125 mEq/L</td><td>&lt; 121 mEq/L</td></lln> | 125 to < 130 mEq/L | 121 to < 125 mEq/L | < 121 mEq/L |
| | 130 to <lln l<="" mmol="" td=""><td>125 to &lt; 130 mmol/L</td><td>121 to &lt; 125 mmol/L</td><td>&lt; 121 mmol/L</td></lln> | 125 to < 130 mmol/L | 121 to < 125 mmol/L | < 121 mmol/L |
| Hypernatremia | >ULN to 150 mEq/L | > 150 to 154 mEq/L | > 154 to 159 mEq/L | > 159 mEq/L |
| | >ULN to 150 mmol/L | > 150 to 154 mmol/L | > 154 to 159 mmol/L | > 159 mmol/L |
| Hypokalemia | 3.0 to <lln l<="" meq="" td=""><td>2.5 to &lt; 3.0 mEq/L</td><td>2.0 to &lt; 2.5 mEq/L</td><td>&lt; 2.0 mEq/L</td></lln> | 2.5 to < 3.0 mEq/L | 2.0 to < 2.5 mEq/L | < 2.0 mEq/L |
| Adult and Pediatric ≥ 1 Year | 3.0 to <lln l<="" mmol="" td=""><td>2.5 to &lt; 3.0 mmol/L</td><td>2.0 to &lt; 2.5 mmol/L</td><td>&lt; 2.0 mmol/L</td></lln> | 2.5 to < 3.0 mmol/L | 2.0 to < 2.5 mmol/L | < 2.0 mmol/L |
| Infant <1 Year | 3.0 to 3.4 mEq/L<br>3.0 to 3.4 mmol/L | 2.5 to < 3.0 mEq/L<br>2.5 to <3.0 mmolL | 2.0 to < 2.5 mEq/L<br>2.0 to <2.5 mmolL | < 2.0 mEq/L<br><2.0 mmolL |
| Hyperkalemia<br>Adult and Pediatric<br>≥ 1 Year | 5.6 to 6.0 mEq/L<br>5.6 to 6.0 mmol/L | > 6.0 to 6.5 mEq/L<br>> 6.0 to 6.5 mmol/L | > 6.5 to 7.0 mEq/L<br>> 6.5 to 7.0 mmol/L | > 7.0 mEq/L<br>> 7.0 mmol/L |
| Infant <1 Year | >ULN to 6.0 mEq/L<br>>ULN to 6.0 mmol/L | > 6.0 to 6.5 mEq/L<br>> 6.0 to 6.5 mmol/L | > 6.5 to 7.0 mEq/L<br>> 6.5 to 7.0 mmol/L | > 7.0 mEq/L<br>> 7.0 mmol/L |
| Hypoglycemia<br>Adult and Pediatric<br>≥ 1 Month | 55 to 64 mg/dL<br>3.03 to 3.58 mmol/L | 40 to < 55 mg/dL<br>2.20 to < 3.03 mmol/L | 30 to < 40 mg/dL<br>1.64 to < 2.20 mmol/L | < 30 mg/dL<br>< 1.64 mmol/L |
| Infant, < 1 Month | 50 to 54 mg/dL<br>2.8 to 3.0 mmol/L | 40 to < 50 mg/dL<br>2.2 to < 2.8 mmol/L | 30 to < 40 mg/dL<br>1.7 to < 2.2 mmol/L | < 30 mg/dL<br>< 1.7 mmol/L |
| Hyperglycemia, Nonfasting | 116 to 160 mg/dL | > 160 to 250 mg/dL | > 250 to 500 mg/dL | > 500 mg/dL |
| | 6.42 to 8.91 mmol/L | > 8.91 to 13.90 mmol/L | > 13.90 to 27.79 mmol/L | > 27.79 mmol/L |
| Hyperglycemia, Fasting | 110 to 125 mg/dL<br>6.08 to 6.96 mmol/L | >125 to 250 mg/dL<br>>6.96 to 13.90 mmol/L | >250 to 500 mg/dL<br>>13.90 to 27.79 mmol/L | >500 mg/dL<br>>27.79 mmol/L |

| | CHEMISTRY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypocalcemia<br>(corrected for albumin if<br>appropriate*)<br>Adult and Pediatric<br>≥2 Years | 7.8 <lln dl<br="" mg="">1.94 to <lln l<="" mmol="" td=""><td>7.0 to &lt; 7.8 mg/dL<br/>1.74 to &lt; 1.94 mmol/L</td><td>6.1 to &lt; 7.0 mg/dL<br/>1.51 to &lt; 1.74 mmol/L</td><td>&lt; 6.1 mg/dL<br/>&lt; 1.51 mmol/L</td></lln></lln> | 7.0 to < 7.8 mg/dL<br>1.74 to < 1.94 mmol/L | 6.1 to < 7.0 mg/dL<br>1.51 to < 1.74 mmol/L | < 6.1 mg/dL<br>< 1.51 mmol/L |
| Pediatric ≥7 days -2 Years | 7.8 to 8.4 mg/dL | 7.0 to <7.8 mg/dL | 6.1 to <7.0 mg/dL | < 6.1 mg/dL |
| | 1.94 to 2.10 mmol/L | 1.74 to <1.94 mmolL | 1.51 to < 1.74 mmolL | < 1.51 mmol/L |
| Infant, < 7 Days | 6.5 to 7.5 mg/dL | 6.0 to < 6.5 mg/dL | 5.5 to < 6.0 mg/dL | < 5.5 mg/dL |
| | 1.61 to 1.88 mmol/L | 1.49 to < 1.61 mmol/L | 1.36 to < 1.49 mmol/L | < 1.36 mmol/L |
| Hypercalcemia (corrected for albumin if appropriate*) Adult and Pediatric ≥ 7 Days | >ULN to 11.5 mg/dL | > 11.5 to 12.5 mg/dL | > 12.5 to 13.5 mg/dL | > 13.5 mg/dL |
| | >ULN to 2.88 mmol/L | > 2.88 to 3.13 mmol/L | > 3.13 to 3.38 mmol/L | > 3.38 mmol/L |
| Infant, < 7 Days | 11.5 to 12.4 mg/dL | > 12.4 to 12.9 mg/dL | > 12.9 to 13.5 mg/dL | > 13.5 mg/dL |
| | 2.86 to 3.10 mmol/L | > 3.10 to 3.23 mmol/L | > 3.23 to 3.38 mmol/L | > 3.38 mmol/L |
| Hypocalcemia (ionized) | 3.0 mg/dL to < LLN | 2.5 to < 3.0 mg/dL | 2.0 to < 2.5 mg/dL | < 2.0 mg/dL |
| | 0.74 mmol/L to < LLN | 0.62 to < 0.74 mmol/L | 0.49 to < 0.62 mmol/L | < 0.49 mmol/L |
| Hypercalcemia (ionized) | > ULN to 6.0 mg/dL | > 6.0 to 6.5 mg/dL | > 6.5 to 7.0 mg/dL | > 7.0 mg/dL |
| | > ULN to 1.50 mmol/L | > 1.50 to 1.63 mmol/L | > 1.63 to 1.75 mmol/L | > 1.75 mmol/L |
| Hypomagnesemia | 1.40 to <lln dl<="" mg="" td=""><td>1.04 to &lt; 1.40 mg/dL</td><td>0.67 to &lt; 1.04 mg/dL</td><td>&lt; 0.67 mg/dL</td></lln> | 1.04 to < 1.40 mg/dL | 0.67 to < 1.04 mg/dL | < 0.67 mg/dL |
| | 1.2 to <lln l<="" meq="" td=""><td>0.9 to &lt; 1.2 mEq/L</td><td>0.6 to &lt; 0.9 mEq/L</td><td>&lt; 0.6 mEq/L</td></lln> | 0.9 to < 1.2 mEq/L | 0.6 to < 0.9 mEq/L | < 0.6 mEq/L |
| | 0.58 to <lln l<="" mmol="" td=""><td>0.43 to &lt; 0.58 mmol/L</td><td>0.28 to &lt; 0.43 mmol/L</td><td>&lt; 0.28 mmol/L</td></lln> | 0.43 to < 0.58 mmol/L | 0.28 to < 0.43 mmol/L | < 0.28 mmol/L |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypophosphatemia<br>Adult and Pediatric<br>> 14 Years | 2.0 to < LLN mg/dL<br>0.63 to < LLN mmol/L | 1.5 to < 2.0 mg/dL<br>0.47 to < 0.63 mmol/L | 1.0 to < 1.5 mg/dL<br>0.31 to < 0.47 mmol/L | < 1.0 mg/dL<br>< 0.31 mmol/L |
| Pediatric 1 Year–14 Years | 3.0 to <lln dl<br="" mg="">0.96 to <lln l<="" mmol="" td=""><td>2.5 to &lt; 3.0 mg/dL<br/>0.80 to &lt; 0.96 mmol/L</td><td>1.5 to &lt; 2.5 mg/dL<br/>0.47 to &lt; 0.80 mmol/L</td><td>&lt; 1.5 mg/dL<br/>&lt; 0.47 mmol/L</td></lln></lln> | 2.5 to < 3.0 mg/dL<br>0.80 to < 0.96 mmol/L | 1.5 to < 2.5 mg/dL<br>0.47 to < 0.80 mmol/L | < 1.5 mg/dL<br>< 0.47 mmol/L |
| Pediatric < 1 Year | 3.5 to <lln dl<br="" mg="">1.12 to <lln l<="" mmol="" td=""><td>2.5 to &lt; 3.5 mg/dL<br/>0.80 to &lt; 1.12 mmol/L</td><td>1.5 to &lt; 2.5 mg/dL<br/>0.47 to &lt; 0.80 mmol/L</td><td>&lt; 1.5 mg/dL<br/>&lt; 0.47 mmol/L</td></lln></lln> | 2.5 to < 3.5 mg/dL<br>0.80 to < 1.12 mmol/L | 1.5 to < 2.5 mg/dL<br>0.47 to < 0.80 mmol/L | < 1.5 mg/dL<br>< 0.47 mmol/L |
| Hyperbilirubinemia<br>Adult and Pediatric<br>> 14 Days | > 1.0 to 1.5 × ULN | > 1.5 to 2.5 × ULN | > 2.5 to 5.0 × ULN | > 5.0 × ULN |
| Infant, ≤ 14 Days (non-hemolytic) | NA | 20.0 to 25.0 mg/dL<br>342 to 428 μmol/L | > 25.0 to 30.0 mg/dL<br>> 428 to 513 μmol/L | > 30.0 mg/dL<br>> 513 μmol/L |
| Infant, ≤ 14 Days (hemolytic) | NA | NA | 20.0 to 25.0 mg/dL<br>342 to 428 µmol/L | > 25.0 mg/dL<br>> 428 μmol/L |
| Blood Urea Nitrogen | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Hyperuricemia | >ULN to 10.0 mg/dL | > 10.0 to 12.0 mg/dL | > 12.0 to 15.0 mg/dL | > 15.0 mg/dL |
| | >ULN to 597 μmol/L | > 597 to 716 μmol/L | > 716 to 895 μmol/L | > 895 μmol/L |
| Hypouricemia Adult and Pediatric ≥ | 1.5 mg/dL to < LLN<br>87 µmol/L to < LLN | 1.0 to < 1.5 mg/dL<br>57 to < 87 μmol/L | 0.5 to < 1.0 mg/dL<br>27 to < 57 μmol/L | < 0.5 mg/dL<br>< 27 μmol/L |
| 1 year Infant < 1 Year | N/A | 1.0 mg/dl to <lln-<br>57 μmol to <lln< td=""><td>0.5 to &lt; 1.0 mg/dL<br/>27 to &lt; 57 μmol/L</td><td>&lt; 0.5 mg/dL<br/>&lt; 27 μmol/L</td></lln<></lln-<br> | 0.5 to < 1.0 mg/dL<br>27 to < 57 μmol/L | < 0.5 mg/dL<br>< 27 μmol/L |
| Creatinine** | > 1.50 to 2.00 mg/dL<br>> 133 to 177 μmol/L | > 2.00 to 3.00 mg/dL<br>> 177 to 265 μmol/L | > 3.00 to 6.00 mg/dL<br>> 265 to 530 μmol/L | > 6.00 mg/dL<br>> 530 μmol/L |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Bicarbonate | 16.0 mEq/L to < LLN | 11.0 to < 16.0 mEq/L | 8.0 to < 11.0 mEq/L | < 8.0 mEq/L |
| Adult and Pediatric<br>≥ 4 Years | 16.0 mmol/L to < LLN | 11.0 to < 16.0 mmol/L | 8.0 to < 11.0 mmol/L | < 8.0 mmol/L |
| Pediatric < 4 Years | NA | 11.0 mEq/L to <lln< td=""><td>8.0 to &lt; 11.0 mEq/L</td><td>&lt; 8.0 mEq/L</td></lln<> | 8.0 to < 11.0 mEq/L | < 8.0 mEq/L |
| | | 11.0 mmol/L to <lln< td=""><td>8.0 to &lt; 11.0 mmol/L</td><td>&lt; 8.0 mmol/L</td></lln<> | 8.0 to < 11.0 mmol/L | < 8.0 mmol/L |
| Triglycerides (Fasting) | NA | 500 to 750 mg/dL<br>5.64–8.47 mmol/L | > 750 to 1200 mg/dL<br>> 8.47–13.55 mmol/L | > 1200 mg/dL<br>> 13.55 mmol/L |
| LDL (Fasting) | 130 to 160 mg/dL | >160 to 190 mg/dL | > 190 mg/dL | NA |
| Adult | 3.35 to 4.15 mmol/L | >4.15 to 4.92 mmol/L | >4.92 mmol/L | |
| LDL (Fasting) | 110 to 130 mg/dL | >130 to 190 mg/dL | > 190 mg/dL | NA |
| Pediatric >2 to <18 years | 2.84 to 3.37 mmol/L | >3.37 to 4.92 mmol/L | >4.92 mmol/L | |
| Hypercholesterolemia | 200 to 239 mg/dL | > 239 to 300 mg/dL | > 300 mg/dL | NA |
| (Fasting) | 5.16 to 6.19 mmol/L | > 6.19 to 7.77 mmol/L | > 7.77 mmol/L | |
| Pediatric < 18 Years | 170 to 199 mg/dL<br>4.39 to 5.15 mmol/L | > 199 to 300 mg/dL<br>> 5.15 to 7.77 mmol/L | > 300 mg/dL<br>> 7.77 mmol/L | NA |
| Creatine Kinase | $3.0 \text{ to} < 6.0 \times \text{ULN}$ | 6.0 to < 10.0 × ULN | 10.0 to < 20.0 × ULN | ≥ 20.0 × ULN |

Calcium should be corrected for albumin if albumin is < 4.0 g/dLAn overlap between the Grade 1 scale and the Lab's normal range for creatinine may result for Male subjects > 70 yrs. Please follow the Gilead convention of grading any result within the LLN and ULN a 0.

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| ALT (SGPT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| GGT | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Alkaline Phosphatase | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Total Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Pancreatic Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Lipase | > 1.0 to 1.5 × ULN | > 1.5 to 3.0 × ULN | > 3.0 to 5.0 × ULN | > 5.0 × ULN |
| Albumin Pediatrics <16 years | - | 2.0 to < LLN g/dL<br>20 to < LLN g/L | < 2.0 g/dL<br>< 20 g/L | NA |
| ≥ 16 years | 3.0 g/dL to < LLN<br>30 g/L to < LLN | 2.0 to < 3.0 g/dL<br>20 to < 30 g/L | < 2.0 g/dL<br>< 20 g/L | NA |

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hematuria (Dipstick) | 1+ | 2+ | 3-4+ | NA |
| Hematuria (Quantitative)<br>See Note below | | | | |
| Females | >ULN - 10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Males | 6-10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Proteinuria (Dipstick) | 1+ | 2–3+ | 4+ | NA |
| Proteinuria, 24 Hour Collection | | | | |
| Adult and Pediatric ≥ 10 Years | 200 to 999 mg/24 h | >999 to 1999 mg/24 h | >1999 to 3500 mg/24 h | > 3500 mg/24 h |
| Pediatric > 3 Mo to < 10 Years | 201 to 499 mg/m <sup>2</sup> /24 h | >499 to 799 mg/m <sup>2</sup> /24 h | >799 to 1000 mg/m <sup>2</sup> /24 h | $> 1000 \text{ mg/ m}^2/24 \text{ h}$ |
| Glycosuria (Dipstick) | 1+ | 2-3+ | 4+ | NA |

#### Notes:

- Toxicity grades for Quantitative and Dipstick Hematuria will be assigned by Covance Laboratory, however for other laboratories, toxicity grades will only be assigned to Dipstick Hematuria.
- With the exception of lipid tests, any graded laboratory test with a result that is between the LLN and ULN should be assigned Grade 0.
- If the severity of a clinical AE could fall under either one of two grades (e.g., the severity of an AE could be either Grade 2 or Grade 3), select the higher of the two grades for the AE.

| | | CARDIOVASCULAR | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac Arrhythmia (general)<br>(By ECG or physical exam) | Asymptomatic AND No intervention indicated | Asymptomatic AND Non-<br>urgent medical intervention<br>indicated | Symptomatic, non-life-<br>threatening AND Non-<br>urgent medical intervention<br>indicated | Life-threatening arrhythmia<br>OR Urgent intervention<br>indicated |
| Cardiac-ischemia/Infarction | NA | NA | Symptomatic ischemia (stable angina) OR Testing consistent with ischemia | Unstable angina OR Acute myocardial infarction |
| Hemorrhage (significant acute blood loss) | NA | Symptomatic AND No transfusion indicated | Symptomatic AND Transfusion of ≤ 2 units packed RBCs (for children ≤ 10 cc/kg) indicated | Life-threatening hypotension<br>OR Transfusion of > 2 units<br>packed RBCs indicated (for<br>children ≤ 10 cc/kg) indicated |
| Hypertension (with repeat testing at same visit) | 140–159 mmHg systolic<br>OR<br>90–99 mmHg diastolic | > 159–179 mmHg systolic<br>OR<br>> 99–109 mmHg diastolic | > 179 mmHg systolic<br>OR<br>> 109 mmHg diastolic | Life-threatening consequences<br>(eg, malignant hypertension)<br>OR Hospitalization (other than<br>ER visit) indicated |
| Pediatric ≤ 17 Years (with repeat testing at same visit) | NA | 91st–94th percentile adjusted<br>for age, height, and gender<br>(systolic and/or diastolic) | ≥ 95th percentile adjusted for age, height, and gender (systolic and/or diastolic) | Life-threatening consequence<br>(eg, malignant hypertension)<br>OR Hospitalization indicated<br>(other than emergency room<br>visit) |
| Hypotension | NA | Symptomatic, corrected with oral fluid replacement | Symptomatic, IV fluids indicated | Shock requiring use of vasopressors or mechanical assistance to maintain blood pressure |
| Pericardial Effusion | Asymptomatic, small effusion requiring no intervention | Asymptomatic, moderate or larger effusion requiring no intervention | Effusion with non-life-<br>threatening physiologic<br>consequences OR Effusion<br>with nonurgent intervention<br>indicated | Life-threatening consequence<br>(eg, tamponade) OR Urgent<br>intervention indicated |

| | CARDIOVASCULAR | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Prolonged PR Interval | PR interval 0.21 to 0.25 sec | PR interval > 0.25 sec | Type II 2nd degree AV<br>block OR Ventricular pause<br>> 3.0 sec | Complete AV block |
| Pediatric ≤ 16 Years | 1st degree AV block<br>(PR > normal for age and<br>rate) | Type I 2nd degree AV block | Type II 2nd degree AV block | Complete AV block |
| Prolonged QTc | Asymptomatic, QTc interval 0.45 to 0.47 sec OR Increase interval < 0.03 sec above baseline | Asymptomatic, QTc interval 0.48 to 0.49 sec OR Increase in interval 0.03 to 0.05 sec above baseline | Asymptomatic, QTc interval ≥ 0.50 sec OR Increase in interval ≥ 0.06 sec above baseline | Life-threatening<br>consequences, eg, Torsade de<br>pointes or other associated<br>serious ventricular<br>dysrhythmia |
| Pediatric ≤ 16 Years | Asymptomatic, QTc interval 0.450 to 0.464 sec | Asymptomatic, QTc interval 0.465 to 0.479 sec | Asymptomatic, QTc interval ≥ 0.480 sec | Life-threatening<br>consequences, eg, Torsade de<br>pointes or other associated<br>serious ventricular<br>dysrhythmia |
| Thrombosis/Embolism | NA | Deep vein thrombosis AND<br>No intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Deep vein thrombosis AND<br>Intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Embolic event (eg, pulmonary embolism, life-threatening thrombus) |
| Vasovagal Episode (associated with a procedure of any kind) | Present without loss of consciousness | Present with transient loss of consciousness | NA | NA |
| Ventricular Dysfunction<br>(congestive heart failure,<br>CHF) | NA | Asymptomatic diagnostic finding AND intervention indicated | New onset with symptoms<br>OR Worsening symptomatic<br>CHF | Life-threatening CHF |

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Bronchospasm (acute) | FEV1 or peak flow reduced to 70% to 80% | FEV1 or peak flow 50% to 69% | FEV1 or peak flow 25% to 49% | Cyanosis OR FEV1 or peak flow < 25% OR Intubation |
| Dyspnea or Respiratory<br>Distress | Dyspnea on exertion with no or minimal interference with usual social & functional activities | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities | Dyspnea at rest causing inability to perform usual social & functional activities | Respiratory failure with ventilatory support indicated |
| Pediatric < 14 Years | Wheezing OR minimal increase in respiratory rate for age | Nasal flaring OR Intercostal retractions OR Pulse oximetry 90% to 95% | Dyspnea at rest causing inability to perform usual social & functional activities OR Pulse oximetry < 90% | Respiratory failure with ventilatory support indicated |

| OCULAR/VISUAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Uveitis | Asymptomatic but detectable on exam | Symptomatic anterior uveitis OR<br>Medical intervention indicated | Posterior or pan-uveitis OR<br>Operative intervention<br>indicated | Disabling visual loss in affected eye(s) |
| Visual Changes (from baseline) | Visual changes causing no or minimal interference with usual social & functional activities | Visual changes causing greater than minimal interference with usual social & functional activities | Visual changes causing inability to perform usual social & functional activities | Disabling visual loss in affected eye(s) |

| SKIN | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alopecia | Thinning detectable by study participant or caregiver (for disabled adults) | Thinning or patchy hair loss detectable by health care provider | Complete hair loss | NA |
| Cutaneous Reaction – Rash | Localized macular rash | Diffuse macular,<br>maculopapular, or<br>morbilliform rash OR Target<br>lesions | Diffuse macular,<br>maculopapular, or morbilliform<br>rash with vesicles or limited<br>number of bullae OR<br>Superficial ulcerations of<br>mucous membrane limited to<br>one site | Extensive or generalized<br>bullous lesions OR<br>Stevens-Johnson syndrome<br>OR Ulceration of mucous<br>membrane involving two<br>or more distinct mucosal<br>sites OR Toxic epidermal<br>necrolysis (TEN) |
| Hyperpigmentation | Slight or localized | Marked or generalized | NA | NA |
| Hypopigmentation | Slight or localized | Marked or generalized | NA | NA |
| Pruritis (itching – no skin lesions) (See also Injection Site Reactions: Pruritis associated with injection) | Itching causing no or<br>minimal interference with<br>usual social & functional<br>activities | Itching causing greater than minimal interference with usual social & functional activities | Itching causing inability to perform usual social & functional activities | NA |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite associated with decreased oral intake without significant weight loss | Loss of appetite associated with significant weight loss | Life-threatening consequences<br>OR Aggressive intervention<br>indicated [eg, tube feeding or<br>total parenteral nutrition] |
| Ascites | Asymptomatic | Symptomatic AND Intervention indicated (eg, diuretics or therapeutic paracentesis) | Symptomatic despite intervention | Life-threatening consequences |
| Cholecystitis | NA | Symptomatic AND Medical intervention indicated | Radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences (eg, sepsis or perforation) |
| Constipation | NA | Persistent constipation requiring regular use of dietary modifications, laxatives, or enemas | Obstipation with manual evacuation indicated | Life-threatening consequences (eg, obstruction) |
| Diarrhea<br>Adult and Pediatric<br>≥ 1 Year | Transient or intermittent episodes of unformed stools OR Increase of ≤ 3 stools over baseline/24 hr | Persistent episodes of unformed to watery stools OR Increase of 4–6 stools over baseline per 24 hrs. | Bloody diarrhea OR Increase<br>of ≥ 7 stools per 24-hour<br>period OR IV fluid<br>replacement indicated | Life-threatening consequences (eg, hypotensive shock) |
| Pediatric < 1 Year | Liquid stools (more<br>unformed than usual) but<br>usual number of stools | Liquid stools with increased<br>number of stools OR Mild<br>dehydration | Liquid stools with moderate dehydration | Liquid stools resulting in<br>severe dehydration with<br>aggressive rehydration<br>indicated OR Hypotensive<br>shock |
| Dysphagia-Odynophagia | Symptomatic but able to eat usual diet | Symptoms causing altered dietary intake without medical intervention indicated | Symptoms causing severely altered dietary intake with medical intervention indicated | Life-threatening reduction in oral intake |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucositis/Stomatitis<br>(clinical exam)<br>See also Proctitis,<br>Dysphagia-Odynophagia | Erythema of the mucosa | Patchy pseudomembranes or ulcerations | Confluent pseudomembranes or ulcerations OR Mucosal bleeding with minor trauma | Tissue necrosis OR Diffuse<br>spontaneous mucosal bleeding<br>OR Life-threatening<br>consequences (eg, aspiration,<br>choking) |
| Nausea | Transient (< 24 hours) or intermittent nausea with no or minimal interference with oral intake | Persistent nausea resulting in decreased oral intake for 24–48 hours | Persistent nausea resulting in minimal oral intake for > 48 hours OR Aggressive rehydration indicated (eg, IV fluids) | Life-threatening consequences (eg, hypotensive shock) |
| Pancreatitis | NA | Symptomatic AND<br>Hospitalization not indicated<br>(other than ER visit) | Symptomatic AND<br>Hospitalization indicated<br>(other than ER visit) | Life-threatening consequences<br>(eg, sepsis, circulatory failure,<br>hemorrhage) |
| Proctitis (functional-<br>symptomatic) Also see Mucositis/<br>Stomatitis for Clinical<br>Exam | Rectal discomfort AND No intervention indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social/ functional activities OR Operative intervention indicated | Life-threatening consequences (eg, perforation) |
| Vomiting | Transient or intermittent vomiting with no or minimal interference with oral intake | Frequent episodes of vomiting with no or mild dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated | Life-threatening consequences (eg, hypotensive shock) |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alteration in Personality-Behavior or in Mood (eg, agitation, anxiety, depression, mania, psychosis) | Alteration causing no or minimal interference with usual social & functional activities | Alteration causing greater than minimal interference with usual social & functional activities | Alteration causing inability to perform usual social & functional activities | Behavior potentially harmful<br>to self or others (eg,<br>suicidal/homicidal ideation or<br>attempt, acute psychosis) OR<br>Causing inability to perform<br>basic self-care functions |
| Altered Mental Status For Dementia, see Cognitive and Behavioral/Attentional Disturbance (including dementia and ADD) | Changes causing no or minimal interference with usual social & functional activities | Mild lethargy or somnolence<br>causing greater than minimal<br>interference with usual social<br>& functional activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR obtundation, OR coma |
| Ataxia | Asymptomatic ataxia detectable on exam OR Minimal ataxia causing no or minimal interference with usual social & functional activities | Symptomatic ataxia causing greater than minimal interference with usual social & functional activities | Symptomatic ataxia causing inability to perform usual social & functional activities | Disabling ataxia causing inability to perform basic self-care functions |
| Cognitive and Behavioral/Attentional Disturbance (including dementia and Attention Deficit Disorder) | Disability causing no or<br>minimal interference with<br>usual social & functional<br>activities OR Specialized<br>resources not indicated | Disability causing greater than minimal interference with usual social & functional activities OR Specialized resources on part-time basis indicated | Disability causing inability to<br>perform usual social &<br>functional activities OR<br>Specialized resources on a<br>full-time basis indicated | Disability causing inability to perform basic self-care functions OR Institutionalization indicated |
| CNS Ischemia (acute) | NA | NA | Transient ischemic attack | Cerebral vascular accident (CVA, stroke) with neurological deficit |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Developmental delay –<br>Pediatric ≤ 16 Years | Mild developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Moderate developmental<br>delay, either motor or<br>cognitive, as determined by<br>comparison with a<br>developmental screening tool<br>appropriate for the setting | Severe developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Developmental regression,<br>either motor or cognitive, as<br>determined by comparison<br>with a developmental<br>screening tool appropriate for<br>the setting |
| Headache | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated (other than ER visit) OR Headache with significant impairment of alertness or other neurologic function |
| Insomnia | NA | Difficulty sleeping causing greater than minimal interference with usual social/functional activities | Difficulty sleeping causing inability to perform usual social & functional activities | Disabling insomnia causing inability to perform basic self-care functions |
| Neuromuscular Weakness<br>(including myopathy &<br>neuropathy) | Asymptomatic with decreased strength on exam OR Minimal muscle weakness causing no or minimal interference with usual social & functional activities | Muscle weakness causing greater than minimal interference with usual social & functional activities | Muscle weakness causing inability to perform usual social & functional activities | Disabling muscle weakness<br>causing inability to perform<br>basic self-care functions OR<br>Respiratory muscle weakness<br>impairing ventilation |
| Neurosensory Alteration<br>(including paresthesia and<br>painful neuropathy) | Asymptomatic with sensory alteration on exam or minimal paresthesia causing no or minimal interference with usual social & functional activities | Sensory alteration or<br>paresthesia causing greater<br>than minimal interference with<br>usual social & functional<br>activities | Sensory alteration or paresthesia causing inability to perform usual social & functional activities | Disabling sensory alteration or<br>paresthesia causing inability to<br>perform basic self-care<br>functions |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Seizure: (new onset) | NA | 1 seizure | 2–4 seizures | Seizures of any kind that are<br>prolonged, repetitive (eg,<br>status epilepticus), or difficult<br>to control (eg, refractory<br>epilepsy) |
| Seizure: (pre-existing) For Worsening of Existing Epilepsy the Grades Should Be Based on an Increase from Previous Level of Control to Any of These Levels | NA | Increased frequency of pre-<br>existing seizures (non-<br>repetitive) without change in<br>seizure character OR<br>infrequent breakthrough<br>seizures while on stable meds<br>in a previously controlled<br>seizure disorder | Change in seizure character<br>from baseline either in<br>duration or quality (eg,<br>severity or focality) | Seizures of any kind that are prolonged, repetitive (eg, status epilepticus), or difficult to control (eg, refractory epilepsy) |
| Seizure – Pediatric < 18 Years | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>< 5 minutes with < 24 hours<br>post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting 5–20<br>minutes with<br>< 24 hours post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>> 20 minutes | Seizure, generalized onset<br>with or without secondary<br>generalization, requiring<br>intubation and sedation |
| Syncope (not associated with a procedure) | NA | Present | NA | NA |
| Vertigo | Vertigo causing no or<br>minimal interference with<br>usual social & functional<br>activities | Vertigo causing greater than minimal interference with usual social & functional activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo causing inability to perform basic self-care functions |

| | MUSCULOSKELETAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Arthralgia<br>See also Arthritis | Joint pain causing no or minimal interference with usual social & functional activities | Joint pain causing greater than minimal interference with usual social & functional activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain causing inability to perform basic self-care functions |
| Arthritis<br>See also Arthralgia | Stiffness or joint swelling causing no or minimal interference with usual social & functional activities | Stiffness or joint swelling causing greater than minimal interference with usual social & functional activities | Stiffness or joint swelling causing inability to perform usual social & functional activities | Disabling joint stiffness or<br>swelling causing inability to<br>perform basic self-care<br>functions |
| Bone Mineral Loss | BMD t-score or z-score<br>-2.5 to -1.0 | BMD t-score or z-score < -2.5 | Pathological fracture<br>(including loss of vertebral<br>height) | Pathologic fracture causing life-threatening consequences |
| Pediatric < 21 Years | BMD z-score<br>-2.5 to -1.0 | BMD z-score < -2.5 | Pathological fracture (including loss of vertebral height) | Pathologic fracture causing life-threatening consequences |
| Myalgia<br>(non-injection site) | Muscle pain causing no or minimal interference with usual social & functional activities | Muscle pain causing greater than minimal interference with usual social & functional activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle pain causing inability to perform basic self-care functions |
| Osteonecrosis | NA | Asymptomatic with radiographic findings AND No operative intervention indicated | Symptomatic bone pain with radiographic findings OR Operative intervention indicated | Disabling bone pain with radiographic findings causing inability to perform basic self-care functions |

| | SYSTEMIC | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Acute Systemic Allergic<br>Reaction | Localized urticaria<br>(wheals) with no medical<br>intervention indicated | Localized urticaria with medical intervention indicated OR Mild angioedema with no medical intervention indicated | Generalized urticaria OR<br>Angioedema with medical<br>intervention indicated OR<br>Symptomatic mild<br>bronchospasm | Acute anaphylaxis OR Life-<br>threatening bronchospasm OR<br>laryngeal edema |
| Chills | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Fatigue<br>Malaise | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating fatigue/malaise<br>symptoms causing inability to<br>perform basic self-care<br>functions |
| Fever (nonaxillary) | 37.7°C to 38.6°C<br>99.8°F to 101.5°F | 38.7°C to 39.3°C<br>101.6°F to 102.8°F | 39.4°C to 40.5°C<br>102.9°F to 104.9°F | > 40.5°C<br>> 104.9°F |
| Pain- Indicate Body Site<br>See also Injection Site<br>Pain, Headache,<br>Arthralgia, and Myalgia | Pain causing no or<br>minimal interference with<br>usual social & functional<br>activities | Pain causing greater than minimal interference with usual social & functional activities | Pain causing inability to perform usual social & functional activities | Disabling pain causing inability to perform basic self-care functions OR Hospitalization (other than ER visit) indicated |
| Unintentional Weight<br>Loss | NA | 5% to 9% loss in body weight from baseline | 10% to 19% loss in body weight from baseline | ≥ 20% loss in body weight<br>from baseline OR Aggressive<br>intervention indicated [eg,<br>tube feeding or total parenteral<br>nutrition] |

| INJECTION SITE REACTION | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Injection Site Pain (pain<br>without touching)<br>Or Tenderness (pain when<br>area is touched) | Pain/tenderness causing no or minimal limitation of use of limb | Pain/tenderness limiting use of limb OR Pain/tenderness causing greater than minimal interference with usual social & functional activities | Pain/tenderness causing inability to perform usual social & functional activities | Pain/tenderness causing inability<br>to perform basic self-care<br>function OR Hospitalization<br>(other than ER visit) indicated<br>for management of<br>pain/tenderness |
| Injection Site Reaction (Localized), > 15 Years | Erythema OR Induration<br>of $5 \times 5$ cm to $9 \times 9$ cm (or<br>$25-81 \times \text{cm}^2$ ) | Erythema OR Induration OR<br>Edema > 9 cm any diameter<br>(or > 81 cm <sup>2</sup> ) | Ulceration OR Secondary<br>infection OR Phlebitis OR<br>Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pediatric ≤ 15 Years | Erythema OR Induration OR Edema present but ≤ 2.5 cm diameter | Erythema OR Induration OR Edema > 2.5 cm diameter but < 50% surface area of the extremity segment (eg, upper arm/thigh) | Erythema OR Induration OR Edema involving ≥ 50% surface area of the extremity segment (eg, upper arm/thigh) OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pruritis Associated with Injection See also Skin: Pruritis (itching—no skin lesions) | Itching localized to injection<br>site AND Relieved<br>spontaneously or with<br>< 48 h treatment | Itching beyond the injection site but not generalized OR Itching localized to injection site requiring ≥ 48 h treatment | Generalized itching causing inability to perform usual social & functional activities | NA |

| ENDOCRINE/METABOLIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Lipodystrophy (eg, back of neck, breasts, abdomen) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious changes on casual visual inspection | NA |
| Diabetes Mellitus | NA | New onset without need to initiate medication OR Modification of current meds to regain glucose control | New onset with initiation of indicated med OR Diabetes uncontrolled despite treatment modification | Life-threatening consequences (eg, ketoacidosis, hyperosmolar non-ketotic coma) |
| Gynecomastia | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |
| Hyperthyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, thyroid storm) |
| Hypothyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, myxedema coma) |
| Lipoatrophy (eg, fat loss from the face, extremities, buttocks) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |

| GENITOURINARY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Intermenstrual Bleeding (IMB) | Spotting observed by participant<br>OR Minimal blood observed<br>during clinical or colposcopic<br>exam | Intermenstrual bleeding not greater in duration or amount than usual menstrual cycle | Intermenstrual bleeding greater in duration or amount than usual menstrual cycle | Hemorrhage with life-<br>threatening hypotension OR<br>Operative intervention<br>indicated |
| Urinary Tract<br>obstruction (eg, stone) | NA | Signs or symptoms of urinary tract obstruction without hydronephrosis or renal dysfunction | Signs or symptoms of urinary tract obstruction with hydronephrosis or renal dysfunction | Obstruction causing life-<br>threatening consequences |

| INFECTION | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Infection (any other than HIV infection) | Localized, no systemic antiµbial treatment indicated AND Symptoms causing no or minimal interference with usual social & functional activities | Systemic antiµbial treatment indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Systemic antiµbial treatment indicated AND Symptoms causing inability to perform usual social & functional activities OR Operative intervention (other than simple incision and drainage) indicated | Life-threatening consequences (eg, septic shock) |

Basic Self-care Functions: Activities such as bathing, dressing, toileting, transfer/movement, continence, and feeding.

Usual Social & Functional Activities: Adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, pursuing a hobby, etc.

Appendix 4. Child-Pugh-Turcotte Classification of the severity of cirrhosisa

| | POINTS* | | |
|---|---|---|---|
| | 1 | 2 | 3 |
| Encephalopathy | None | Grade 1-2<br>(or precipitant-induced) | Grade3-4<br>(or chronic) |
| Ascites | None | Mild/Moderate<br>(diuretic-responsive) | Severe<br>(diuretic-refractory) |
| Bilirubin (mg/dL) | < 2 | 2-3 | > 3 |
| Albumin (g/dL) | > 3.5 | 2.8-3.5 | < 2.8 |
| PT (sec prolonged) or INR | < 4<br>< 1.7 | 4-6<br>1.7-2.3 | > 6<br>> 2.3 |

CPT score is obtained by adding the score for each parameter

CPT  $\overline{\text{class}}$ : A = 5-6 points

B = 7-9 points

C = 10-15 points

a U.S. Department of Veterans Affairs. Child -Pugh-Turcotte Classification of the severity of cirrhosis. Available at http://www.hepatitis.va.gov/provider/tools/child-pugh-calculator.asp, Accessed May 29, 2012.

# Appendix 5. Banff Criteria\*

Table 1. Grading of Acute Liver Allograft Rejection

| Global Assessment* | Criteria |
|---|---|
| Indeterminate | Portal inflammatory infiltrate that fails to meet the<br>criteria for the diagnosis of acute rejection (see text) |
| Mild | Rejection infiltrate in a minority of the triads, that is<br>generally mild, and confined within the portal<br>spaces |
| Moderate | Rejection infiltrate, expanding most or all of the triads |
| Severe | As above for moderate, with spillover into periportal<br>areas and moderate to severe perivenular<br>inflammation that extends into the hepatic<br>parenchyma and is associated with perivenular<br>hepatocyte necrosis |

NOTE. Global assessment of rejection grade mode on a review of the biopsy and after the diagnosis of rejection has been established.

<sup>\*</sup> Verbal description of mild, moderate, or severe acute rejection could also be labeled as Grade I, II, and III, respectively.

<sup>\*</sup> Demetris et al., Banff Schema for Grading Liver Allograft Rejection: An International Consensus Document. Hepatology 1997;25:658-663

# Appendix 6. Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements

# 1) Definitions

# a. Definition of Female of Childbearing Potential

For the purposes of this study, a female born subject is considered of childbearing potential following the initiation of menarche until becoming post-menopausal, unless permanently sterile or with medically documented ovarian failure.

Women are considered to be in a postmenopausal state when they are  $\geq$  54 years of age with cessation of previously occurring menses for  $\geq$  12 months without an alternative cause.

#### b. Definition of Male Fertility

For the purposes of this study, a male born subject is considered of fertile after the initiation of puberty unless permanently sterile by bilateral orchidectomy or medical documentation.

#### 2) Study Drug Effects on Pregnancy and Hormonal Contraception

Data from clinical pharmacokinetic interaction studies of SOF have demonstrated that there is no reduction in the clinical efficacy of hormonal contraception. Non-clinical toxicity studies of SOF have demonstrated no adverse effect on fertility or embryo-fetal development.

Data from clinical pharmacokinetic interaction studies of VEL have demonstrated that there is no reduction in the clinical efficacy of hormonal contraception. Non-clinical toxicity studies of GS-5816 have demonstrated no adverse effect on fertility or embryo-fetal development

However, the risks of treatment with SOF/VEL during pregnancy in humans have not been evaluated. Please refer to the latest version of the investigator's brochure for additional information.

# 3) Contraception Requirements for Female Subjects of Childbearing Potential

The inclusion of female subjects of childbearing potential requires using at least an acceptable effective contraceptive measure. They must have a negative serum pregnancy test at Screening and a negative pregnancy test on the Baseline/Day 1 visit prior to randomization. A pregnancy test will be performed at the Post Treatment Week 4 visit. They must also agree to one of the following from Screening until 30 days after the last dose of SOF/VEL.

• Complete abstinence from intercourse of reproductive potential. Abstinence is an acceptable method of contraception only when it is in line with the subject's preferred and usual lifestyle.

Or

- Consistent and correct use of 1 of the following methods of birth control listed below, in addition to a male partner who correctly used a condom from the date of Screening until 30 days after the last dose of SOF/VEL.
  - Intrauterine device (IUD)
  - Intrauterine hormone-releasing system (IUS)
  - Tubal sterilization
  - Essure micro-insert system
  - Vasectomy in the male partner
  - Barrier methods
    - Female barriers: Diaphragm with spermicide or Cervical cap with spermicide
    - Male barriers: Male condom (with or without spermicide)
  - Hormonal methods
    - Oral contraceptives (either combined or progesterone only)
    - Injectable progesterone
    - Implants of levonorgestrel or etonorgestrel
    - Transdermal contraceptive patch
    - Contraceptive vaginal ring

Female subjects must also refrain from egg donation and in vitro fertilization during study treatment and until at least 30 days after the last dose of SOF/VEL.

# 4) Contraception Requirements for Male Subjects

During the study, male subjects with female partners of childbearing potential should use condoms until 30 days after the last dose of SOF/VEL treatment when engaging in intercourse of reproductive potential. If their female partner is of childbearing potential (as defined above), their female partner must use 1 of the methods of birth control listed above from the date of Screening until 30 days after the last dose of SOF/VEL.

Male subjects must agree to refrain from sperm donation for at least 30 days after the last dose of SOF/VEL.

# 5) Unacceptable Birth Control Methods

Birth control methods that are unacceptable include periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM). Female condom and male condom should not be used together.

# 6) Procedures to be Followed in the Event of Pregnancy

Subjects will be instructed to notify the investigator if they become pregnant at any time during the study or if they become pregnant within 30 days of last dose of SOF/VEL. Subjects who become pregnant or who suspect that they are pregnant during the study must report the information to the investigator and discontinue study drug immediately. Subjects whose partner has become pregnant or suspects she is pregnant must report the information to the investigator.

Instructions for reporting pregnancy, partner pregnancy, and pregnancy outcome are outlined in Section 7.6.2.1.